Statistical Analysis Plan

AC-080A201

Multi-center, double-blind, double-dummy, randomized, placebo- and active-reference, parallel group, Phase 2 dose-finding study with ACT-132577 in subjects with essential hypertension (grade 1 and 2)

ClinicalTrials.gov Identifier: NCT02603809

This study was sponsored by Actelion Pharmaceuticals - study sponsorship was transferred to Idorsia Pharmaceuticals Ltd.



# STATISTICAL ANALYSIS PLAN FOR CLINICAL STUDY REPORT

# **STUDY AC-080A201**

Multi-center, double-blind, double-dummy, randomized, placebo- and active-reference, parallel group, Phase 2 dose-finding study with ACT-132577 in subjects with essential hypertension (grade 1 and 2)

Purpose of Analysis
Investigational Drug
ACT-132577
Protocol Number
AC-080A201
Actelion Document Number
D-17.304
Document Status/Version Number
Final Version 2.0
15 May 2017

Authors

, Expert Statistician

, Medical Science Expert

, Senior Clinical Project

Scientist

, Senior Expert Statistician

, Head of Biostatistics

, Senior Trial Data Scientist

, Senior Drug Safety Physician

, Global Clinical Project Management

, Senior Clinical

Pharmacologist

, Global DRA Project Leader


May not be used, divulged, published or otherwise disclosed without the consent of Actelion Pharmaceuticals Ltd

# TABLE OF CONTENTS

| LI | ST OF ABBE | VIATIONS AND ACRONYMS | 7 |
|----|------------|-----------------------------------------------------|----|
| 1 | INTRODUC | TION | 9 |
| 2 | STUDY DE | SIGN AND FLOW | 9 |
| | 2.1 Stu | dy design | 9 |
| | | dy visit and assessment schedule | |
| 3 | OBJECTIVE | ES | 13 |
| | 3.1 Prii | mary objective(s) | 13 |
| | | condary objectives | |
| | 3.3 Oth | ner objectives | 13 |
| 4 | | OR CLARIFICATIONS TO ANALYSES PLANNED IN T | |
| | STUDY PRO | OTOCOL | 13 |
| | 4.1 Cha | anges to the analyses planned in the study protocol | 13 |
| | 4.1.1 | Analysis sets | |
| | 4.1.2 | Analyses of the secondary efficacy variables | 13 |
| | 4.1.3 | | 15 |
| | 4.2 Cha | anges in the conduct of the study / data collection | 15 |
| 5 | DEFINITIO | NS OF VARIABLES | 15 |
| | 5.1 Sub | pjects disposition | 15 |
| | | oject characteristics | |
| | 5.2.1 | Demographics | 16 |
| | 5.2.2 | Baseline disease characteristics | 16 |
| | 5.2.3 | Other baseline characteristics | |
| | 5.2.4 | Medical history | |
| | 5.2.5 | Previous and concomitant therapies | |
| | 5.2.6 | Other subject characteristics | |
| | | dy treatment duration and compliance | |
| | 5.3.1 | Study treatment duration | |
| | 5.3.2 | Compliance with study treatment | |
| | 5.3.3 | Study treatment discontinuation | |
| | 5.3.4 | Study treatment adjustments or interruptions | |
| | | dy discontinuation | |
| | | icacy variables | |
| | 5.5.1 | Primary efficacy endpoint(s) | 20 |

| | 5.5.2 Secondary efficacy endpoints | |
|---|--------------------------------------------------------------------|----|
| | 5.5.3 Other efficacy endpoints | 22 |
| | 5.5.3.1 Illustration of derivation of ABPM endpoints | |
| | 5.6 Safety variables | 25 |
| | 5.6.1 Adverse events | 25 |
| | 5.6.1.1 Treatment-emergent adverse events | 26 |
| | 5.6.1.2 Frequency of treatment-emergent adverse events | 26 |
| | 5.6.1.3 Intensity of treatment-emergent adverse events | |
| | 5.6.1.4 Relationship of treatment-emergent adverse events | |
| | 5.6.2 Deaths | |
| | 5.6.3 Serious adverse events | 27 |
| | 5.6.4 Adverse events leading to discontinuation of study treatment | |
| | 5.6.5 Other adverse events | |
| | 5.6.6 Physical examination, vital signs and body weight | |
| | 5.6.7 Electrocardiogram | |
| | 5.6.7.1 Treatment-emergent ECG abnormalities | |
| | 5.6.8 Laboratory | |
| | 5.6.8.1 Treatment-emergent marked laboratory abnormalities | |
| | 5.6.9 Other safety variables | |
| | 5.7 Quality of life variables | |
| | 5.8 Pharmacoeconomic variables | |
| | 5.9 Pharmacodynamic variables | |
| | 5.10 Pharmacokinetic variables | |
| 6 | DEFINITION OF PROTOCOL DEVIATIONS | 32 |
| 7 | ANALYSIS SETS | 33 |
| | 7.1 Definitions of analysis sets | |
| | 7.1.1 Screened Set | |
| | 7.1.2 Run-in Set | |
| | 7.1.3 All Randomized Set | |
| | 7.1.4 Full Analysis Set | |
| | 7.1.5 Per-Protocol Set | |
| | 7.1.6 Safety Set | |
| | 7.1.7 Pharmacokinetic Set | 34 |
| 3 | DEFINITION OF SUBGROUPS | 34 |
| ) | GENERAL STATISTICAL METHODOLOGY | 34 |
| | 9.1 Missing data | 35 |
| | 9.2 Dose-response analysis for the primary endpoint | |
| | 1 J T T T T T T T T T T T T T T T T T T | |

| | 9.3 | Dose-1 | response analyses for continuous data | 38 |
|---|---|---|---|---|
| | 9.4 | | response analyses for binary data | |
| 10 | STATIS | STICAL | ANALYSES | 40 |
| | 10.1 | Overa | Il testing strategy | 40 |
| | 10.2 | | al rules for data presentations | |
| | 10.3 | | y of subject disposition, protocol deviations and analysis sets | |
| | 10. | 3.1 | Subject disposition | |
| | 10. | 3.2 | Protocol deviations | 4 |
| | 10. | 3.3 | Analysis sets | 42 |
| | 10.4 | Analy | ses of subject characteristics | |
| | 10. | 4.1 | Demographics | 42 |
| | 10. | 4.2 | Baseline disease characteristics | 42 |
| | 10. | 4.3 | Other baseline characteristics. | 42 |
| | 10. | 4.4 | Medical history | 42 |
| | 10. | 4.5 | Previous and concomitant therapies | 43 |
| | 10. | 4.6 | Other subject characteristics | 43 |
| | 10.5 | Analy | sis of study treatment duration and compliance | |
| | 10. | 5.1 | Study treatment duration | |
| | 10. | 5.2 | Compliance with study treatment | 44 |
| | 10. | 5.3 | Study treatment discontinuation | |
| | 10. | 5.4 | Study treatment adjustments or interruptions | 44 |
| | 10. | 5.5 | Study withdrawal | |
| | 10.6 | Analy | sis of the primary efficacy variable(s) | |
| | 10. | 6.1 | Hypothesis and statistical model | |
| | | 6.2 | Handling of missing data | |
| | | 6.3 | Main analysis | |
| | | 6.4 | Supportive/sensitivity analyses | |
| | | 6.5 | Subgroup analyses | |
| | 10.7 | | sis of the secondary efficacy variables | |
| | 10.8 | | sis of other efficacy variables | |
| | 10.9 | | sis of safety variables | |
| | | 9.1 | Adverse events | |
| | 10. | 9.2 | Deaths, other serious adverse events | |
| | | 10.9.2 | | |
| | | 10.9.2 | | 5 |
| | | 10.9.2 | | |
| | | 1005 | discontinuations | |
| | 4.0 | 10.9.2 | | |
| | | 9.3 | Electrocardiography (ECG) | 52 |
| | 10. | 9.4 | Laboratory tests | |
| | | 1094 | 1 Treatment-emergent marked laboratory abnormalities | - 50 |

| | 10.9. | Physical examination, vital signs and body weight | 53 |
|---|---|---|---|
| | 10.9.0 | 6 Other safety variables | 54 |
| | 10.10 A | Analysis of quality of life variables (TSQM vII) | 54 |
| | 10.11 A | Analysis of pharmacoeconomic variables | 54 |
| | 10.12 A | Analysis of epidemiological measures and risk-benefit evaluations | 54 |
| | | Analysis of pharmacodynamic variables | |
| | | Analysis of pharmacokinetic variables | |
| 11 | GENERA | L DEFINITIONS AND DERIVATIONS | 55 |
| | 11.1 Т | ime windows | 55 |
| | 11.2 F | Run-in treatment start date/time | 56 |
| | | Run-in treatment end date/time | |
| | 11.4 F | Randomization date/time | 56 |
| | | Oouble-blind treatment start date/time | |
| | | Double-blind treatment end date/time | |
| | | Vithdrawal period start date/time | |
| | | Vithdrawal period end date/time | |
| | | Study day | |
| | | Ouration of essential hypertension (years) | |
| | | Jnit conversion rules | |
| | | Body Mass Index (BMI) | |
| 12 | HANDLI | NG OF MISSING/INCOMPLETE DATE AND TIME FIELDS | 58 |
| 13 | LIST OF S | SUMMARY TABLES, LISTINGS AND FIGURES | 61 |
| | 13.1 S | Subject disposition | 61 |
| | | Protocol deviations | |
| | | Subject characteristics | |
| | 13.3. | <b>.</b> | |
| | 13.3.2 | | |
| | 13.3.3 | | |
| | 13.3.4 | | |
| | 13.3.5 | , | |
| | 13.3.0 | 1 | |
| | 13.3. | | |
| | | Study treatment duration and compliance | |
| | 13.4. | · | |
| | 13.4.2 | · | |
| | 13.4.3 | F | |
| | 13.4.4 | • | |
| | | Study withdrawal | |

| 13.6 | Primary efficacy analyses | 67 |
|---|---|---|
| | 13.6.1 Main analysis | |
| 1 | 13.6.2 Supportive/sensitivity analyses | 70 |
| 1 | 13.6.3 Subgroup analyses | 74 |
| 13.7 | Secondary efficacy analyses | |
| 13.8 | Other efficacy analyses | 84 |
| 13.9 | | |
| 1 | 13.9.1 Adverse events | 87 |
| 1 | 13.9.2 Deaths | 88 |
| 1 | 13.9.3 Serious adverse events | 88 |
| 1 | 13.9.4 Adverse events leading to treatment discontinuation | 89 |
| 13.10 | Electrocardiogram (ECG) | 90 |
| 13.11 | Laboratory tests | 90 |
| 13.12 | Physical examination, vital signs and body weight | 93 |
| 13.13 | 3 Other safety variables | 93 |
| 13.14 | 4 Other evaluations | 92 |
| 1 | 13.14.1 PK | 94 |
| 1 | 13.14.2 PD | 92 |
| 14 REFI | ERENCES | 95 |
| 15 APPI | ENDICES | 97 |
| | LIST OF TABLES | |
| Table 1 | Visit and assessment schedule | 11 |
| Table 2 | Thresholds for marked laboratory abnormalities | |
| Table 3 | Parameterization of models considered in MCP-Mod analyses | |
| Table 4 | Summary of efficacy analyses | |
| Table 5 | Visit time windows | |
| | LIST OF FIGURES | |
| Figure 1 | Example DBP and SBP measured by ABPM | 2/ |
| Figure 2 | Dose-response curves considered in MCP-Mod procedure | 22<br>3 <i>6</i> |
| Figure 3 | Examples of E <sub>max</sub> dose-response relationships | |
| | LIST OF APPENDICES | |
| A. | Protocol synopsis | 97 |
| B. | Calculation of mean blood pressure measurements based on ABPM | 105 |
| C. | Calculation of trough-peak ratios based on ABPM | |
| D. | Document history | 110 |

AC-080A201 15 May 2017, page 7/110

# LIST OF ABBEVIATIONS AND ACRONYMS

Statistical Analysis Plan

Doc No D-17.304

**ABPM** Ambulatory blood pressure monitoring Adverse event AΕ Akaike's Information Criterion AIC ALT Alanine aminotransferase Analysis of covariance ANCOVA AP Alkaline phosphatase Aspartate aminotransferase **AST** ATC Anatomic therapeutic chemical Below the limit of quantification BLQ **Body Mass Index** BMI Baseline observation carried forward **BOCF** BP Blood pressure CI Confidence interval DB Double-blind DBP Diastolic blood pressure **ECG** Electrocardiogram eCRF **Electronic Case Report Form** Maximum effect  $E_{max}$ EOS End-of-Study **End-of-Treatment** EOT ET Endothelin **EudraCT** European Clinical Trials Database **FAS** Full Analysis Set **FDA** Food and Drug Administration (US) HR Heart rate Interactive Voice Response System **IVRS** Last observation carried forward LOCF Least Squares Means LSMeans MAR Missing at random MCP-Mod Multiple Comparison Procedure – Modeling MCT Multiple Contrast Test MedDRA Medical Dictionary for Regulatory Activities o.d. Once a day **OBPM** (automated) Office blood pressure measurement

Observed cases

OC

| ACT-132577 | | Statistical Analysis Plan |
|------------------------|--------------|---------------------------|
| AC-080A201 | Confidential | Doc No D-17.304 |
| 15 May 2017 nage 8/110 | | |

| PD | Protocol deviation |
|-------|------------------------------------------------|
| PK | Pharmacokinetic |
| PPS | Per-Protocol Set |
| PR | Pulse rate |
| RIS | Run-in Set |
| RND | All Randomized Set |
| SAE | Serious adverse event |
| SAF | Safety Analysis Set |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analysis Software |
| SB | Single-blind |
| SBP | Systolic blood pressure |
| SCR | Screened Set |
| SD | Standard deviation |
| SiDBP | (Mean trough) sitting diastolic blood pressure |
| SiSBP | (Mean trough) sitting systolic blood pressure |
| SOC | System organ class |
| UACR | Urine albumin-to-creatinine ratio |
| ULN | Upper limit of normal |
| WD | Withdrawal |
| WHO | World Health Organization |

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) describes the statistical analyses and data presentation for the Clinical Study Report of Study AC-080A201, the Phase 2 dose-finding trial with ACT-132577 in subjects with essential hypertension (grade 1 and 2).

This SAP is based on Version 3 of the protocol dated 30 May 2016 [D-16.063].

For the layouts of the tables Biostatistics Standards for Analysis Datasets and Outputs (Project Code: PR 070; version 3.0) will be used.

#### 2 STUDY DESIGN AND FLOW

#### 2.1 Study design

Study AC-080A201 is a prospective, multi-center, double-blind, double-dummy, randomized, placebo- and active-reference, parallel group, Phase 2 dose-finding study with ACT-132577 in subjects with essential hypertension (grade 1 and 2).

Approximately 1000 subjects are enrolled into the study, in order to have at least 540 subjects randomized in the 6 following groups using a 1:1:1:1:1:1 ratio: placebo, 5 mg ACT-132577, 10 mg ACT-132577, 25 mg ACT-132577, 50 mg ACT-132577 and lisinopril 20 mg. At least 420 subjects are expected to complete the trial. There are no stratification factors

The study consists of the following study periods:

#### Screening

The screening period starts with the signature of the "study" informed consent form and lasts until Visit 1. During this period study assessments (e.g., laboratory test) are performed to determine whether the subject is eligible for the study.

#### Run-in period (Period I)

Period I is a single-blind (SB) placebo period of 4 to 6 weeks starting at Visit 1 and ends at Visit 4 / Randomization (after completion of the baseline 24-hour ambulatory blood pressure monitoring [ABPM] recording on the last dose of SB study treatment [placebo]).

The run-in period lasts 4 weeks for anti-hypertensive treatment naïve subjects.

The run-in period lasts 6 weeks for subjects on anti-hypertensive treatment including a 2-week wash-out period for anti-hypertensive treatment. The anti-hypertensive treatment must be discontinued (according to its label) at Visit 1, if there is no contraindication to stop it.

#### **Treatment period (Period II)**

Period II is a double-blind (DB) treatment period of 8 weeks which starts at Visit 4 with the first dose of DB study treatment and ends at Visit 7 at the first dose of SB withdrawal treatment.

# Withdrawal period (Period III)

Period III is a SB placebo period of 2 weeks, which starts at Visit 7 with the first administration of first placebo dose (withdrawal [WD] study treatment) and ends at Visit 8 (WD-End-of-Treatment [EOT]).

# Follow-up period

The follow-up period, including follow-up telephone call, or follow-up visit only for women of childbearing potential to perform the pregnancy test at the site, starts after the last dose of SB WD study treatment (placebo) and ends at 30–33 days after the last dose of the DB treatment.

# **End-of-Study (EOS)**

End-of-Study (EOS) for a single subject is defined as the date of the follow-up telephone call or follow-up visit.

If a subject withdraws consent and does not wish to participate in the study visits, the date of consent withdrawal is EOS for this subject. If a subject is declared lost to follow-up date of last contact is EOS for this subject.

In addition, unscheduled visits may take place at any time during the study, in which case appropriate assessments may be performed at the discretion of the investigator and must be recorded in the electronic Case Report Form (eCRF).

At the end of the study, the investigator/delegate will explain to the subject what treatment(s) / medical care is necessary and available according to local regulations.

#### 2.2 Study visit and assessment schedule

Table 1 shows a schematic representation of the assessments during the study.

Table 1 Visit and assessment schedule

| PERIODS | Name / duration | Period | I: Run-in / | 4–6 weeks | 6 | Period II: Double-blind / 8 weeks Period III: withdrawal / 2 weeks | | | | | Premature<br>EOT | | Follow-up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISITS | Number<br>Name | 1 <sup>6</sup><br>Week –6 | 2 <sup>6</sup><br>Week –4 | 3<br>Week −1 | 4 | ļ | 5<br>Week 2 | 6<br>Week 4 | Wee | 7<br>ek 8 | 8<br>Week 10 | 9 | U1, 2, 3, etc. <sup>10</sup> | Telephone call <sup>9</sup> or visit <sup>11</sup> |
| | Name | Screening** | | | Randon | nization | | | DB- | EOT | WD-EOT | Within 7 days | Unscheduled | EOS |
| | TIME / Week | Day -42 | Day -28<br>(± 3 d) | Day -7<br>(± 4 d) | Pre-<br>Day –1 | Day 1 | 2<br>Day 14<br>(± 3 d) | 4<br>Day 28<br>(± 3 d) | Part 1 Day 55 (± 5 d) | Part 2<br>Day 56 | 10<br>Day 70<br>(± 3 d) | after last study<br>treatment<br>intake | Any time | 30–33 d after last<br>dose of DB treatment |
| Infor | med consent | X | | | | | | | | | | | | |
| F | Eligibility | X | X | X | X | | | | | | | | | |
| Med | dical history | X | | | | | | | | | | | | |
| Physic | al examination | X | X | X | X | | X | X | X | | X | X | X | |
| Concomi | itant medications | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HR*, bod | ly weight, height <sup>1</sup> | X | X | X | X | | X | X | X | | X | X | X | |
| 12- | lead ECG* | $X^4$ | | | $X^9$ | | | X | X | | X | $X^9$ | X | |
| Laboratory in | ncl. pregnancy tests*2 | $X^5$ | | X <sup>9</sup> | $X^9$ | | X | X | X | | X | $X^9$ | X | X <sup>2</sup> |
| U | Jrinalysis | | X <sup>7, 9</sup> | | $X^9$ | | X | X | X | | X | $X^9$ | X | |
| Office B | P measurement* | X | X | X | X | | X | X | X | | X | X | X | |
| Home | e BP device <sup>12</sup> | X | | | | | | | | | | | <b></b> | |
| Ambulatory | BP measurement* | | | | X | | | | X | | | | | |
| PK and PD sampling <sup>13</sup> | | | | | | | X | X | X | | | | | |
| Compliance with study treatment | | | X <sup>9</sup> | X <sup>9</sup> | X | | X | X | X | | X | X | X | |
| Study treatment dispensing/return | | X | $X^8$ | | X | X | | X | X | X | X | X | X | |
| Adv | erse events <sup>3</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serious | adverse events <sup>3</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |

15 May 2017, page 12/110

- \*Electronically transferred to sponsor.
- \*\* Visit 1 (Screening) can last up to 72 h for obtaining informed consent and performing required assessments.
- 1. Height is only measured at Visit 1.
- 2. Serum pregnancy test only for women of childbearing potential. Result is transferred electronically to sponsor.
- 3. All AEs and SAEs that occur after signing the Informed Consent Form and up to 30 days after last DB study treatment intake must be reported.
- 4. Historical ECG is accepted if not older than 6 months.
- 5. Historical blood laboratory data is accepted to check exclusion criterion 15, if not older than 3 months. In such a case, for women of childbearing potential a urine pregnancy test must be performed. If no historical report is available, a blood sample to be taken for laboratory analysis (including pregnancy test for women of childbearing potential) by central laboratory.
- 6. Run-in period is 4 weeks before randomization for anti-hypertensive treatment naïve subjects. Visit 1 is combined with Visit 2. Run-in period is 6 weeks before randomization for subjects on anti-hypertensive treatment. Visit 1 and Visit 2 must be performed.
- 7. Only urine pregnancy test for women of childbearing potential. Result is captured in the eCRF.
- 8. Only for subjects who were on anti-hypertensive drugs at Visit 1 (i.e., had to perform a Visit 2).
- 9. If subject discontinued study treatment during run-in period (i.e., between run-in visits) or at an in-person run-in visit (e.g., Visit 3), these tests may not be performed
- 10. Unscheduled visits may be performed at any time during the study and may include all or some of the indicated assessments, based on the judgment of the investigator.
- 11. For women of childbearing potential a visit must be organized instead of the telephone call to perform the serum pregnancy test at the site. However, if a woman of childbearing potential discontinued study treatment during the run-in period, a telephone call can be made instead of the visit.
- 12. Upon investigator's judgment, a home monitoring device will be dispensed to monitor BP at home, if necessary.
- 13. Sample to be taken at trough (i.e., prior to study treatment intake).

AE = adverse event; BP = blood pressure; DB = double-blind; ECG = electrocardiogram; eCRF = electronic Case Report Form; EOS = End-of-Study; EOT = End-of-Treatment; HR = heart rate; PD = pharmacodynamics; PK = pharmacokinetics; SAE = serious adverse event; WD = withdrawal.

#### 3 OBJECTIVES

# 3.1 Primary objective(s)

The primary objective of the study is to explore the dose-response of ACT-132577 on diastolic blood pressure (DBP) in subjects with grade 1 or 2 essential hypertension.


# 3.2 Secondary objectives

- Evaluate the dose-response of ACT-132577 on:
  - Systolic blood pressure (SBP)
  - Control and response rate of blood pressure (BP)
  - 24-h ABPM.
- Evaluate the safety and tolerability of a once a day (o.d.) oral regimen of 4 doses of ACT-132577.

# 3.3 Other objectives

- Evaluate steady-state trough plasma concentrations of ACT-132577 in hypertensive subjects.
  - Evaluate steady-state trough endothelin (ET)-1 in hypertensive subjects.
- Investigate the correlation between ET-1 and ACT-132577 plasma concentrations.

# 4 CHANGES OR CLARIFICATIONS TO ANALYSES PLANNED IN THE STUDY PROTOCOL

# 4.1 Changes to the analyses planned in the study protocol

#### 4.1.1 Analysis sets

In addition to the analysis sets described in the section 11.1 of the protocol a 'Run-in Set' (RIS) and an 'All Randomized Set' (RND) are defined to be used in summaries of disposition and premature study discontinuation [see Section 7.1.2 and Section 7.1.3].

# 4.1.2 Analyses of the secondary efficacy variables

Where indicated, analyses based on analysis of covariance (ANCOVA) models, mixed models or logistic regression models planned in the protocol for the secondary variables, were supplemented by a Multiple Comparison Procedure – Modeling (MCP-Mod) analysis of the Least Squares Means (LSMeans) obtained from these models. MCP-Mod was qualified as an efficient statistical methodology for model-based design and analysis of Phase 2 dose finding studies [EMA 2014]. This approach replaces the Dunnett tests that were planned in the protocol for these endpoints.

In addition, a dose-response analysis was performed for the average change from baseline over time (Weeks 2, 4 and 8).

*BP control rates.* After completion of the protocol, the Canadian Hypertension Education Program (CHEP) issued guidelines proposing cut-offs of 85 mmHg for DBP and 135 mmHg for SBP, specifically focusing on measurement by automated office blood pressure measurement (OBPM) [Leung 2016]. These were added to the secondary endpoints.

Analysis data set for ABPM. ABPM is performed over a 24-h period with the ABPM device set to record DBP and SBP at a pre-defined inflation sequence over the 24-h period including three measurements per hour during the day and two per hour during the night. ABPM data are electronically transferred to and subsequently to Actelion. The supplements each ABPM reading with an indicator of whether the reading satisfied the quality control criteria agreed

- 1. Start time of ABPM is between 06:00 and 11:00
- 2. Duration of ABPM is at least 24 hours
- 3. Percentage of valid readings in the period of duration is at least 75%
- 4. Number of required hours (i.e., hours with at least one reading) is at least 22
- 5. Number of exception hours (i.e., hours without a reading) is at most 2
- 6. No two consecutive exception hours

It should be noted that when an ABPM reading does not satisfy all 6 criteria this does not necessarily mean that this reading should be excluded from the analysis, as the ABPM analysis primarily focuses on the 24 hour means (according to report dated For the analysis of 24 hour means, criteria 3 and 6 are considered to be the most relevant ones by Actelion.

For this reason, the ABPM analyses will be based on the subset of subjects from the Per-Protocol Set (PPS) with baseline and Week 8 ABPM readings satisfying quality criteria 3 and 6 (i.e., ABPM readings having less than 75% valid readings and/or two consecutive exception hours will be excluded).

Trough to peak ratios based on ABPM. In the protocol it was assumed that trough to peak ratios of DBP and SBP measured by ABPM would be derived on a subject level. However, the definition of subject-specific trough to peak ratios [Omboni 1995] appears to be problematic because of individual ABPM variation over time. Based on clinical rationale and following the reasoning in recent FDA reviews such as FDA 2007, the trough to peak ratios of DBP (and SBP) were re-defined on a treatment group level based on the time course of the 24 hours ABPM. As a consequence, the analysis in the protocol (which assumed a definition on a subject level) was replaced by descriptive statistics [Section 10.7].

#### 4.1.3 Safety analysis

As exploratory analyses, the change from baseline to Week 8 in hemoglobin and weight will be analyzed using the MCP-Mod approach [see Sections 10.9.4 and 10.9.5] to explore whether there is a dose-response relationship for these variables which are associated with the safety of ACT-132577.

# 4.2 Changes in the conduct of the study / data collection

A blinded sample size re-estimation was introduced in Version 3 of the protocol. This sample size re-estimation was based on the standard deviation (SD) of the primary endpoint, change from baseline to Week 8 in DBP as measured by OBPM in the PPS. As a consequence the number of randomized subjects was lowered to 490 (instead of the foreseen 540). The lower sample size did not affect the conduct of the study or the analysis of the data.

After database lock but before unblinding, it was noticed that one subject who had a Week 8 sitting diastolic blood pressure (SiDBP) outside of the analysis window was, however, included in the PPS (after accounting for the protocol deviations [PDs] present in the database). The decision was taken by management not to unlock the database and to maintain the PPS as it was. The subject remained in the PPS, with a missing value for the Week 8 SiDBP.

#### 5 DEFINITIONS OF VARIABLES

**Baseline** assessments refer to the last available measurement before the start of double-blind treatment.

If date and time of the measurement are collected, baseline is the last one up to the start date and time of the double-blind treatment. If only the date is collected, baseline is the last one before the start date of the double-blind treatment. For ABPM baseline is the period from date/time of last run-in placebo intake up to the date/time of the first double-blind treatment intake, i.e., a maximum of 25 hours.

**Screening** assessments refer to last available measurement before or on run-in start date (Visit 1) before the start of placebo run-in medication.

# 5.1 Subjects disposition

Screened subjects: are all subjects who received a subject number.

<u>Screening failures</u>: are all subjects with answer 'NO' to the question 'Is the subject eligible for the Run-in period?' in the **Eligibility - Run-in Period** eCRF).

Reason for screening failure is collected in the same eCRF form.

Subjects who failed screening twice will only be counted once (and only the reason for the last screening failure will be tabulated).

<u>Subjects in Run-in</u>: are all subjects with answer 'YES' to the question 'Is the subject eligible for the Run-in period?' in the **Eligibility - Run-in Period** eCRF.

<u>Run-in failures</u>: are all subjects in Run-in with answer 'NO' to the question 'Was the subject randomized?' in the **Randomization** eCRF. Reason for run-in failure is collected in the same eCRF form.

<u>Randomized subjects</u>: are all subjects who received a randomization number from the Interactive Voice Response System (IVRS).

# 5.2 Subject characteristics

# **5.2.1** Demographics

Demographic variables are those collected at Screening on the **Demographics** eCRF pages 12–13 (or on page 14 in the event of Re-Screening):

- Sex
- Age
- Race (Black or African American; American Indian or Alaska Native; Native Hawaiian or Other Pacific Islander; Asian; White; Other)
- Ethnicity
- Country (derived from site number)

#### **5.2.2** Baseline disease characteristics

Baseline disease characteristics include:

- Duration of essential hypertension (years) at Screening [see Section 11.8 for definition]
- Treatment for hypertension ongoing at Screening (Y/N), as collected in the **Treatment of Hypertension Summary** eCRF.
- Mean trough sitting diastolic blood pressure (SiDBP) at Screening as measured by ORPM
- Mean trough sitting systolic blood pressure (SiSBP) at Screening as measured by OBPM

#### 5.2.3 Other baseline characteristics

Other baseline characteristics, recorded on the **Height, Body Weight & BMI** eCRF page 22, at Screening and/or Re-Screening include:

- Height (cm) at Screening
- Body weight (kg) at Screening
- Body Mass Index (BMI; kg/m<sup>2</sup>) at Screening

When necessary, height and body weight are converted into cm and kg, respectively [according to conversion rules detailed in Section 11.9]. BMI (kg/m²), derived according to the formula in Section 11.10, is collected in the eCRF and will not be (re-) calculated.

In the event of re-screening, the last available measurement has to be considered in the analysis.

# 5.2.4 Medical history

Medical history includes previous and/or concomitant diseases or diagnoses collected on the **Medical History** eCRF page 15. Reported terms are coded using the MedDRA dictionary, Version 19.0.

Any disease or diagnosis is defined as previous if 'Ongoing at Screening' is not answered with 'Yes'; all other diseases/diagnoses are considered as concomitant.

# 5.2.5 Previous and concomitant therapies

Therapies are collected in the **Previous/Concomitant Medication** eCRF, and terms are coded using the WHO drug code dictionary and the anatomic therapeutic chemical (ATC) class code using the versions available at database lock

A <u>previous</u> therapy is any treatment for which the end date is prior to the start of study (i.e., signing of informed consent). If the end date is missing and the start date of therapy is prior to the date of informed consent, then the therapy is considered as previous if 'Ongoing at start of treatment?' is not ticked with 'Yes'.

A <u>study-concomitant</u> therapy is any treatment that is ongoing or initiated after signing of informed consent, or initiated up to 30 days after the DB study treatment discontinuation (Visit 8).

A <u>double-blind treatment concomitant</u> therapy is any treatment that is either ongoing at the start of DB study treatment (i.e., Day 1 – Visit 4 / Randomization) or is initiated during the DB treatment period.

Rules for handling partial or missing dates are detailed in Section 12.

#### Forbidden concomitant therapies

The following concomitant therapies are forbidden from Screening Visit (i.e., Visit 1) until the WD-EOT Visit (i.e., Visit 8):

• Any drug which may affect BP e.g., ophthalmic preparation, sympathomimetics (any formulation of decongestants), corticosteroids (intermittent use of topical/nasal applications excluded), cyclosporin, tacrolimus, erythropoietin, diet pills, herbal supplements, homeopathic compounds, treatment for psychiatric diseases [see protocol synopsis Appendix A].

- Endothelin receptor antagonists, and phosphodiesterase type-5 inhibitors.
- Strong inhibitors or inducers of cytochrome P450 3A4 isoenzyme [see protocol synopsis Appendix A].

These definitions will be used in the clinical review to identify potential PDs. Forbidden medication will not be tabulated as such.

### **Specific previous and concomitant therapies**

Not applicable.

# 5.2.6 Other subject characteristics

Not applicable.

# 5.3 Study treatment duration and compliance

# **5.3.1** Study treatment duration

Double-blind treatment duration is defined as the number of days between the first dose of double-blind study treatment [see definition in Section 11.2] and the last dose of double-blind study treatment [see definition in Section 11.4] plus one day, without taking into account interruptions. For the purpose of tabulation treatment duration will also be expressed in weeks, calculated by dividing the above treatment duration (in days) by 7.

In addition, run-in treatment duration is defined as the number of days between the first dose and last dose of open-label placebo run-in treatment.

# **5.3.2** Compliance with study treatment

Double-blind treatment compliance is based on the **Study Drug Dispensing & Accountability** eCRF. Run-in treatment compliance is based on the same eCRF.

As per section 5.1.4.2 of the protocol, all subjects had to take 2 capsules o.d. every morning from the morning of Visit 4 / Randomization (i.e., Day 1, after completion of the baseline 24-hour ABPM recording) to the morning of Visit 7 / Part 1.

Compliance between Visit 4 and Visit 7 / Part 1 will be then calculated as follows:

#### Compliance =

[(number of capsules dispensed at Visit 4 – number of capsules returned at Visit 6 + number of capsules dispensed at Visit 6 – number of capsules returned at Visit 7)/ (Total number of capsules that should have been taken)] × 100.

The number of capsules that should have been taken during the double-blind period is the double-blind treatment duration (in days) as defined in Section 5.3.1, multiplied by 2.

Run-in compliance between Visit 1 and Visit 4 / Part 1 will be calculated similarly.

Here the expected number of capsules is the run-in treatment duration (in days) as defined in Section 5.3.1, multiplied by 2.

#### **5.3.3** Study treatment discontinuation

A subject is considered to have prematurely discontinued double-blind study treatment if the 'reason for treatment end' in the **Study drug Log** eCRF is 'PREMATURE DISCONTINUATION' and the 'Study Period' is 'DB TREATMENT'. The reason for premature discontinuation will be taken from the **Premature Discontinuation of Study Treatment** eCRF and the study period is 'DB TREATMENT'.

Discontinuation from run-in study treatment is defined similarly and the reason will be taken from the same eCRF, but with study period = 'RUN-IN TREATMENT'. Discontinuation from withdrawal study treatment (listed only) is defined similarly with study period = 'SB WITHDRAWAL'. In those cases where a subject completed the double-blind treatment period, but did not start the withdrawal period, the reason for treatment discontinuation will be allocated to the withdrawal period.

# 5.3.4 Study treatment adjustments or interruptions

Study treatment interruptions in the double-blind period are recorded in the **Study drug Log** when 'Study Period' is 'DB TREATMENT'. A subject is considered to have had a study treatment interruption if the reason for treatment end is either 'Temporarily interrupted due to an AE' or 'Temporarily interrupted not due to an AE'.

# 5.4 Study discontinuation

Subjects who completed the study as per protocol are those with the question "Did the subject complete the study?" answered "Yes" in the **End-of-Study** eCRF.

On the other hand, a subject is considered to have prematurely discontinued the study if the answer to the question 'Did the subject complete the study?' in the **End-of-Study** eCRF is 'No'. The reason for study stop is derived from the same form. Reasons for study withdrawal are: Death, Lost to follow up, Subject decision, Physician decision, Sponsor decision.

# 5.5 Efficacy variables

All efficacy data are collected electronically and are transferred to Actelion by



OBPM, SiDBP and SiSBP (mmHg) are measured at the study site by the BpTRU<sup>®</sup> device using six measurements per subject / visit. These measurements and their average (excluding the first measurement) are uploaded into the database. The data

transfer from to Actelion includes the separate measurements as well as the average which will be used as the subject's SiDBP or SiSBP value for that visit. The average will not be re-calculated by the sponsor. The sponsor will perform spot checks to confirm that the average was been correctly calculated

ABPM is performed over a 24-h period with the ABPM device set to record DBP and SBP at a pre-defined inflation sequence over the 24-h period including three measurements per hour during the day and two per hour during the night. ABPM data are electronically transferred to and subsequently to Actelion. The supplements each ABPM reading with an indicator of whether the reading satisfied the quality control criteria agreed between and Actelion

- 1. Start time of ABPM is between 06:00 and 11:00
- 2. Duration of ABPM is at least 24 hours
- 3. Percentage of valid readings in the period of duration is at least 75%
- 4. Number of required hours (i.e., hours with at least one reading) is at least 22
- 5. Number of exception hours (i.e., hours without a reading) is at most 2
- 6. No two consecutive exception hours

In addition, there is an indicator (Y/N) for the overall quality of the ABPM reading. This is only set to Y if all six criteria are met.

It should be noted that when an ABPM reading does not satisfy all 6 criteria, this does not necessarily mean that this reading should be excluded from the analysis as the ABPM analysis primarily focuses on the 24 hour means

For the analysis of 24 hour means, criteria 3 and 6 are considered to be the most relevant ones by Actelion.

For this reason, the ABPM analyses will be based on the subset of subjects from the PPS with baseline and Week 8 ABPM readings satisfying quality criteria 3 and 6 (i.e., ABPM readings having less than 75% valid readings and/or two consecutive exception hours will be excluded). As this subset is likely to be comprised of < 50% of subjects, formal dose-response analyses for the ABPM endpoints will be carried out as needed.

All assessments (including the unscheduled ones) are considered and re-assigned to the most appropriate visit according to the time windows described in Section 11; reference to visits are to be intended as references to re-mapped visit, i.e., time window visits.

#### 5.5.1 Primary efficacy endpoint(s)

The primary efficacy endpoint is the change from baseline to Week 8 of DB treatment period (Period II) in mean trough (i.e., 24 hours post-dose) SiDBP, measured by OBPM.

Baseline is defined as described in Section 5. Week 8 is the time window of Visit 7 [Section 11.1].

SiDBP is retrieved from the SDTM VS domain selecting VSTESTCD="DIABP" and VSSCAT = 'Average'.

# 5.5.2 Secondary efficacy endpoints

- Change from baseline to Week 8 of DB treatment period (Period II) in mean trough SiSBP, measured by OBPM and collected as described for SiDBP.
  - SiSBP is retrieved from the SDTM VS domain selecting VSTESTCD="SYSBP" and VSSCAT = "Average".
- Control and response status at Week 8 of DB treatment period (Period II) based on trough SiDBP, measured by OBPM;
  - Controlled, if mean SiDBP < 90 mmHg;</li>
  - Responder, if the reduction from baseline in mean SiDBP ≥ 10 mmHg;
  - Controlled according to CHEP guidelines [Leung 2016], if mean SiDBP < 85 mmHg.</li>
- Control and response status at Week 8 of DB treatment period (Period II) based on trough SiSBP, measured by OBPM;
  - Controlled, if mean SiSBP < 140 mmHg;
  - Responder, if the reduction from baseline in mean SiSBP  $\geq$  20 mmHg;
  - Controlled according to CHEP guidelines [Leung 2016], if mean SiSBP < 135 mmHg.</li>
- Change from baseline to Week 8 of DB treatment period (Period II) in 24-hour mean DBP, measured by ABPM;
  - ABPM will be measured before start of treatment (Day -1, Visit 4) and after the last dose (Day 55, Visit 7). At each visit the 24-hour mean DBP will be derived from the area under the DBP-time curve, divided by the time span. [See Figure 1 for clarification.] Time points later than 25 hours after the first time point will be excluded from the calculation. The change from baseline to Week 8 will be obtained as the difference in 24-hour mean DBP ABPM between Visit 7 and Visit 1.
- Change from baseline to Week 8 of DB treatment period (Period II) in 24-hour mean SBP, measured by ABPM;
  - The change from baseline to Week 8 will be obtained as the difference in 24-hour mean SBP ABPM between Visit 7 and Visit 1, where the 24-hour mean SBP ABPM is calculated similar to the 24-hour mean DBP ABPM.

- Trough to peak ratio for DBP based on ABPM.
  - The trough to peak ratio will be derived on treatment group level [FDA 2007] based on the time course of ABPM and will be corrected for baseline according to the following steps:
    - O Patient level: for each visit (Visit 4 / Day -1 and Visit 7 / Part 1) the patient's ABPM-DBP will be averaged by hour after drug intake (0, 1, ..., 24), applying a window of 30 minutes around each hour (lower limit excluded; upper limit included).
    - O Group level: for each visit (Visit 4 / Day -1 and Visit 7 / Part 1) and hour after drug intake (0, 1, ..., 24) the ABPM-DBP will be averaged by treatment group.
    - o Group level: for each hour after drug intake (0, 1, ..., 24) and the treatment group the difference in mean ABPM-DBP between Week 8 (Visit 7 Part 1) and baseline (Visit 4 Part 1) will be obtained.
    - o Group level: the trough to peak ratio will be calculated as the average of the (five) differences at hours 20–24 (expected trough) divided by the average of the (five) differences at hours 2–6 (expected peak at 4 hours ± 2 hours) [See Appendix C for illustration.]

Baseline is defined as described in Section 5 and Week 8 is the time window of Visit 7 [Section 11.1].

In the evaluation of changes from baseline and control/response status, only subjects with both the baseline and the time point assessments available will be included.

# 5.5.3 Other efficacy endpoints

- Changes from baseline to time window Visit 5 (Week 2) and time window Visit 6 (Week 4) of DB treatment period (Period II) in mean trough SiSBP and SiDBP (measured by OBPM);
- Change from baseline to Week 8 of DB treatment period (Period II) in mean daytime ABPM;
  - Change from baseline in mean daytime DBP. All ABPM measurements taken between 09:00 and 21:00 will be included in this calculation [O'Brien 2013]; there may be two parts of the daytime DBP-time curve to be considered for a subject at a given visit, one for each calendar day of Visits 4 and 7. At each visit the mean daytime DBP will be derived from the area under the DBP-time curve(s), divided by the time span(s) [see Appendix B for clarification]. The change from baseline to Week 8 will be obtained as the difference in mean daytime DBP ABPM between Visit 7 and Visit 4.
  - Change from baseline in mean daytime SBP. Similar to change from baseline in mean daytime DBP.

- Change from baseline to Week 8 of DB treatment period (Period II) in mean night time ABPM;
  - Change from baseline in mean night time DBP. All ABPM measurements taken between 01:00 and 06:00 will be included in this calculation [O'Brien 2013]; there should be one night time part of the DBP-time curve to be considered for each subject at a given visit; in the unlikely event that there are two, only the first one will be used). At each visit the mean night time DBP will be derived from the area under the DBP-time curve, divided by the time span [see Appendix B for further specification]. The change from baseline to Week 8 will be obtained as the difference in mean daytime DBP ABPM between Visit 7 and Visit 4.
  - Change from baseline in mean night time SBP. Similar to change from baseline in mean night time DBP.
- Trough to peak ratio for SBP based on ABPM;
  - The trough to peak ratio for SBP will be derived on treatment group level based on the time course of ABPM as similar to the trough to peak ratio for DBP.
- Changes from baseline to time window Visit 8 (Week 10 i.e., Week 2 of withdrawal period Period III) in mean trough SiSBP and SiDBP (measured by OBPM);
- Changes from Week 8 of Period II to time window Visit 8 (Week 10 i.e., Week 2 of withdrawal period Period III) in mean trough SiSBP and SiDBP (measured by OBPM).

# 5.5.3.1 Illustration of derivation of ABPM endpoints

The derivation of the various endpoints based on ABPM is illustrated by means of an example. Figure 1 displays the DBP and SBP measured by ABPM in one subject at one visit. The data underlying this example figure are included in Appendix B.

Since ABPM measurements are obtained during 24 hours at two consecutive calendar days, the time on the horizontal axis runs from 0–48 hours, clock times 0:00–23:59 corresponding to the first day and times 24:00–48:00 to the second day The ABPM started on 10:29 on the first day and finished on 11:04 on the second day [35:04 in Appendix B].

Figure 1 Example DBP and SBP measured by ABPM



Example DBP (blue lines) and SBP (red lines) measured by ABPM in one subject at one visit. Vertical lines indicate inclusion of measurements in the calculation of daytime ABPM (solid) and night time ABPM (dotted).

The derivation of the 24-hour mean DBP (SBP), mean daytime DBP (SBP) and mean night time DBP (SBP) for these example data are as follows.

- The total duration of this ABPM (24 hours 35 minutes) was greater than 24 hours, but less than 25 hours, so all measurements were included in the calculation of 24-hours mean ABPM.
- The 24-hour mean DBP (SBP) is derived from the area under the DBP (SBP) curve, divided by the time span. The area under the curve is calculated by the trapezoidal rule. The implementation of this rule in SAS is given in Appendix B. For the example data the areas under the DBP and SBP curves are 8,640,870 and 12,956,970 mmHg sec, respectively. Dividing both areas by the time span of

88,500 sec gives a 24-hour means of 97.6 and 146.4 mmHg for DBP and SBP, respectively.

- The trapezoidal rule will be applied up to the last measurement within 25 hours. If there is another measurement after 25 hours, there will be NO interpolation up to 25 hours exactly.
- The mean daytime DBP (SBP) is based on two periods: from 10:29 to 21:00 (limits included) on the first day and from 09:00 to 11:04 on the second day (limits included; 33:00 to 35:04 in Appendix B). The mean daytime DBP and SBP are 99.5 mmHg and 143.9 mmHg, respectively.
- The mean night time DBP (SBP) is based on the measurements between 01:00 and 06:00 on the second day (limits included; 25:00 to 30:00 in Appendix B). The mean night time DBP and SBP are 78.4 mmHg and 135.5 mmHg, respectively.
- Note that measurements between 21:00 on the first day and 01:00 on the second day (limits excluded) and between 06:00 and 09:00 on the second day (limits excluded) are only included in the calculation of the 24-hour means, but not in the calculation of the daytime or night time means.

# 5.6 Safety variables

All assessments are considered and re-assigned to the most appropriate visit according to the time windows described in Section 11; reference to visits are to be intended as references to re-mapped visit, i.e., time window visits.

The following safety variables will be evaluated:

- Treatment-emergent adverse events (AEs);
- AEs leading to premature discontinuation of study treatment;
- Treatment-emergent deaths;
- Treatment-emergent serious adverse events (SAEs);
- Treatment-emergent electrocardiogram (ECG) abnormalities;
- Treatment-emergent marked laboratory abnormalities;
- Changes from baseline to time window Visits 5, 6 and 7 (Weeks 2, 4 and 8, respectively) of DB treatment period (Period II) in laboratory parameters;
- Changes from baseline to time window Visits 6 and 7 (Week 4 and Week 8, respectively) of DB treatment period (Period II) in ECG parameters (pulse rate [PR], QRS, QT, QTcB, QTcF);
- Changes from baseline to time window Visits 5, 6 and 7 (Weeks 2, 4 and 8, respectively) of DB treatment period (Period II) in body weight and PR (BpTRU®).

#### **5.6.1** Adverse events

An AE is defined as any term reported by the investigator in the **Adverse Event** eCRF. The original terms used by the investigators to describe AEs are assigned preferred terms for classification and tabulation using the MedDRA dictionary, Version 19.0.

#### 5.6.1.1 Treatment-emergent adverse events

Double-blind treatment-emergent AEs are defined as those AEs with onset on or after the double-blind treatment start date [see definition in Section 11.2] up to the double-blind treatment end date [see definition in Section 11.4] plus 30 days (included). Run-in treatment-emergent AEs are AEs with onset dates between the start and end dates of the run-in placebo (or the start of double-blind treatment, if applicable; limits included).

# 5.6.1.2 Frequency of treatment-emergent adverse events

Except otherwise specified, the counting of treatment-emergent AEs in the summary table is handled as follows:

- Subjects who experienced the same AE more than once (as qualified by the same preferred term[s]) are counted only once.
- In the event that the reported AE is assigned to several preferred terms, subjects are counted for each individual preferred term.

#### 5.6.1.3 Intensity of treatment-emergent adverse events

The intensity of an AE is determined by the investigator as 'mild', 'moderate' or 'severe'.

AEs reported more than once (as qualified by the same preferred term) for a subject within a specified time period but with different intensities are counted only once, with the worst reported intensity in the corresponding analysis. If intensity is missing, the event is considered severe.

# 5.6.1.4 Relationship of treatment-emergent adverse events

Relationship to study treatment is determined by the investigator as 'related' or 'not related'. An event is considered related if the response to the question 'Relationship to study treatment?' is answered 'Related'.

For AEs reported more than once (as qualified by the same preferred term) for a subject within a specified time period, the worst relationship reported is taken. AEs with missing relationship are considered in any analysis as 'Related'.

#### **5.6.2** Deaths

Death information is taken from the **Death** eCRF. The primary cause of death is reported on the same form.

The original terms used by the investigators to describe the primary death cause are assigned preferred terms for classification and tabulation using the MedDRA dictionary.

Double-blind treatment-emergent deaths are those with occurrence on or after the double-blind treatment start date [see definition in Section 11.2] up to the double-blind treatment end date [see definition in Section 11.4] plus 30 days (included). Run-in

treatment-emergent deaths are deaths that occur between the start and end of the run-in placebo (or the start of double-blind treatment, if applicable; limits included).

#### **5.6.3** Serious adverse events

An SAE is defined as an AE with "Serious?" = "Yes" on the **Adverse Events** eCRF.

Double-blind treatment-emergent SAEs are all SAEs with onset on or after the double-blind treatment start date [see definition in Section 11.2] up to the double-blind treatment end date [see definition in Section 11.4] plus 30 days (included). Run-in treatment-emergent SAEs are SAEs with onset date between the start and end dates of the run-in placebo (or the start of double-blind treatment, if applicable; limits included).

#### 5.6.4 Adverse events leading to discontinuation of study treatment

These are AEs with 'Action taken with study drug' recorded as 'permanently discontinued' on the **Adverse Event** eCRF.

#### 5.6.5 Other adverse events

Not applicable.

# 5.6.6 Physical examination, vital signs and body weight

Vital signs include PR measured by BpTRU<sup>®</sup> (simultaneously with BP; the mean is provided in the same way, i.e., based on the last 5 of 6 measurements) and body weight (DBP and SBP are evaluated as efficacy endpoints). For PR, the value is retrieved from the SDTM VS domain by selecting VSTESTCD = "HR" and VSSCAT = 'Average'.

All assessments (including the unscheduled ones) are considered and re-assigned to the most appropriate visit according to the time windows described in Section 12.

#### 5.6.7 Electrocardiogram

A standard 12-lead ECG is performed as defined in the Schedule of Assessments. Historical ECG is accepted for Visit 1, if not older than 6 months. Digital 12-lead ECG devices will be provided to each site by the central ECG laboratory for the duration of the study. All assessments (including the unscheduled ones) are considered and re-assigned to the most appropriate visit according to the rules described in Section 11.1.

The following variables will be evaluated: heart rate (HR; bpm), PR (ms), QRS (ms), QT (ms), QTc (ms). In addition, the percentage of subjects with any ECG findings will be evaluated.

QTc (ms) will be calculated according to Fridericia's formula QTcF =  $QT/(RR)^{1/3}$ .

ECG data will be electronically transferred from the ECG laboratory database to Actelion and will not be (re-)calculated. Note that ECG HR will be evaluated only in the context of the ECG. For vital signs, PR will be used based on BpTRU<sup>®</sup>.

# 5.6.7.1 Treatment-emergent ECG abnormalities

Double-blind treatment-emergent ECG abnormalities are defined as follows:

- QTcF (Fridericia's formula) maximum value > 450 ms (H), > 480 ms (HH), or > 500 ms (HHH);
- Maximum increase from baseline in QTcF (Fridericia's formula) > 30 ms (HH), > 60 ms (HHH).

In addition, each of the six combinations of maximum QTcF and increase in QTcF will be considered.

Note that, in order to allow appropriate interpretation of overall incidence of abnormalities > 450 ms, the marked abnormalities are presented cumulatively, e.g., a QTc value of 501 ms is reported in > 450 ms (H), > 480 ms (HH) and > 500 ms (HHH) categories; the same holds for abnormalities related to changes from baseline (i.e., they are presented cumulatively).

Treatment-emergent ECG abnormalities are defined as those abnormalities with onset on or after the double-blind treatment start date [see definition in Section 11.2] up to the double-blind treatment end date [see definition in Section 11.4] plus 30 days (included): i.e., the highest QTc absolute value and the highest QTc change value at any post-baseline time point of assessment up to 30 days after study treatment discontinuation are considered in the evaluation of the categories, as defined above.

#### 5.6.8 Laboratory

Laboratory data are evaluated in standard international units as provided by the central laboratory. The following tests are considered:

- Hematology: hemoglobin, hematocrit, erythrocyte count, leukocyte count with differential counts, platelet count.
- Chemistry: aminotransferases (aspartate aminotransferase [AST] / alanine aminotransferase [ALT]), alkaline phosphatase [AP], total and direct bilirubin, lactate hehydrogenase, creatinine, creatinine clearance, uric acid, glucose, sodium, potassium, total protein, albumin, thyroid hormones (triiodothyronine [free T3], thyroxine [free T4]) and thyroid-stimulating hormone.
- Urinalysis: Urine albumin-to-creatinine ratio (UACR).

For woman of childbearing potential, urine as well as serum pregnancy tests are performed, but these results will not be summarized as part of the laboratory data. Positive pregnancy tests (if any) will be reported.

Results of local laboratory tests (collected on the **Local Laboratory** eCRF) may be used to identify marked abnormalities, but only if no central laboratory test has been performed in the same time window. Local laboratory test results will not be used in summaries, but will still be listed.

# 5.6.8.1 Treatment-emergent marked laboratory abnormalities

The marked laboratory abnormalities are given in Table 2, copied from appendix 1 of the protocol.

Table 2 Thresholds for marked laboratory abnormalities

| Parameter LL | | LLL | нн | ннн | нннн |
|---|---|---|---|---|---|
| Hematology | | | | | |
| Hemoglobin | < 100 g/L<br>(< 10 g/dL;<br>< 6.2 mmol/L) | < 80<br>(< 8 g/dL;<br>< 4.9 mmol/L;) | Increase in > 20 g/L<br>above ULN or above<br>baseline if baseline is<br>above ULN | Increase in > 40 g/L<br>above ULN or above<br>baseline if baseline is<br>above ULN | |
| Hematocrit | < 28% for females<br>< 32% for males | < 20% | > 60% in men<br>> 55% in women | > 65% | |
| Leukocytes | < 3.0 × 10 <sup>9</sup> /L<br>(< 3000/mm <sup>3</sup> ) | $< 2.0 \times 10^9 / L$<br>( $< 2000 / mm^3$ ) | $> 20.0 \times 10^9 / L$<br>(> 20,000/mm <sup>3</sup> ) | > 100.0 × 10 <sup>9</sup> /L<br>(> 100,000/mm <sup>3</sup> ) | |
| Platelet count | $< 75 \times 10^9 / L$<br>( $< 75,000 / mm^3$ ) | $< 50 \times 10^9/L$<br>( $< 50,000/mm^3$ ) | > 600× 10 <sup>9</sup> /L | > 999× 10 <sup>9</sup> /L | |
| Neutrophils | < 1.5 10 <sup>9</sup> /L<br>(< 1500/mm <sup>3</sup> ) | <1.010 <sup>9</sup> /L<br>(<1000/mm <sup>3</sup> ) | NA | NA | |
| Eosinophils | NA | NA | $> 5.0 \times 10^9 \text{ or}$<br>> 5% ( > 5000 cells/mm <sup>3</sup> ) | NA | |
| Lymphocytes | $< 0.8 \times 10^9 / L$<br>( $< 800 / mm^3$ ) | $< 0.5 \times 10^9 / L$<br>( $< 500 / mm^3$ ) | $> 4.0 \times 10^9 / L$<br>(> 4000/mm <sup>3</sup> ) | $> 20 \times 10^9/L$<br>(> 20,000/mm <sup>3</sup> ) | |

| Parameter LL | | LLL | нн | ннн | нннн |
|---|---|---|---|---|---|
| Blood Chemistry | | | | | |
| AST (U/L) | NA | NA | > 3 × ULN | > 5 × ULN | >8 × ULN |
| ALT (U/L) | NA | NA | > 3 × ULN | > 5 × ULN | > 8 × ULN |
| AP | NA | NA | > 2.5 × ULN | > 5 × ULN | |
| Bilirubin Total (µmol/L) | NA | NA | > 2 × ULN | > 5 × ULN | |
| Creatinine | NA | NA | > 1.5 × ULN or<br>> 1.5 × baseline | > 3 × ULN or<br>> 3 × baseline | |
| Creatinine clearance | < 60 mL/min | < 30 mL/min | NA | NA | |
| Glucose | < 3.0 mmol /L<br>(< 55 mg/dL) | < 2.2 mmol /L<br>(< 40 mg/ dL) | > 8.9 mmol /L<br>(> 160 mg/dL) | > 13.9 mmol /L<br>(> 250 mg/ dL) | |
| Sodium | | < 130 mmol/L<br>(< 130 mEq/L) | > 150 mmol/L<br>(> 150 mEq/L) | > 155 mmol/L<br>(> 155 mEq/L) | |
| Potassium | < 3.2(mmol/L) | < 3.0(mmol/L) | > 5.5(mmol/L) | > 6.0(mmol/L) | |
| Uric acid | NA | NA | > 590 (umol/L)<br>(> 10 mg/dL) | > 720 (umol/L)<br>(> 12 mg/dL) | |
| Albumin | < 30 g/L<br>(< 3.0 g/dL) | < 20(g/L<br>(< 2.0 g/dL) | - | - | |

ALT = alanine aminotransferase; AP = alkaline phosphatase; AST = aspartate aminotransferase; NA = not applicable; ULN = upper limit of normal.

Treatment-emergent marked laboratory abnormalities are those marked abnormalities with onset date after the double-blind treatment start date [see definition in Section 11.2] and before or on double-blind treatment end date [see definition in Section 11.4] plus 30 days (included), that were not present at baseline.

Baseline for laboratory data is defined in Section 5. Each condition is triggered at any post-baseline time point of measurement up to the double-blind treatment end date plus 30 days (included). When determining double-blind treatment-emergent marked laboratory abnormalities, all assessments (including the unscheduled ones) are considered.

# 5.6.9 Other safety variables

Not applicable.

# 5.7 Quality of life variables

Not applicable.

#### 5.8 Pharmacoeconomic variables

Not applicable.

# 5.9 Pharmacodynamic variables

Trough plasma concentrations of ET-1, measured at steady state at Weeks 2, 4 and 8 in DB treatment period (Period II). Trough is defined as a sample taken in the morning of the visit prior to study treatment administration of that visit.

#### 5.10 Pharmacokinetic variables

plasma concentrations of ACT-132577 , measured at steady state at Weeks 2, 4 and 8 in DB treatment period (Period II)

#### 6 DEFINITION OF PROTOCOL DEVIATIONS

PDs include deviations from inclusion and/or exclusion criteria and deviations from the protocol during the conduct of the study, classified as per latest version of PD code list. Each PD is reported in the SDTM DV domain and categorized according to time period:

- 1. PD at Screening
- 2. PD during Run-in period
- 3. PD at Visit 4 / Pre-randomization

- 4. PD during DB treatment period
- 5. PD during withdrawal period and follow-up

Each PD is classified as important or not. Only important PDs during time periods 3, 4 and 5 will be summarized by treatment group for the RND set. (All PDs will be listed.)

Note that an important PD does not necessarily lead to exclusion from the PPS [see Section 7.1.6], whereas an unimportant PD may lead to exclusion from the PPS. The subset of PDs *leading to exclusion* from the PPS are:

- 1. Double-blind treatment duration less than 49 days: PV PP.535.
- 2. No or no valid Week 8 SiDBP (hence, no primary endpoint): PV\_PP.501 and PV MM.501.
- 3. Anti-hypertensive treatment still ongoing at randomization: PV\_MM.307.
- 4. Taking medication during the double-blind treatment interfering with the primary efficacy parameter (SiDBP): PV\_MM.503, PV\_MM.504, PV\_MM.506, PV\_MM.507, PV\_MM.508, PV\_MM.509, PV\_MM.534.
- 5. Compliance with double-blind treatment < 80% or > 120% or treatment not taken as per protocol: PV\_PP.502 and PV\_MM.515.

Note that exclusion will be done on a subject basis (rather than on subject / visit basis). In this particular study this approach is not unreasonable since PDs 1–5 are related to the 8 week DB treatment period and the primary efficacy endpoint is measured at the end of that period.

The one PD *leading to exclusion* from the Pharmacokinetic (PK) Set [see Section 7.1.6] is that the PK sample for that subject/visit was not taken at trough: PV\_MM.512.

#### 7 ANALYSIS SETS

# 7.1 Definitions of analysis sets

#### 7.1.1 Screened Set

The Screened Set (SCR) includes all subjects who received a subject number.

#### 7.1.2 Run-in Set

The RIS includes all subjects who received at least one dose of SB placebo in Period I.

#### 7.1.3 All Randomized Set

The RND includes all subjects who received a randomization number from the IVRS.

#### 7.1.4 Full Analysis Set

The Full Analysis Set (FAS) includes all subjects in the RND Set who have a baseline mean trough SiDBP. Subjects are evaluated according to the study treatment they have been assigned to (which may be different from the study treatment they have received).

#### 7.1.5 Per-Protocol Set

The PPS includes all subjects from the FAS who have a mean trough SiDBP at Week 8 of Period II and do not have any important PD as defined in Section 6. Subjects are evaluated according to the study treatment they have been assigned to.

#### 7.1.6 Safety Set

The Safety Set (SAF) includes all subjects who received at least one dose of study treatment in Period II. Subjects are evaluated according to the study treatment they have received

#### 7.1.7 Pharmacokinetic Set

The PK Set includes all subjects from the PPS who had at least one evaluable PK trough sample. Subjects are evaluated according to the study treatment they have received.

#### 8 DEFINITION OF SUBGROUPS

All subgroup analyses will be performed to investigate the consistency of the treatment across subgroups defined by:

Age  $< 65 \text{ versus} \ge 65 \text{ years}$ 

18-64, 65-84 and  $\geq 85$  years; for European Clinical Trials (EudraCT)

Database purposes only

Sex Female, male

Race Black or African American; American Indian or Alaska Native; Native

Hawaiian or Other Pacific Islander; Asian; White; Other.

Categories containing less than 5% of randomized subjects will be considered

in the category 'Other' for purpose of analysis.

Country United States (including Puerto Rico, USA); Canada (CAN); Israel (ISR)

#### 9 GENERAL STATISTICAL METHODOLOGY

This section describes the general statistical methodology, independent of which analysis data set is used. These aspects will be addressed in Section 10. SAS and R programming statements are provided to specify the details of the analyses.

# 9.1 Missing data

All analyses based on the PPS will be based on observed cases (OC). It is acknowledged that the PPS analyses are based on a selected subset of patients who completed the 8 weeks of DB treatment with sufficient compliance and who have no missing data at Week 8. For the assessment of dose-response reliance on this subset was deemed appropriate.

In analyses based on the FAS missing data will be imputed using last observation carried forward (LOCF). This may be justified as a conservative analysis since in this study the majority of patients are expected to improve over time [EMA 2010].

Baseline observation carried forward (BOCF) will be used as a sensitivity analyses for missing data imputation. Another sensitivity analysis is provided by a mixed model which does not impute the missing data and, in that sense, can be seen as a OC analysis. Mixed models are based on the missing at random (MAR) assumption, i.e.: missing data can be fully accounted for by baseline covariates and prior measurements. The MAR assumption is not unreasonable in the hypertension context, although it cannot be proven.

# 9.2 Dose-response analysis for the primary endpoint

Dose-response data include changes from baseline to Week 8 of DB treatment period in mean trough SiDBP (primary endpoint) and mean trough SiSBP (secondary endpoint). These data will be analyzed using the MCP-Mod approach [Bretz 2005, Pinheiro 2006]. In brief, this methodology consists of two steps:

- 1. MCPs step to establish a dose-response signal (i.e., the dose-response curve is not flat) using MCPs.
- 2. Modeling (Mod) step to estimate the dose-response curve and target doses using modeling techniques.

In this study six models have been pre-specified in the protocol for consideration in all MCP-Mod analyses: linear, linear in log (linlog), quadratic, maximum effect ( $E_{max}$ ), sigmoidal  $E_{max}$  and logistic. See Table 3 for the parameterization of the dose-response models and Figure 2 as an illustration of their basic shapes. The initial values for the parameters are needed in the MCP step of the procedure. They will be estimated in the Mod step based on the actual data.
Table 3 Parameterization of models considered in MCP-Mod analyses

| Model | Response* | Initial value(s) |
|---|---|---|
| | | for parameters |
| Linear | E0 + delta • dose | NA* |
| Linear in log | E0 + delta • $\log(dose + 0.5)$ | NA* |
| Quadratic | E0 + beta1 • $dose$ + beta2 • $dose^2$ | beta2/beta1 = -0.005 |
| $E_{\text{max}}$ | $E0 + E_{\text{max}} \cdot dose/(ED50 + dose)$ | ED50 = 50 |
| Sigmoidal E <sub>max</sub> | $E0 + E_{max} \cdot dose^h/(ED50^h + dose^h)$ | ED50 = 50, h = 0.5 |
| Logistic | $E0 + E_{\text{max}}/(1 + \exp[\{\text{ED50 - } dose\}/\text{delta}])$ | ED50 = 50, |
| | | delta = 50 |

Dose = 0, 5, 10, 25 and 50 mg of ACT-132577;

Figure 2 Dose-response curves considered in MCP-Mod procedure



<sup>\*</sup>Not applicable for E0, delta (in linear and linlog models), and Emax

The Lisinopril group will be excluded from all analyses of the dose-response. Note that the 'Model means' on the vertical axis are plotted on a scale from 0 to -1 for illustrative purposes. The actual scale will depend on the endpoint analyzed.

The null hypothesis of 'no dose-response' will be rejected if at least one of the six Multiple Contrast Tests (MCTs) has a multiplicity adjusted p-value < 0.05. All statistically significant models (i.e., with an adjusted p-value < 0.05) are fitted in the Mod step and for each model Akaike's Information Criterion (AIC) is calculated. The smaller the value of AIC (= model deviance + 2 times the number of model parameters), the better the fit. The analysis will be performed using the R-package *DoseFinding* [Bornkamp 2016]. The basic R-code is:

In the Mods function call the candidate models are specified, together with the assumed direction of the effect (decreasing for change from baseline in blood pressure). In the call to the MCPMod function, DF is a data frame with objects dose, resp (for response), and base (for the baseline value) and Delta is a target difference vs placebo (Delta=3 for DBP; Delta=5 for SBP). The object *MMfit* will be summarized to obtain the MCP test, parameter estimates, target dose and AIC. These elements will go in a summary table. The object will be plotted to display the fitted dose-response curves.

Subgroup analyses based on MCP-Mod can be performed by fitting the selected model by subgroup using the *fitMod* function for which the basic R-code is:

```
MMfit1 <- fitMod(dose=dose, resp=resp, data=DF[DF$subg==1,], addCovars=~base,
model=MMfit$selMod)
MMfit2 <- fitMod(dose=dose, resp=resp, data=DF[DF$subg==2,], addCovars=~base,
model=MMfit$selMod)</pre>
```

As a supportive analysis to MCP-Mod, change from baseline to Week 8 in DBP and SBP will also be analyzed in an ANCOVA model using the Dunnett test.

```
proc mixed data=dset;
  class treat;
  model outcome=treat base;
  lsmeans treat/ adjust=Dunnett diff=control('0') cl;
  where week=8 and treat in (0,1,2,3,4);
run;
```

## 9.3 Dose-response analyses for continuous data

Changes from baseline to Week 8 for other continuous OBPM endpoints will be analyzed using the general MCP-Mod approach which consists of two steps.

First an ANCOVA model is fitted with a factor for treatment group and a covariate for the baseline value. The SAS statements (using mock variable names and values) for this model are:

```
ods output Ismeans=Ism, * export data set Ism as xpt file; proc mixed data=dset; class treat; model outcome=treat base; Ismeans treat/cov; where week=8 and treat in (0,1,2,3,4);
```

Here, treat=0, 1, 2, 3, and 4 for placebo, 5 mg, 10 mg, 25 mg and 50 mg of ACT-132577, respectively. Note that the active comparator (treat=5) is excluded from this analysis.

Then the LSMeans from this model will be analyzed using the general MCP-Mod approach. The R statements for this analysis are (Delta=3 for DBP; Delta=5 for SBP):

```
# read data frame lsm from xpt file
est <- lsm$ESTIMATE # LSMeans
C <- lsm[,c("COV1","COV2","COV3","COV4","COV5")] # covariance matrix
doses <- c(0,5,10,25,50)
MMfit <- MCPMod(type="general", dose=doses, resp=est, S=as.matrix(C),
models=candMod, Delta=3, alpha=0.05)</pre>
```

Repeated measurements (e.g., changes from baseline to Weeks 2, 4 and 8) will be analyzed in two ways: focusing on the last time point (e.g., Week 8 and using Week 2 and Week 4 only to predict missing data, if needed) and estimating the average effect over time. In both cases the general MCP-Mod approach was used.

Last time point. First a mixed model is fitted with factors for treatment group, time and treatment by time interaction and covariates for the baseline value and the interaction between baseline and time. An unstructured covariance matrix will be used to account for the correlation between repeated measurements from the same subject. The SAS statements for this model are:

```
ods output lsmeans=lsml (where=(week=8)); * export data set lsml as xpt file; proc mixed data=dset noclprint=6; class treat week subjid; model outcome=treat week treat*week base base*week; repeated week/ subject=subjid type=un; lsmeans treat*week/ cov; where treat in (0,1,2,3,4); run;
```

The LSMeans at Week 8 will then be analyzed using the general MCP-Mod approach. The R statements for this analysis are the same as above, except for:

```
C <- lsm[,c("COV3","COV6","COV9","COV12","COV15")] # covariance matrix</pre>
```

Average over time. First the same mixed model is fitted, but without the treatment by time interaction. The SAS statements for this model are:

```
ods output Ismeans=Ism2; * export data set Ism2 as xpt file; proc mixed data=dset noclprint=6; class treat week subjid; model outcome=treat week base base*week; repeated week/ subject=subjid type=un; Ismeans treat/ cov; where treat in (0,1,2,3,4); run;
```

Then the LSMeans (averages over time) will be analyzed using the same R statements as above with:

```
C <- lsm[,c("COV1","COV2","COV3","COV4","COV5")] # covariance matrix</pre>
```

## 9.4 Dose-response analyses for binary data

Binary outcomes include the control and response status for DBP (or SBP) at a fixed time point and will also be analyzed using the general MCP-Mod approach. First a logistic regression model is fitted with a factor for treatment group and a covariate for the baseline value of DBP (or SBP). The SAS statements (using mock variable names and values) for this model are:

```
ods output lsmeans=lsm, * export data set lsm as xpt file; proc logistic data=dset descending; class treat/param=glm, model resp=treat base; lsmeans trt01pn/ ilink cov; where week=8 and treat in (0,1,2,3,4); run;
```

Then the estimated differences vs placebo (in data set diff) will be analyzed using the general MCP-Mod approach [Pinheiro 2014].

```
# read data frame lsm from xpt file
est <- lsm$MU #LSMeans
C <- diag(lsm$STDERRMU^2)
candMod <- Mods(linear = NULL, linlog = NULL, quadratic = -0.005, emax = 50,</pre>
```

Since control and response statuses are not expected to change much over time (i.e., from Week 2 to 8) a repeated measures analysis of these binary endpoints was omitted.

### 10 STATISTICAL ANALYSES

## **10.1** Overall testing strategy

All statistical testing will be performed at a two-sided significance level of 0.05 using 95% confidence intervals (CIs).

In the main analysis of the primary endpoint in the PPS the type I error is controlled by the MCT part of the MCP-Mod methodology. The primary objective of the trial will be evaluated based on this analysis.

The type I error of the MCP-Mod analysis in the FAS is similarly protected. In the other supportive analysis of the primary endpoint Dunnett's test will be used to correct for testing multiple doses vs placebo. The alpha is formally controlled only for the main analysis; all other analyses are considered exploratory.

In all analyses of secondary and other efficacy variables, no correction will be made for multiple testing.

## 10.2 General rules for data presentations

This section describes the general rules applied for all data displays.

SAS version 9.3 is used for the statistical analyses except for the primary endpoint (dose-response analysis) that is analyzed by means of the R package.

Unless otherwise specified in this document:

- All listings are sorted by randomized treatment, subject number and, when appropriate, by visit / date of assessment. If a listing includes non-randomized subjects, these will appear after the randomized subjects. All data collected are displayed, including unscheduled visits (if any).
- In summary tables and graphical representations, subjects are grouped by randomized treatment group, except for the SAF for which the actual treatment is used.
- In summary tables based on the RND, FAS, PPS and SAF, the order of the treatment groups is: placebo, ACT-132577 5 mg, ACT-132577 10 mg, ACT-132577 25 mg, ACT-132577 50 mg and Lisionpril 20 mg, followed by Total (if required). In summary tables based on the RIS or SCR, only a total column will be given.

- The absolute change from baseline to Visit X is defined as the difference between the post-baseline Visit X value and the baseline value.
- In order to analyze the data at the relevant planned (scheduled) visits, all recorded assessments for each subject up to the Week 10 visit are reassigned to the most appropriate visit according to the time window for that visit. The windows are consecutive (i.e., there are no gaps) and are based on the study day corresponding to the date of assessment. Any unscheduled visit is also mapped to a time window. Details of the visit mapping are given in Section 11.1.
- According to section 11.3.2.2 of the protocol, imputation rules for missing data are defined for the evaluation of efficacy endpoints at Week 8. Subjects without a value in the defined Week 8 time window are included in the analysis according to the rules highlighted in Section 9.

## 10.3 Display of subject disposition, protocol deviations and analysis sets

### **10.3.1** Subject disposition

Summary tables are provided, on the SCR, RIS and RND sets [see Section 7 for terminology], by treatment group (where applicable) and overall, to display the following information:

- Disposition of subjects (screened, entered in run-in, randomized, treated i.e., who received at least one dose of study treatment, who completed treatment see Section 5.3.3 for definition, who completed study see Section 5.4 for details). This summary table is also provided by site.
- Reasons for screening failures [see definition in Section 5.1, overall only].
- Reasons for run-in failures [see definition in Section 5.1, overall only].

Percentages are calculated based on screened subjects [see definition in Section 5.1] or run-in subjects where appropriate. A listing of screening failures is provided for the SCR and a listing of run-in failures for the RIS. Randomization scheme and codes and code break or subject unblinding (if any) are provided in separate listings on the RND set.

### 10.3.2 Protocol deviations

All important PDs (as defined by the PD list) will be summarized on the FAS by categories, displaying counts and percentages of subjects with at least a PD, by treatment group and overall. This summary table is sorted, within each PD temporal category, by overall frequency, in descending order; if a tie occurs, the tied characteristics will be sorted alphabetically.

All reported PDs will be reported in a subject listing on the SCR set. Important PDs will be flagged accordingly.

### 10.3.3 Analysis sets

A summary table is provided on the RND set to display the composition of FAS, PPS and SAF analysis sets, by treatment group and overall. A listing of subject participation in the different analysis sets is also provided.

A separate summary table is provided on the RND set to display the reasons for exclusion from the above analysis sets, by treatment group and overall. In addition, the same table is provided by site.

## 10.4 Analyses of subject characteristics

### 10.4.1 Demographics

All data [see definition in Section 5.2.1] will be reported in a subject listing based on the RND. The listing will include the other baseline characteristics defined in Section 5.2.3.

Demographic characteristics will be summarized using descriptive statistics by treatment group as well as overall for the FAS and PPS.

Note that age will be summarized as a continuous variable as well as a categorical variable ( $< 65, \ge 65$  years). Age as per EudraCT categories ( $18-64, 65-84, \ge 85$  years) will be tabulated separately based on the FAS.

#### 10.4.2 Baseline disease characteristics

All data [see definition in Section 5.2.2] will be reported in a subject listing based on the SCR. Baseline disease characteristics will be summarized by treatment group as well as overall for the FAS and PPS.

### 10.4.3 Other baseline characteristics.

Other baseline disease characteristics [see definition in Section 5.2.3] will be summarized by treatment group and overall using descriptive statistics for the FAS and PPS.

### 10.4.4 Medical history

All previous or ongoing diseases / diagnoses [see definition in Section 5.2.4] will be reported in a subject listing. Ongoing diseases / diagnoses will be flagged accordingly. Previous and ongoing diseases / diagnoses will be summarized in separate tables. This will be done for the FAS and PPS.

Previous or ongoing diseases / diagnoses will be summarized by treatment group and overall, together displaying counts and percentages of subjects having experienced at least one disease. Counts and percentages of subjects having experienced at least one disease are presented by system organ class (SOC) and individual preferred term within each SOC. The summary table is presented in descending order according to the

incidence in the highest-dose of active test treatment (e.g., SOC and individual preferred term within each SOC with the highest number of occurrences appears first). Equal frequency of different SOC / individual preferred terms is sorted in alphabetical order of the SOC / individual preferred term.

The counting of the diseases is handled as follows:

- Subjects with two or more occurrences of the same disease (as qualified by the same preferred term[s]) are counted only once.
- In the event that the reported disease is assigned to several preferred terms, subjects are counted for each individual preferred term.

## 10.4.5 Previous and concomitant therapies

For study reporting purposes, all previous and/or concomitant therapies will be reported in a subject listing.

Counts and percentages of subjects having taken at least one previous, study concomitant and double-blind treatment concomitant therapy [see definition in Section 5.2.5] are presented by treatment group, by ATC class and individual preferred term within each ATC class, separately.

The summary tables are presented in descending order according to the incidence in the highest-dose of active test treatment (e.g., ATC and individual preferred term within each ATC with the highest number of occurrences appear first). Equal frequency of different ATC / individual preferred terms is sorted in alphabetical order of the ATC / individual preferred term.

The counting of the therapies is handled as follows:

- Subjects who took the same therapy more than once (as qualified by the same preferred term[s]) are counted only once.
- In the event of the reported medication being assigned to several preferred terms, subjects are counted for each individual preferred term.

For each preferred term the class are allocated using the 3 digits of the ATC code.

Specific previous and concomitant therapies will be displayed separately as described above.

### 10.4.6 Other subject characteristics

Not applicable.

## 10.5 Analysis of study treatment duration and compliance

### 10.5.1 Study treatment duration

The duration of double-blind study treatment [see definition in Section 5.3.1] will be summarized on the PPS and SAF using descriptive statistics. Additionally, double-blind study treatment will be summarized as categorical variable, presenting the cumulative distribution by class interval categorized as 0-2, > 2-4, > 4-8 and > 8 weeks and displaying counts and percentages of subjects in each class interval.

In addition, run-in study treatment duration will be summarized for the RIS.

### **10.5.2** Compliance with study treatment

Double-blind treatment compliance [see definition in Section 5.3.2] will be summarized on the FAS and PPS displaying counts and percentages of subjects with compliance categorized as: < 80%, 80-120%, and > 120%. Run-in treatment compliance will be summarized similarly for the RIS.

### 10.5.3 Study treatment discontinuation

A summary table is provided for the SAF to display counts and percentages of subjects who prematurely discontinued double-blind study treatment, as well as the associated reasons [see definition in Section 5.3.3], by treatment group and overall.

Note that premature double-blind study treatment discontinuation does not necessarily imply study withdrawal.

In addition, premature run-in treatment discontinuation will be summarized for the RIS.

### 10.5.4 Study treatment adjustments or interruptions

The number and percentage of subjects with DB study treatment interruptions will be provided for the SAF. The associated reasons will be summarized similarly.

### 10.5.5 Study withdrawal

A summary table is provided for the RND to display counts and percentages of subjects who prematurely discontinued the study after randomization, as well as the associated reasons by treatment group and overall. A listing of discontinued subjects is provided on the RND set. A similar table and listing based on the RIS will be provided for premature study discontinuation during run-in.

### 10.6 Analysis of the primary efficacy variable(s)

The primary efficacy variable (change from baseline to Week 8 of DB treatment in mean trough SiDBP, measured by OBPM) will be analyzed in the PPS and the FAS. The PPS analysis is the primary analysis, the analysis in the FAS is supportive.

The primary efficacy variable will be summarized by treatment group using descriptive statistics for the PPS and FAS.

## 10.6.1 Hypothesis and statistical model

The null hypothesis associated with the primary endpoint is that there is no dose-response relationship.

$$H_0$$
:  $\mu_0 = \mu_1 = \mu_2 = \mu_3 = \mu_4$ 

Here,  $\mu_i$  denotes the mean change from baseline to Week 8 in mean trough SiDBP ( $\mu$ ) for ACT-132577 dose (i) (where I = 0 corresponds to placebo). A value of  $\mu_i$  < 0 corresponds to a decrease in SiDBP.

The alternative hypothesis is that there is a monotonic dose-response for the primary endpoint.

H<sub>1</sub>: 
$$\mu_0 \ge \mu_1 \ge \mu_2 \ge \mu_3 \ge \mu_4$$
 and  $\mu_i > \mu_j$  for at least one  $i > j$  or  $\mu_0 \le \mu_1 \le \mu_2 \le \mu_3 \le \mu_4$  and  $\mu_i < \mu_j$  for at least one  $i > j$ 

Note that larger values of  $\mu_i$  – corresponding to less decrease (or more increase) from baseline to Week 8 in mean trough SiDBP with increasing dose of ACT-132577 – are less favorable. The first part of the alternative hypothesis corresponds to ACT-132577 being superior to placebo, whereas the second part corresponds to ACT-132577 being worse than placebo.

## 10.6.2 Handling of missing data

In the PPS there will be no missing data from the primary endpoint given the definition of PPS. For the handling of missing data in the FAS, refer to Section 9.1.

#### 10.6.3 Main analysis

The change from baseline to Week 8 of DB treatment period (Period II) in mean trough SiDBP will be analyzed using the MCP-Mod approach [Bretz 2005, Pinheiro 2006] described in Section 9.1.

A placebo-corrected mean reduction from baseline of at least 4 mmHg is considered clinically relevant.

Some examples of  $E_{max}$  dose-response relationships are given in Figure 3, where it is assumed that the minimum response will be obtained with placebo (mean change from baseline -4 mmHg) and the maximum response (change from baseline -8 or -9 mmHg) will be reached at the highest dose of ACT-132577 (50 mg).

Figure 3 Examples of  $E_{max}$  dose-response relationships



Six candidate dose-response models were pre-specified in the protocol: linear, linear in log-dose, quadratic,  $E_{max}$ , sigmoidal  $E_{max}$  and logistic. The analysis will be performed using the R-package DoseFinding [Bornkamp 2016]. A dose-response relationship is demonstrated if at least one of the six MCTs has an adjusted p-value < 0.05. The best fitting model will be selected based on AIC. That model will be used to estimate the minimum effective dose, defined as the dose that achieves a placebo-corrected mean reduction from baseline of at least 4 mmHg with a 95% CI excluding 0.

## 10.6.4 Supportive/sensitivity analyses

Supportive analyses. The analysis of the primary endpoint in the FAS using LOCF to impute missing Week 8 data will be performed as described in the previous section.

In the PPS as well as the FAS (with LOCF), change from baseline to Week 8 of DB treatment period (Period II) in mean trough SiDBP will be analyzed using an ANCOVA model with a factor for treatment group (placebo and four doses of ACT-132577) and a covariate for baseline mean trough SiDBP. Each of the four doses of ACT-132577 will be compared to placebo applying Dunnett's test. The active comparator will be compared separately versus placebo using an ANCOVA model with a factor for treatment group

(placebo or active comparator) and a covariate for baseline mean trough SiDBP. In the FAS missing data will be imputed by LOCF.

*Sensitivity analysis*. As a sensitivity analysis for missing data imputation by LOCF an MCP-Mod analysis based on BOCF will be performed in the FAS.

Also in the FAS, changes from baseline to time window Visit 5 (Week 2), time window Visit 4 (Week 4) and Week 8 of DB treatment period (Period II) in mean trough SiDBP will also be analyzed using repeated measurements model. A mixed model will be applied with factors for treatment group, time (Week 2, 4 or 8), treatment by time interaction and a covariate for baseline mean trough SiDBP. An unstructured covariance matrix will be used to account for the correlation between repeated measurements from the same subject. This can be seen as an OC analysis. The treatment group LSMeans obtained from this model will be analyzed using the general MCP-Mod approach [Pinheiro 2014].

Average effect over time. In order to investigate the dose-response on the average treatment effect over time, the same mixed model will be used, but without the treatment by time interaction. Treatment group LSMeans will be analyzed using the general MCP-Mod approach.

### 10.6.5 Subgroup analyses

Subgroup analyses will be performed on the PPS by age (< 65 versus  $\geq$  65 years), sex, race and country.

In the absence of a published, consolidated approach for subgroup analyses for dose-response, subgroup analyses will be performed by fitting the 'best' model from the overall analysis [see Section 10.6.3] in each of the subgroups. The fitted dose-response curves will be compared visually between subgroups. Dose-response by subgroup interaction may be investigated in an ad hoc fashion based on AIC.

## 10.7 Analysis of the secondary efficacy variables

Secondary efficacy variables will be analyzed for the PPS at  $\alpha$  = 0.05 (two-sided) using 95% CIs. Additionally, change from baseline to Week 8 in mean trough SiSBP will be analyzed for the FAS. No correction for multiple testing will be applied for these analyses.

Change from baseline to Week 8 of DB treatment period (Period II) in mean trough SiSBP will be analyzed similarly to the primary endpoint (SiDBP), i.e., MCP-Mod will be applied, supplemented by the ANCOVA and the repeated measurements models described above. The correlation between the changes from baseline in SiDBP and SiSBP will be displayed in a scatter plot for each post-baseline time point.

Control (< 90 mmHg and < 85 mmHg, separately) and response (Y/N) at Week 8 of DB treatment period (Period II) based on trough SiDBP will be analyzed using a logistic regression model with a factor for treatment group and a covariate for baseline mean trough SiDBP. Control and response status at Week 8 of Period II based on trough SiSBP will be analyzed similarly.

Change from baseline to Week 8 of DB treatment period (Period II) in 24-hour mean DBP based on ABPM will be analyzed using an ANCOVA with a factor for treatment group and a covariate for baseline 24-hour mean DBP. Change from baseline to Week 8 of DB treatment period (Period II) in 24-hour mean SBP based on ABPM will be analyzed similarly.

The baseline and Week 8 average ABPM-DBP curves over time (by hour) will be plotted by treatment group [averaging as described in Section 5.5.2]. Additionally, the Week 8 minus baseline difference will be plotted vs time. Trough to peak ratios for DBP will be calculated by treatment group as described in Section 5.5.2.

## 10.8 Analysis of other efficacy variables

Other efficacy analyses will be performed on the PPS.

Changes from baseline to Week 2 (time window Visit 5) and Week 4 (time window Visit 6) of DB treatment period (Period II) in mean trough SiSBP and SiDBP (OBPM) will be obtained from the repeated measurements model as described in Section 10.6.4 under *sensitivity analysis*.

Change from baseline to Week 8 of DB treatment period (Period II) in mean daytime DBP (SBP) measured by ABPM will be analyzed using an ANCOVA with a factor for treatment group and a covariate for baseline mean daytime ABPM. Change from baseline to Week 8 of DB treatment period (Period II) in mean night time DBP (SBP) measured by ABPM will be analyzed similarly.

ABPM-SBP curves will be plotted and trough to peak ratios for SBP will be calculated as described for DBP based on ABPM.

Changes from baseline to Week 10 (time window Visit 8; Week 2 of withdrawal period - Period III) in mean trough SiSBP and SiDBP (OBPM) will be obtained by extending the repeated measurements model described in Section 10.6.4 with an additional time point for time window Visit 8 (Week 10 i.e., Week 2 of withdrawal period - Period III).

Changes from Week 8 of Period II to time Week 10 (time window Visit 8; Week 2 of withdrawal period - Period III) in mean trough SiSBP and SiDBP (OBPM) will be obtained from the same model using appropriate treatment and time contrasts.

All efficacy analyses are summarized in Table 4.

Table 4 Summary of efficacy analyses

| Efficacy<br>analysis | Endpoint | Measure | Week | Model | Dataset | t(imputation) |
|---|---|---|---|---|---|---|
| Primary | SiDBP | OBPM | 8 | MCP-Mod | PPS | |
| - Supportive | SiDBP | OBPM | 8 | MCP-Mod | | FAS<br>(LOCF) |
| | SiDBP | OBPM | 8 | ANCOVA (Dunnett) | PPS | FAS<br>(LOCF) |
| - Sensitivity | SiDBP | OBPM | 8 | MCP-Mod | | FAS<br>(BOCF) |
| | SiDBP | OBPM | 8 | MCP-Mod based on mixed model <sup>a</sup> | | FAS (OC) |
| - Average over time | SiDBP | OBPM | 2,4,8 | MCP-Mod based on mixed model <sup>b</sup> | PPS | FAS (OC) |
| - Subgroup | SiDBP | OBPM | 8 | MCP-Mod by subgroup | PPS | |
| Secondary | SiSBP | OBPM | 8 | MCP-Mod | PPS | FAS<br>(LOCF) |
| | SiSBP | OBPM | 8 | ANCOVA (Dunnett) | PPS | FAS<br>(LOCF) |
| | SiSBP | OBPM | 8 | MCP-Mod based on mixed model <sup>a</sup> | | FAS (OC) |
| | Average<br>SiSBP over<br>time | OBPM | 2,4,8 | MCP-Mod based on mixed model <sup>b</sup> | PPS | FAS (OC) |
| | Subgroup<br>SiSBP | OBPM | 8 | MCP-Mod | PPS | |
| | Control/<br>response of<br>SiDBP | OBPM | 8 | MCP-Mod based on logistic regression | PPS | |
| | Control/<br>response of<br>SiSBP | OBPM | 8 | MCP-Mod based on logistic regression | PPS | |
| | 24-hour mean DBP | ABPM | 8 | ANCOVA | PPS <sup>c</sup> | |
| | 24-hour mean SBP | ABPM | 8 | ANCOVA | PPS <sup>c</sup> | |
| | Trough to peak ratio DBP | ABPM | 8 | Descriptive statistics | PPS <sup>c</sup> | |
| Other | Mean daytime<br>DBP | ABPM | 8 | ANCOVA | PPS <sup>c</sup> | |

#### Confidential

| Efficacy | Endpoint | Measure | Week | Model | Dataset(imputation) |
|---|---|---|---|---|---|
| analysis | | | | | |
| | Mean night | ABPM | 8 | ANCOVA | PPS <sup>c</sup> |
| | time DBP | | | | |
| | Mean daytime | ABPM | 8 | ANCOVA | PPS <sup>c</sup> |
| | SBP | | | | |
| | Mean night | ABPM | 8 | ANCOVA | PPS <sup>c</sup> |
| | time SBP | | | | |
| | Trough to | ABPM | 8 | Descriptive statistics | PPS <sup>c</sup> |
| | peak ratio SBP | | | | |
| | SiDBP | OBPM | 8,10 | ANCOVA | PPS |
| | SiSBP | OBPM | 8,10 | ANCOVA | PPS |

<sup>\*</sup> If applicable. In the PPS all analyses are based on OC.

ABPM = ambulatory blood pressure monitoring; ANCOVA = analysis of covariance; BOCF = baseline observation carried forward; DBP = diastolic blood pressure; FAS = Full Analysis Set; LOCF = last observation carried forward; MCP-Mod = Multiple Comparison Procedure - Modeling; OBPM = automated office blood pressure measurement; OC = observed cases; PPS = Per-Protocol Set; SBP = systolic blood pressure; SiDBP = sitting diastolic blood pressure; SiSBP = sitting systolic blood pressure.

MCP-Mod based on mixed model (logistic regression, ANCOVA) implies that first the mixed model (logistic regression, ANCOVA) is performed and then the estimated differences vs placebo are analyzed using the general MCP-Mod approach [Pinheiro 2014].

## 10.9 Analysis of safety variables

All safety analyses described below will be performed on the SAF. All safety data will be listed, with flags for abnormalities, when applicable.

### 10.9.1 Adverse events

All reported AEs will be listed, together with the assigned preferred term/SOC. The listings will indicate the period of onset of the AE (run-in, DB treatment or placebo WD).

Treatment-emergent AEs [see definition in Section 5.6.1.1] will be summarized displaying, for each treatment group, counts and percentages of subjects having experienced at least one treatment-emergent AE. Counts and percentages of subjects having experienced at least one treatment-emergent AE are presented by SOC and individual preferred term within each SOC. The summary tables are presented in descending order according to the incidence in the highest-dose of active test treatment (e.g., SOC and individual preferred term within each SOC with the highest number of

<sup>&</sup>lt;sup>a</sup> Also including Week 2 and 4 data, but only to predict missing Week 8 data.

<sup>&</sup>lt;sup>b</sup> Including Week 2, 4 and 8 data to estimate the average effect of time.

<sup>&</sup>lt;sup>c</sup> ABPM analyses are based on the subset of the PPS described in Section 5.5.

occurrences appears first). Equal frequency of different SOC/individual preferred terms is sorted in alphabetical order of the SOC/individual preferred term.

Treatment-emergent AEs related to study treatment, treatment-emergent AEs leading to premature discontinuation of study treatment and treatment-emergent AEs with fatal outcome will be summarized, separately, by SOC and individual preferred term.

Treatment-emergent AEs, treatment-emergent AEs leading to premature discontinuation of study treatment and treatment-emergent AEs with fatal outcome will be summarized also by preferred term only. Treatment-emergent AEs are also summarized by maximum intensity.

For the disclosure of the results to EudraCT and ClinicalTrials.gov (rather than for the purpose of the clinical study report), a summary table with an overview of treatment-emergent AEs is provided displaying, for each treatment group, counts and percentages of subjects having experienced at least a treatment-emergent AE, a severe AE, a study-treatment related AE, an AE leading to study treatment discontinuation, a non-serious frequent AE, a serious AE, a study-treatment related serious AE, a fatal SAE.

The occurrence of non-serious, frequent (i.e., the percentage of subjects in at least one of the treatment groups equals or exceeds five percent) treatment-emergent AEs will be tabulated by SOC and individual preferred term within each SOC.

### 10.9.2 Deaths, other serious adverse events

#### 10.9.2.1 Deaths

The primary cause of death coded according to MedDRA dictionary [see Section 5.6.2] will be summarized displaying, for each treatment group, counts and percentages of subjects by class and individual preferred term within each class; the summary table is presented in descending order according to the incidence in the highest-dose of active test treatment (equal frequencies are sorted in alphabetical order).

All deaths will be listed. The listings will indicate the period in which the death occurred (run-in, DB treatment, placebo WD).

### 10.9.2.2 Serious adverse events

All reported SAEs will be listed and tabulated as described above for AEs.

The occurrence of treatment-emergent serious AEs will be summarized by SOC and individual preferred term within each SOC. The table is presented in descending order according to the incidence in the highest-dose of active test treatment (i.e., SOC and individual preferred term within each SOC with the highest number of occurrences appears first). Ties are sorted in alphabetical order.

Treatment-emergent SAEs will also be summarized by preferred term only.

For the disclosure of the results to EudraCT and ClinicalTrials.gov (rather than for the purpose of the clinical study report), treatment-emergent SAEs will be summarized displaying, for each treatment group, counts and percentages of subjects with at least a treatment-emergent SAE plus the number of events (counted exactly the number of times they occurred also within a subject) by SOC and individual preferred term. The summary table is presented in descending order according to the incidence in the highest-dose of active test treatment (i.e., SOC and individual preferred term within each SOC with the highest number of occurrences appears first). Equal frequency of different individual preferred terms is sorted in alphabetical order of the individual preferred term. Similarly, a separate summary is presented for treatment-emergent SAEs related to study treatment. In addition, treatment-emergent SAEs with fatal outcome and treatment-emergent SAEs with fatal outcome related to study treatment will be summarized separately, similarly to treatment-emergent SAEs.

### 10.9.2.3 Adverse events leading to study treatment discontinuations

A separate subject listing is provided with treatment-emergent AEs leading to study treatment discontinuation. Treatment-emergent AEs leading to premature study treatment discontinuation will be summarized by SOC and preferred term as well as by preferred term only.

#### 10.9.2.4 Other adverse events

Not applicable.

### 10.9.3 Electrocardiography (ECG)

Double-blind treatment-emergent ECG abnormalities [see definition in Section 5.6.7.1] will be summarized, by treatment group, displaying counts and percentages of subjects (and 95% confidence limits according to the Clopper-Pearson method) with at least one treatment-emergent ECG abnormality. Values from unscheduled visits are included. Subjects may be included in more than one category as the marked abnormality are presented cumulatively.

ECG variables are displayed in a subject listing on the SCR set; a separate listing is provided of all ECG variables, restricted to subjects with at least one abnormality [see Section 5.6.7 for details].

### **10.9.4** Laboratory tests

All hematology and chemistry parameters provided by the central and local laboratory are displayed in a subject listing. Marked laboratory abnormalities will be flagged

accordingly. Laboratory values below the limit of detection (i.e., preceded by '<') will be replaced by half that limit in calculations as well as in determining abnormalities.

Hematology, chemistry and urine parameters UACR will be summarized by treatment group for each time window visit. Changes from baseline in these parameters will be summarized for each post-baseline assessment, displaying:

- observed values at baseline and at the post-baseline visit window
- absolute change from baseline to post-baseline visit window

In each evaluation only subjects who had both the assessments at baseline and the considered post-baseline time point are included.

## 10.9.4.1 Treatment-emergent marked laboratory abnormalities

For each category (i.e., LL, LLL, HH, HHH, HHHH), treatment-emergent marked laboratory abnormalities [see definition in Section 5.6.8.1] will be summarized by treatment group, displaying counts and percentages of subjects with at least a treatment-emergent marked laboratory abnormality for each parameter for which the marked abnormality is defined. Values from unscheduled visits are included. Subjects may be included in more than one category for the same parameter.

In addition, the number of patients with ALT  $> 3 \times$  upper limit of normal (ULN) and bilirubin  $> 2 \times$  ULN will be tabulated by treatment group and time point (baseline, Week 8).

Percentages are calculated as number of subjects with at least one abnormality for the parameter under consideration divided by the number of subjects with any post-baseline laboratory measurement.

The distribution of the changes from baseline in hemoglobin will be plotted for each post-baseline visit. As an exploratory analysis, dose trends in the change from baseline to Week 8 in hemoglobin will be analyzed using the MCP-Mod approach. The active comparator will be excluded from these analyses.

### 10.9.5 Physical examination, vital signs and body weight

Physical examination data performed during the course of the study will be reported in a subject listing. Pulse rate and body weight measurements will be reported in a subject listing and summarized by time window visit.

Furthermore, for each post-baseline assessment, average PR (from BpTRU®) and body weight will be summarized displaying, for each treatment group, descriptive statistics for:

- observed values at baseline and at the post-baseline visit window
- absolute change from baseline to post-baseline visit window

In each evaluation only subjects who had both the assessment at baseline and the considered post-baseline assessment are included. Only measurements obtained in sitting position will be taken into account.

The density of the changes from baseline in body weight will be plotted for each post-baseline visit. As an exploratory analysis, dose trends in the change from baseline to Week 8 in body weight ([kg]) will be analyzed using the MCP-Mod approach. The active comparator will be excluded from these analyses.

### 10.9.6 Other safety variables

Not applicable.

## 10.10 Analysis of quality of life variables (TSQM vII)

Not applicable.

## 10.11 Analysis of pharmacoeconomic variables

Not applicable.

## 10.12 Analysis of epidemiological measures and risk-benefit evaluations

Not applicable.

## 10.13 Analysis of pharmacodynamic variables

For the analysis of ET-1 the PK set will be used. ET-1 plasma concentrations will be summarized by active treatment and visit by arithmetic mean, SD of the mean, minimum, maximum, median, coefficient of variation of the arithmetic mean (CV%), and number of observations. A subject listing presenting ET-1 data will also be provided. Data presentations will follow the general rules as described in Section 10.2.

## 10.14 Analysis of pharmacokinetic variables

ACT-132577 plasma concentrations and, if applicable, summarized for ACT-132577 treated groups only.

The data will be summarized by active treatment and visit by arithmetic mean, SD of the mean, minimum, maximum, median, coefficient of variation of the arithmetic mean (CV%), and number of observations. For mean value calculations, all values below the limit of quantification (BLQ values) will be set to zero. If  $\leq 50\%$  of the values at a given time point are BLQ, these values will be set to zero for calculation of the mean value. If  $\geq 50\%$  of the values at a given time point are BLQ, no mean value will be calculated. Additionally, summaries will be created by sex, race and age.

### 11 GENERAL DEFINITIONS AND DERIVATIONS

### 11.1 Time windows

To allow analysis of data at the relevant planned (scheduled) visits, all recorded assessments, including unscheduled ones, are re-assigned to the most appropriate visit according to the best fitting time window for that visit [see Table 5]. Note that there are no 'gaps' between the visit windows in order to keep all values in the analysis.

**Table 5** Visit time windows

| Visit | Target day* | Min. day | Max. day |
|----------|-------------|-----------------|------------|
| 1 | -42 | - | -35 |
| 2 | -28 | -34 | -18 |
| 3 | -7 | -17 | -4 |
| 4 | 1 | -3 | 1 |
| 5 | 14 | 1 | 21 |
| 6 | 28 | 22 | 42 |
| 7 - I | 55 | 43 | EOT*** |
| 7 - II** | 56 | EOT + 01 m | EOT + 25 h |
| 8 | 70 | EOT + 25 h 01 m | No limit |

<sup>\*</sup> Number of days from start of double-blind treatment.

ABPM = ambulatory blood pressure monitoring; EOT = End-of-Treatment; OBPM = office blood pressure measurement; SiDBP = sitting diastolic blood pressure.

For assessments for which time is collected, please use the following rules:

- Target day = Target day and time 12:00
- Min. day = Min. day and time 0:00
- Max. day = Max. day and time 23:59

<sup>\*\*</sup> Only for ABPM.

<sup>\*\*\*</sup> For OBPM use EOT + 05 m (for the time of the average SiDBP)

Visit 4 / Day 1

- Target day 1 = Start date/time of DB treatment
- Max. day1 = Start date/time of DB treatment

Visit 5 / Day 1

• Min. day 1 = Start date/time of DB treatment + 1 minute

Visit 7 - I / EOT

• Max. day = End date/time of DB treatment

Visit 7 - II / EOT

• Min. day = End date/time of DB treatment + 1 minute

In the event that there is more than one value within the same time window, the value closest to the planned assessment date will be taken. In the event of equidistant values from the planned time point, the last assessment will be considered for the analyses. Where multiple assessments fall on the same day the latest is then used.

#### 11.2 Run-in treatment start date/time

The run-in treatment start date is the first day of intake of study treatment during the run-in period. It is derived from the first treatment start date (in chronological order) in the **Study Drug Log** eCRF where the 'Study Period' is 'SB RUN-IN'. If the start time of the run-in period is missing, it will be set to 00:00.

### 11.3 Run-in treatment end date/time

The run-in treatment end date is the last day of intake of run-in study treatment. It is derived from the last DB treatment end date (in chronological order) in the **Study Drug Log** eCRF where the 'Study Period' is 'SB RUN-IN'. If the end time of the run-in period is missing, it will be set to the start time of the DB period minus 1 minute, in the event that the DB period is missing it will be set to 23:59.

### 11.4 Randomization date/time

The randomization date/time is taken from IVRS.

### 11.5 Double-blind treatment start date/time

It is the first day of intake of study treatment during the double-blind period. It is derived from the first treatment start date (in chronological order) in the **Study Drug Log** eCRF where the 'Study Period' is 'DB TREATMENT'.

If the date is missing the randomization date (see definition below) is used. If the subject is listed as run-in failure [see definition in Section 5.1] the date is set to 'missing'. If the start time of the double-blind treatment is missing and the start date of DB period corresponds to the date of Randomization, the Randomization time will be used. In other cases the start time of DB will be set to 00:00.

### 11.6 Double-blind treatment end date/time

The double-blind treatment end date is the last day of intake of DB study treatment. It is derived from the last DB treatment end date (in chronological order) in the **Study Drug Log** eCRF where the 'Study Period' is 'DB TREATMENT' and the reason for treatment end is ≠ "TEMPORARILY INTERRUPTED DUE TO AN AE" or "TEMPORARILY INTERRUPTED NOT DUE TO AN AE".

If the study treatment end date is still missing after this derivation, the earliest of the date of Visit 7 - Week 8 / EOT /Part 1 and the date of death (if any) is to be imputed. If the end date is still missing, the EOS date as defined in the Section 2.1 will be used. If the end time of double-blind treatment is missing and DB end date corresponds to the date of the first assessment of ABPM at Visit 7, the time of the first ABPM assessment will be used, otherwise, it will be set to 23:59.

## 11.7 Withdrawal period start date/time

The withdrawal period start date is the first day of intake of placebo during the withdrawal period. It is derived from the first treatment start date (in chronological order) in the **Study Drug Log** eCRF where the 'Study Period' is 'SB WITHDRAWAL'. If the time of the WD period is missing the time of last assessment of ABPM at Visit 7 will be used, otherwise it will be set to 23:59.

## 11.8 Withdrawal period end date/time

The withdrawal period end date is the date of Visit 8, collected in the **Visit Date** eCRF. If the time is missing it will be set to 23:59.

### 11.9 Study day

The study day is the number of days elapsed since the day of first DB treatment plus 1 (start of DB treatment is considered Day 1). For dates prior to Day 1, study day is the negative number of days between the date under consideration and the date of first DB treatment. Therefore, the study day is always different from zero.

## 11.10 Duration of essential hypertension (years)

Duration of essential hypertension (years) = (date of Visit 1 - date of diagnosis)/365.25 with the date of diagnosis collected in the **Essential Hypertension Relevant Disease History** form of the eCRF.

### 11.11 Unit conversion rules

Height (cm) = height (in)  $\times 2.54$ 

Weight (kg) = weight (lbs)  $\times$  0.4536

## 11.12 Body Mass Index (BMI)

BMI  $(kg/m^2)$  = weight  $(kg) / (height [cm] / 100)^2$ 

## 12 HANDLING OF MISSING/INCOMPLETE DATE AND TIME FIELDS

All dates and times used in the analyses are supposed to be complete, apart from the types included in the table below.

The dates in these types that are missing or incomplete are derived as follows:

- Dates are split in 3 parts: year, month and day. Year is the top-level, month is the medium level and day is the low level. If a part expected to contain a number is numeric but the value is outside a valid range, the complete date is handled as missing. For example, if date = 44Nov2000 the whole date is considered to be missing.
- 2 If a part is expected to contain a number is not numeric, i.e., contains values, for example, ND, NA, --, ??, 2?, it is considered as missing.
- If a part is missing, all lower level parts are considered to be missing. This means that a ddmmyy date '21ND99' is considered as '----99'.
- 4 Missing parts are changed into acceptable non-missing values in a way depending on the type of date to be replaced.

In the following, 'lower limit' and 'upper limit' refer to the minimum or maximum, respectively, of a possible date. For example, if the day is missing, the lowest limit is the first day of the given month and the upper limit is the last day of the given month. If the day and month are missing, the lower limit refers to the first day of the given year and the upper limit to the last day of the given year. The earliest and the latest of different dates refer to the first or last date, respectively, when ordered in sequence.

| Type of date | Date is incomplete | Date is missing |
|---|---|---|
| AE resolution date | The upper limit. | No replacement, the AE is considered as ongoing in the analysis. |

| Type of date | Date is incomplete | Date is missing |
|---|---|---|
| AE onset date | If the end date of the AE is not before<br>the start of double-blind treatment,<br>and if the study treatment start falls in<br>the range of possible dates, the study<br>treatment start date is used. In all the<br>other cases the lower limit is used. | Whichever is the earlier of the date of resolution of the AE and the study treatment start date. |
| Medical<br>history end<br>date | The upper limit. | No replacement. |
| Medical<br>history start<br>date | The lower limit. | No replacement. |
| Concomitant medication end date | If the answer to the question 'Ongoing at start of treatment?' in the <b>Previous/Concomitant Medication</b> eCRF is answered 'No' or if the study treatment start date-1 falls in the range of possible dates, the study treatment start date-1 is used. In all the other cases the upper limit is used. | No replacement. If the answer to the question 'Ongoing at start of treatment?' in the <b>Previous/Concomitant Medication</b> eCRF is answered 'Yes' the therapy is considered to have finished after the start of treatment. |
| Concomitant medication start date | If the end date of the medication is not before the informed consent signature date and if the informed consent date falls in the range of possible dates, the informed consent date is used. If the end date of the medication is not before the study treatment start date and if the study treatment start date falls in the range of possible dates, the study treatment start date is used. In all the other cases the lower limit is | No replacement. The medication is considered to have started before the date of consent. |
| | used. | |

| Type of date | Date is incomplete | Date is missing |
|---|---|---|
| Hospitalization discharge date | The upper limit is used. | No replacement. The hospitalization is considered as ongoing in the analysis. |
| Hospitalization admission date | If the onset date of the AE leading to hospitalization falls in the range of possible dates, the onset date of the AE is used. In all the other cases the lower limit is used. | The onset date of the AE leading to hospitalization is used. |

## 13 LIST OF SUMMARY TABLES, LISTINGS AND FIGURES

The table, listing, and figure naming conventions have three components: **Display** (T, L, F), **Name** (free text, in general not more than eight characters, but if required to maintain uniqueness up to a maximum of ten characters), **Suffix** (for example, for analysis sets, or subgroups, not longer than four characters). Multiple suffixes can be added; components/suffixes are separated by '\_'. Example:  $T_{TEAE}_{SAF}$ , summary table (T) of treatment-emergent adverse events (TEAE) on the SAF.

The mock layout column refers to the BST standard Outputs Version 3.0 as of March 31, 2016.

A number of outputs have been identified as key outputs based on which an initial assessment of the dose-response relationship can be made. These are indicated with a 'Yes' in the 'Key' columns of the tables below.

## 13.1 Subject disposition

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DISP | T | Disposition of subjects | SCR | Yes | LAYDISP001 |
| DISP_SITE | T | Disposition of subjects by site | SCR | | LAYDISP001 |
| SCRFAIL | T | Reasons for screening failure | SCR | | LAYDISP002 |
| SCRFAIL | L | Listing of reasons for screening failure | SCR | | LSTCSR011 |
| RUNFAIL | Т | Reasons for run-in failure | RIS | | LAYDISP002 |
| RUNFAIL | L | Listing of run-in failures | RIS | | LSTCSR011 |
| ANSETOV | T | Overview of FAS,<br>PPS, SAF and PK<br>analysis sets | RND | Yes | LAYDISP001 |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| ANSET | L | Listing of subject participation in the different analysis sets | RND | | LSTCSR031 |
| RAND | L | Randomization scheme and codes | RND | | LSTRAN |
| UNBLIND | L | Listing of code break or subject unblinding | RND | | LSTCSR032 |

\* T = Summary Table; L = Listing. FAS = Full Analysis Set; PK = Pharmacokinetic; PPS = Per-Protocol Set; RIS = Run-in Set; RND = All Randomized Set; SAF = Safety Set; SCR = Screened Set.

## 13.2 Protocol deviations

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s)** | Key | Mock layout |
|---|---|---|---|---|---|
| PRDEVA | Т | Important protocol deviations during the double-blind period | FAS | | LAYPD001 |
| PRDEVI | Т | Protocol deviations<br>leading to exclusion<br>from PPS | FAS | Yes | LAYPD002 |
| PRDEVA | Т | Important protocol deviations during run-in period | RIS | | LAYPD001 |
| PRDEV | L | Listing of protocol deviations | SCR | | LSTCSR021 |

<sup>\*</sup> T = Summary Table; L = Listing.

FAS = Full Analysis Set; PPS = Per-Protocol Set; RIS = Run-in Set; SCR = Screened Set.

## 13.3 Subject characteristics

## 13.3.1 Demographics

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DEMOG | T | Demographic characteristics | FAS,<br>PPS, PK | Yes | LAYDEM001 |
| DEMOG | L | Listing of demographic characteristics | RIS | | LSTCSR041 |
| AGECATEU | Т | EudraCT age categories | FAS | | LAYDEM004 |

<sup>\*</sup> T = Summary Table; L = Listing.

FAS = Full Analysis Set; PK = Pharmacokinetic; PPS = Per-Protocol Set; RIS = Run-in Set.

### 13.3.2 Baseline disease characteristics

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| BASDC | T | Essential hypertension at Screening | FAS,<br>PPS | | LAYMIX001 |
| BASDC | L | Listing of essential hypertension at Screening | SCR | | LSTCSR091 |

\* T = Summary Table; L = Listing. FAS = Full Analysis Set; PPS = Per-Protocol Set; SCR = Screened Set.

### 13.3.3 Other baseline characteristics

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| OBASDC | Т | Height at Screening,<br>weight and BMI at<br>baseline | FAS,<br>PPS, PK | | LAYDEM001 |

<sup>\*</sup> T = Summary Table; L = Listing.

BMI = body mass index; FAS = Full Analysis Set; PK = Pharmacokinetic; PPS = Per-Protocol Set;

# 13.3.4 Medical history

| Output<br>name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| MHSCPR | T | Medical history by<br>primary system organ<br>class (SOC) and<br>preferred term | FAS | | LAYMH001 |
| CDSCPR | T | Concomitant disease by<br>primary system organ<br>class (SOC) and<br>preferred term | FAS | | LAYMH001 |
| PCMHIST | L | Listing of subjects with previous and concomitant medical history | SCR | | LSTCSR043 |

\* T = Summary Table; L = Listing. FAS = Full Analysis Set; SCR = Screened Set; SOC = system organ class.

# 13.3.5 Previous and concomitant therapies

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| PTATCPR | T | Previous therapies by<br>anatomical<br>therapeutic chemical<br>(ATC) class and<br>preferred term | FAS | | LAYCONMED001 |
| DBCATCPR | T | Double-blind<br>treatment concomitant<br>therapies by<br>anatomical<br>therapeutic chemical<br>(ATC) class and<br>preferred term | FAS | | LAYCONMED001 |

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| STCATCPR | T | Study-concomitant<br>therapies by<br>anatomical<br>therapeutic chemical<br>(ATC) class and<br>preferred term | FAS | | LAYCONMED001 |
| PCTHER | L | Listing of subjects with previous and concomitant therapies | RIS | | LSTCSR044 |

<sup>\*</sup> T = Summary Table; L = Listing.

ATC = anatomical therapeutic chemical; FAS = Full Analysis Set; RIS = Run-in Set.

## 13.3.6 Specific previous and concomitant therapies

Not applicable.

## 13.3.7 Other subject characteristics

Not applicable.

# 13.4 Study treatment duration and compliance

## 13.4.1 Study treatment duration

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock<br>layout |
|---|---|---|---|---|---|
| TREXP | T | Double-blind treatment duration | FAS,<br>PPS, SAF | Yes | LAYEX001 |
| TREXP | T | Run-in treatment duration | RIS | | LAYEX001 |
| TREXP | L | Listing of run-in and double-<br>blind treatment duration | RIS | | LSTCSR052 |

<sup>\*</sup> T = Summary Table; L = Listing.

FAS = Full Analysis Set; PPS = Per-Protocol Set; RIS = Run-in Set; SAF = Safety Set.

## 13.4.2 Compliance with study treatment

| Output<br>name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| COMPA | T | Compliance with double-<br>blind study treatment | PPS,<br>FAS | | LAYCAT001 |
| COMPA | Т | Compliance with run-in study treatment | RIS | | LAYCAT001 |
| COMPA | L | Listing of compliance with double-blind study treatment | SAF | | LSTCSR051a |

<sup>\*</sup> T = Summary Table; L = Listing.

FAS = Full Analysis Set; PPS = Per-Protocol Set; RIS = Run-in Set; SAF = Safety Set.

# 13.4.3 Study treatment discontinuation

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| PDISCTR | T | Reasons for premature discontinuation of double-blind study treatment | SAF | Yes | LAYDISP003b |
| PDISCTR | T | Reasons for premature discontinuation of run-in treatment | RIS | | LAYDISP003b |
| PDISCTR | L | Listing of subjects who discontinued treatment | RIS | | LSTCSR012 |

<sup>\*</sup> T = Summary Table; L = Listing. RIS = Run-in Set; SAF = Safety Set.

## 13.4.4 Study treatment adjustments or interruptions

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| TREINT | Т | Reasons for double-blind treatment interruptions | SAF | | LAYMIX001 |
| TREINT | L | Listing of subjects with double-blind treatment interruptions | SAF | | L_TREINT |

<sup>\*</sup> T = Summary Table; L = Listing. SAF = Safety Set.

## 13.5 Study withdrawal

| Output<br>name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| PDISCST | T | Reasons for premature study discontinuation after randomization | RND | | LAYDISP004b |
| PDISCST | T | Reasons for premature study discontinuation before randomization | RIS | | LAYDISP004b |
| PDISC | L | Listing of subjects who discontinued the study prematurely | RIS | | LSTCSR012 |

<sup>\*</sup> T = Summary Table; L = Listing.

RIS = Run-in Set; RND = All Randomized Set.

# 13.6 Primary efficacy analyses

## 13.6.1 Main analysis

All outputs for the main analysis will be based on the PPS. Some outputs will also be generated for the FAS. These are listed in 13.6.2.

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DBP_VIS | T | Mean trough sitting<br>diastolic blood pressure<br>(SiDBP) as measured<br>by OBPM by visit and<br>treatment group | PPS | | LAYCON001 |
| DBP_CHG | T | Change from baseline<br>to post-baseline visits<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) as measured<br>by OBPM by treatment<br>group | PPS | Yes | LAYBASE001 |
| DBP_MCHG | F | Mean change from baseline to post- baseline visits in mean trough sitting diastolic blood pressure (SiDBP) as measured by OBPM by treatment group | PPS | Yes | LAYTIME |
| DBP_CHG | F | Density of change from<br>baseline to post-<br>baseline visits in mean<br>trough sitting diastolic<br>blood pressure<br>(SiDBP) as measured<br>by OBPM by treatment<br>group | PPS | | LAYDENS |
| DBP_MCPMOD1 | T | MCP-Mod test for<br>dose-response in<br>change from baseline<br>to Week 8 in mean<br>trough sitting diastolic<br>blood pressure<br>(SiDBP) | PPS | Yes | LAYMCP1 |

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DBP_MCPMOD2 | T | MCP-Mod estimation<br>of dose-response in<br>change from baseline<br>to Week 8 in mean<br>trough sitting diastolic<br>blood pressure<br>(SiDBP) | PPS | Yes | LAYMCP2 |
| DBP_MCPMOD | F | MCP-Mod estimation<br>of dose-response in<br>change from baseline<br>to Week 8 in mean<br>trough sitting diastolic<br>blood pressure<br>(SiDBP) | PPS | | LAYMCP3 |
| DBP_MCPMOD_SEL | F | MCP-Mod estimation of dose-response in change from baseline to Week 8 in mean trough sitting diastolic blood pressure (SiDBP) - Best fitting model | PPS | Yes | LAYMCP4 |
| DBP_MCPMOD_SEL | T | MCP-Mod estimation<br>of dose-response in<br>change from baseline<br>to Week 8 in mean<br>trough sitting diastolic<br>blood pressure<br>(SiDBP) - Best fitting<br>model | PPS | | LAYMCP5 |

<sup>\*</sup> T = Summary Table; F = Figure.

PPS = Per-Protocol Set; MCP-Mod = Multiple Comparison Procedure – Modeling; OBPM = automated office blood pressure measurement; SiDBP = sitting diastolic blood pressure.

# 13.6.2 Supportive/sensitivity analyses

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock<br>layout |
|---|---|---|---|---|---|
| DBP_VIS | T | Mean trough sitting<br>diastolic blood pressure<br>(SiDBP) as measured by<br>OBPM by visit and<br>treatment group | FAS | | LAYCON0<br>01 |
| DBP_CHG | T | Change from baseline to post-baseline visits in mean trough sitting diastolic blood pressure (SiDBP) as measured by OBPM by treatment group | FAS | Yes | LAYBASE0<br>01 |
| DBP_MCHG | F | Mean change from<br>baseline to post-baseline<br>visits in mean trough<br>sitting diastolic blood<br>pressure (SiDBP) as<br>measured by OBPM by<br>treatment group | PPS | Yes | LAYTIME |
| DBP_CHG | F | Density of change from<br>baseline to post-baseline<br>visits in mean trough<br>sitting diastolic blood<br>pressure (SiDBP) as<br>measured by OBPM by<br>treatment group | FAS | | LAYDENS |
| DBP_MCPMOD 1 | T | MCP-Mod test for dose-<br>response in change from<br>baseline to Week 8 in<br>mean trough sitting<br>diastolic blood pressure<br>(SiDBP) | FAS | Yes | LAYMCP1 |

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock<br>layout |
|---|---|---|---|---|---|
| DBP_MCPMOD 2 | T | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) | FAS | Yes | LAYMCP2 |
| DBP_MCPMOD | F | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) | FAS | | LAYMCP3 |
| DBP_MCPMOD<br>_SEL | F | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) - Best fitting<br>model | FAS | Yes | LAYMCP4 |
| DBP_MCPMOD<br>_SEL | T | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) - Best fitting<br>model | FAS | | LAYMCP5 |
| DBP_ANCOVA | T | ANCOVA for change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) - ACT-132577<br>vs placebo | PPS,<br>FAS | Yes | LAYBETW<br>001 |
| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock<br>layout |
|---|---|---|---|---|---|
| DBP_ANCOVA | F | ANCOVA for change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) - ACT-132577<br>vs placebo | PPS,<br>FAS | Yes | LAYFOR |
| DBP_ANCOVA<br>_L | T | ANCOVA for change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) - Lisinopril vs<br>placebo | PPS,<br>FAS | Yes | LAYBETW<br>001 |
| DBP_MCPMBO<br>CF1 | T | MCP-Mod test for dose-<br>response in change from<br>baseline to Week 8 in<br>mean trough sitting<br>diastolic blood pressure<br>(SiDBP, BOCF) | FAS | | LAYMCP1 |
| DBP_MCPMBO<br>CF2 | T | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP, BOCF) | FAS | | LAYMCP2 |
| DBP_MCPMBO<br>CF | F | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP, BOCF) | FAS | | LAYMCP3 |

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock<br>layout |
|---|---|---|---|---|---|
| DBP_MIXED_W<br>2_W4_W8 | T | Mixed Model for changes<br>from baseline to Weeks 2,<br>4 and 8 in mean trough<br>sitting diastolic blood<br>pressure (SiDBP, OC) -<br>ACT-132577 vs placebo | FAS | | LAYBETW<br>001 |
| DBP_MIXED_W<br>2_W4_W8_MCP<br>1 | | Mixed Model for changes<br>from baseline to Weeks 2,<br>4 and 8 in mean trough<br>sitting diastolic blood<br>pressure (SiDBP, OC) -<br>MCP-Mod test for dose-<br>response at Week 8 | FAS | | LAYMCP1 |
| DBP_MIXED_W<br>2_W4_W8_MCP<br>2 | | Mixed Model for changes<br>from baseline to Weeks 2,<br>4 and 8 in mean trough<br>sitting diastolic blood<br>pressure (SiDBP, OC) -<br>MCP-Mod estimation of<br>dose-response at Week 8 | FAS | | LAYMCP2 |
| DBP_MIXED_W<br>2_W4_W8_L | T | Mixed Model for changes<br>from baseline to Weeks 2,<br>4 and 8 in mean trough<br>sitting diastolic blood<br>pressure (SiDBP, OC) -<br>Lisinopril vs placebo | FAS | | LAYBETW<br>001 |
| DBP_MIXED_A | T | Mixed Model for average | PPS, | | LAYBETW |
| VER8 | | change from baseline to Weeks 2, 4 and 8 in mean trough sitting diastolic blood pressure (SiDBP, OC) - ACT-132577 vs placebo | FAS | | 001 |

| Output | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock<br>layout |
|---|---|---|---|---|---|
| DBP_MIXED_<br>AVER8_MCP1 | T | Mixed Model for average<br>change from baseline to<br>Weeks 2, 4 and 8 in mean<br>trough sitting diastolic<br>blood pressure (SiDBP,<br>OC) - MCP-Mod test for<br>dose-response | PPS,<br>FAS | | LAYMCP1 |
| DBP_MIXED_A<br>VER8_MCP2 | T | Mixed Model for average<br>change from baseline to<br>Weeks 2, 4 and 8 in mean<br>trough sitting diastolic<br>blood pressure (SiDBP,<br>OC) - MCP-Mod<br>estimation of dose-<br>response | PPS,<br>FAS | | LAYMCP2 |
| DBP_MIXED_A<br>VER8_L | T | Mixed Model for average change from baseline to Weeks 2, 4 and 8 in mean trough sitting diastolic blood pressure (SiDBP, OC) - Lisinopril vs placebo | PPS,<br>FAS | | LAYBETW<br>001 |

\* T = Summary Table; L = Listing; F = Figure.

ANCOVA = analysis of covariance; BOCF = baseline observation carried forward; FAS = Full Analysis Set; MCP-Mod = Multiple Comparison Procedure – Modeling; OBPM = automated office blood pressure measurement; PPS = Per-Protocol Set; SiDBP = sitting diastolic blood pressure.

### 13.6.3 Subgroup analyses

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DBP_MCPMOD<br>_AGE | T | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) by Age | PPS | | LAYMCP2 |

| Output<br>name | Display * | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DBP_MCPMOD<br>_AGE | F | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) by Age | PPS | | LAYMCP6 |
| DBP_MCPMOD<br>_SEX | T | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) by Sex | PPS | | LAYMCP2 |
| DBP_MCPMOD<br>_SEX | F | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) by Sex | PPS | | LAYMCP6 |
| DBP_MCPMOD<br>_RACE | T | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) by Race | PPS | | LAYMCP2 |
| DBP_MCPMOD<br>_RACE | F | MCP-Mod estimation of<br>dose-response in change<br>from baseline to Week 8<br>in mean trough sitting<br>diastolic blood pressure<br>(SiDBP) by Race | PPS | | LAYMCP6 |

\* T = Summary Table; F = Figure. MCP-Mod = Multiple Comparison Procedure – Modeling; PPS = Per-Protocol Set; SiDBP = sitting diastolic blood pressure. Age category:  $< 65 \text{ vs} \ge 65 \text{ years}$ .

# 13.7 Secondary efficacy analyses

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| SBP_VIS | T | Mean trough sitting systolic<br>blood pressure (SiSBP) as<br>measured by OBPM by visit<br>and treatment group | PPS,<br>FAS | | LAYCON001 |
| SBP_CHG | Т | Change from baseline to post-<br>baseline visits in mean trough<br>sitting systolic blood pressure<br>(SiSBP) as measured by<br>OBPM by treatment group | PPS,<br>FAS | Yes | LAYBASE00 |
| SBP_MCHG | F | Mean change from baseline to<br>post-baseline visits in mean<br>trough sitting systolic blood<br>pressure (SiSBP) as measured<br>by OBPM by treatment group | PPS,<br>FAS | Yes | LAYTIME |
| SBP_CHG | F | Density of change from<br>baseline to post-baseline visits<br>in mean trough sitting systolic<br>blood pressure (SiSBP) as<br>measured by OBPM by<br>treatment group | PPS,<br>FAS | | LAYDENS |
| SBP_MCPMOD 1 | T | MCP-Mod test for dose-<br>response in change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) | PPS,<br>FAS | Yes | LAYMCP1 |
| SBP_MCPMOD 2 | T | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in sitting<br>systolic blood pressure<br>(SiSBP) | PPS,<br>FAS | Yes | LAYMCP2 |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| SBP_MCPMO<br>D | F | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in sitting<br>systolic blood pressure<br>(SiSBP) | PPS,<br>FAS | | LAYMCP3 |
| SBP_MCPMO<br>D_SEL | F | MCP-Mod estimation of response at study doses in change from baseline to Week 8 in mean trough sitting systolic blood pressure (SiSBP) - Best fitting model | PPS,<br>FAS | Yes | LAYMCP4 |
| SBP_MCPMO<br>D_SEL | F | MCP-Mod estimation of response at study doses in change from baseline to Week 8 in mean trough sitting systolic blood pressure (SiSBP) - Best fitting model | PPS,<br>FAS | | LAYMCP5 |
| SBP_ANCOVA | T | ANCOVA for change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) - ACT-<br>132577 vs placebo | PPS,<br>FAS | Yes | LAYBETW00<br>1 |
| SBP_ANCOVA | F | ANCOVA for change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) - ACT-<br>132577 vs placebo | PPS,<br>FAS | Yes | LAYFOR |
| SBP_ANCOVA _L | T | ANCOVA for change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) - Lisinopril<br>vs placebo | PPS,<br>FAS | Yes | LAYBETW00<br>1 |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| SBP_MIXED_<br>W2_W4_W8 | T | Mixed Model for changes<br>from baseline to Weeks 2, 4<br>and 8 in sitting systolic blood<br>pressure (SiSBP, OC) - ACT-<br>132577 vs placebo | FAS | | LAYBETW00 |
| SBP_MIXED_<br>W2_W4_W8_M<br>CP1 | T | Mixed Model for changes<br>from baseline to Weeks 2, 4<br>and 8 in sitting systolic blood<br>pressure (SiSBP, OC) - MCP-<br>Mod test for dose-response at<br>Week 8 | FAS | | LAYMCP1 |
| SBP_MIXED_<br>W2_W4_W8_M<br>CP2 | T | Mixed Model for changes<br>from baseline to Weeks 2, 4<br>and 8 in sitting systolic blood<br>pressure (SiSBP, OC) - MCP-<br>Mod estimation of dose-<br>response at Week 8 | FAS | | LAYMCP2 |
| SBP_MIXED_<br>W2_W4_W8_L | T | Mixed Model for changes<br>from baseline to Weeks 2, 4<br>and 8 in mean trough sitting<br>systolic blood pressure<br>(SiSBP, OC) - Lisinopril vs<br>placebo | FAS | | LAYBETW00 |
| SBP_MIXED_<br>AVER8 | T | Mixed Model for changes<br>from baseline to Weeks 2, 4<br>and 8 in sitting systolic blood<br>pressure (SiSBP, OC) - ACT-<br>132577 vs placebo | PPS,<br>FAS | | LAYBETW00<br>1 |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| SBP_MIXED_<br>AVER8_MCP1 | T | Mixed Model for average<br>change from baseline to<br>Weeks 2, 4 and 8 in sitting<br>systolic blood pressure<br>(SiSBP, OC) - MCP-Mod test<br>for dose-response | PPS,<br>FAS | | LAYMCP1 |
| SBP_MIXED_<br>AVER8_MCP2 | T | Mixed Model for average<br>change from baseline to<br>Weeks 2, 4 and 8 in sitting<br>systolic blood pressure<br>(SiSBP, OC) - MCP-Mod<br>estimation of dose-response | PPS,<br>FAS | | LAYMCP2 |
| SBP_MIXED_<br>AVER8_L | T | Mixed Model for average change from baseline to Weeks 2, 4 and 8 in mean trough sitting systolic blood pressure (SiSBP, OC) - Lisinopril vs placebo | PPS,<br>FAS | | LAYBETW00<br>1 |
| SBP_MCPMOD<br>_AGE | T | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) by Age | PPS | | LAYMCP2 |
| SBP_MCPMOD<br>_AGE | F | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) by Age | PPS | | LAYMCP6 |
| SBP_MCPMOD<br>_SEX | T | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) by Sex | PPS | | LAYMCP2 |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| SBP_MCPMOD<br>_SEX | F | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) by Sex | PPS | | LAYMCP6 |
| SBP_MCPMOD<br>_RACE | T | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) by Race | PPS | | LAYMCP2 |
| SBP_MCPMOD<br>_RACE | F | MCP-Mod estimation of dose-<br>response in change from<br>baseline to Week 8 in mean<br>trough sitting systolic blood<br>pressure (SiSBP) by Race | PPS | | LAYMCP6 |
| COR_DBP_SB P | F | Correlation between change<br>from baseline in Diastolic and<br>Systolic Blood Pressure by<br>Visit and Treatment Group | PPS | | LAYCORR |
| CRR_DBP | T | Control and response rates at<br>Week 8 for sitting diastolic<br>blood pressure (SiDBP) as<br>measured by OBPM | PPS | | LAYCAT002 |
| CR_DBP_LOG<br>REG1 | T | Logistic regression for control<br>rates at Week 8 for sitting<br>diastolic blood pressure<br>(SiDBP) as measured by<br>OBPM < 90 mmHg | PPS | | LAYLOGR |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| CR_DBP_LOG<br>REG2 | T | Logistic regression for control<br>rates at Week 8 for sitting<br>diastolic blood pressure<br>(SiDBP) as measured by<br>OBPM < 85 mmHg | PPS | | LAYLOGR |
| CR_DBP_LOG<br>REG_MCP1 | T | Logistic regression for control<br>rates at Week 8 for sitting<br>diastolic blood pressure<br>(SiDBP) as measured by<br>OBPM < 90 mmHg - MCP-<br>Mod test for dose-response | PPS | | LAYMCP1 |
| CR_DBP_LOG<br>REG_MCP2 | T | Logistic regression for control<br>rates at Week 8 for sitting<br>diastolic blood pressure<br>(SiDBP) as measured by<br>OBPM < 90 mmHg - MCP-<br>Mod estimation of dose-<br>response | PPS | | LAYMCP2 |
| RR_DBP_LOG<br>REG | T | Logistic regression for<br>response rates at Week 8 for<br>sitting diastolic blood pressure<br>(SiDBP) as measured by<br>OBPM | PPS | | LAYLOGR |
| CRR_SBP | Т | Control and response rates at<br>Week 8 for sitting systolic<br>blood pressure (SiSBP) as<br>measured by OBPM | PPS | | LAYCAT002 |
| CR_SBP_LOG<br>REG1 | T | Logistic regression for control rates at Week 8 for sitting systolic blood pressure (SiSBP) as measured by OBPM < 140 mmHg | PPS | | LAYLOGR |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| CR_SBP_LOG<br>REG2 | T | Logistic regression for control<br>rates at Week 8 for sitting<br>systolic blood pressure<br>(SiSBP) as measured by<br>OBPM < 135 mmHg | PPS | | LAYLOGR |
| CR_SBP_LOG<br>REG_MCP1 | T | Logistic regression for control<br>rates at Week 8 for sitting<br>systolic blood pressure<br>(SiSBP) as measured by<br>OBPM < 140 mmHg - MCP-<br>Mod test for dose-response | PPS | | LAYMCP1 |
| CR_SBP_LOG<br>REG_MCP2 | T | Logistic regression for control<br>rates at Week 8 for sitting<br>systolic blood pressure<br>(SiSBP) as measured by<br>OBPM < 140 mmHg - MCP-<br>Mod estimation of dose-<br>response | PPS | | LAYMCP2 |
| RR_SBP_LOG<br>REG | T | Logistic regression for<br>response rates at Week 8 for<br>sitting systolic blood pressure<br>(SiSBP) as measured by<br>OBPM | PPS | | LAYLOGR |
| 24H_DBP_CH<br>G | T | Change from baseline to Week<br>8 in 24-hour mean diastolic<br>blood pressure (DBP) as<br>measured by ABPM by<br>treatment group | PPS | | LAYBASE00 |
| 24H_DBP_AN<br>COVA | T | ANCOVA for change from<br>baseline to Week 8 in 24-hour<br>mean diastolic blood pressure<br>(DBP) as measured by ABPM<br>- ACT-132577 vs Placebo | PPS | Yes | LAYBETW00 |

| Output name | Display * | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| 24H_DBP_AN<br>COVA_L | T | ANCOVA for change from<br>baseline to Week 8 in 24-hour<br>mean diastolic blood pressure<br>(DBP) as measured by ABPM<br>- Lisinopril vs Placebo | PPS | Yes | LAYBETW00 |
| 24H_SBP_CHG | T | Change from baseline to Week<br>8 in 24-hour mean systolic<br>blood pressure (SBP) as<br>measured by ABPM by<br>treatment group | PPS | | LAYBASE00 |
| 24H_SBP_ANC<br>OVA_L | T | ANCOVA for change from<br>baseline to Week 8 in 24-hour<br>mean systolic blood pressure<br>(SBP) as measured by ABPM<br>- Lisinopril vs Placebo | PPS | Yes | LAYBETW00 |
| OBPM | L | Listing of mean trough sitting diastolic (SiDBP), mean trough sitting systolic blood pressure (SiSBP) and pulse rate measured by OBPM with control and response rates | FAS | | L_OBPM |
| ABPM24_DBP<br>_BAS | F | Mean diastolic blood pressure<br>(DBP) per hour as measured<br>by ABPM at baseline | PPS | | LAY_ABPM |
| ABPM24_DBP<br>_WK8 | F | Mean diastolic blood pressure<br>(DBP) per hour as measured<br>by ABPM at Week 8 | PPS | | LAY_ABPM |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| ABPM24_DBP<br>_WK8_DIF | F | Difference in mean diastolic<br>blood pressure (DBP) per hour<br>as measured by ABPM | PPS | | LAY_ABPM |
| ABPM24_DBP<br>_TTPR | T | Trough to peak ratio for diastolic blood pressure (DBP) measured by ABPM | PPS | | LAY_TTPR |
| ABPM24_SBP_<br>BAS | F | Mean systolic blood pressure<br>(SBP) per hour as measured by<br>ABPM at baseline | PPS | | LAY_ABPM |
| ABPM24_SBP_<br>WK8 | F | Mean systolic blood pressure<br>(SBP) per hour as measured by<br>ABPM at Week 8 | PPS | | LAY_ABPM |
| ABPM24_SBP_<br>WK8_DIF | F | Difference in mean systolic<br>blood pressure (SBP) per hour<br>as measured by ABPM | PPS | | LAY_ABPM |
| ABPM24_SBP_<br>TTPR | T | Trough to peak ratio for systolic blood pressure (SBP) measured by ABPM | PPS | | LAY_TTPR |

<sup>\*</sup> T = Summary Table; F = Figure.

ABPM = ambulatory blood pressure monitoring; ANCOVA = analysis of covariance; DBP = diastolic blood pressure; FAS = Full Analysis Set; MCP-Mod = Multiple Comparison Procedure – Modeling; OBPM = automated office blood pressure measurement; PPS = Per-Protocol Set; SBP = systolic blood pressure; SiDBP = sitting diastolic blood pressure; SiSBP = sitting systolic blood pressure.

ABPM analyses are based on the subset of the PPS described in Section 5.5.

Age category:  $< 65 \text{ vs} \ge 65 \text{ years}.$ 

## 13.8 Other efficacy analyses

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DAY_DBP_<br>CHG | T | Change from baseline to<br>Week 8 in 24-hour mean<br>daytime diastolic blood<br>pressure (DBP) as measured<br>by ABPM by treatment group | PPS | | LAYBASE0<br>01 |

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DAY_DBP_<br>ANCOVA | T | ANCOVA for change from<br>baseline to Week 8 in mean<br>daytime diastolic blood<br>pressure (DBP) as measured<br>by ABPM | PPS | | LAYBETW0<br>01 |
| NIGHT_DBP<br>_CHG | T | Change from baseline to<br>Week 8 in 24-hour mean<br>night time diastolic blood<br>pressure (DBP) as measured<br>by ABPM by treatment group | PPS | | LAYBASE0<br>01 |
| NIGHT_DBP<br>_ANCOVA | T | ANCOVA for change from<br>baseline to Week 8 in mean<br>night time diastolic blood<br>pressure (DBP) as measured<br>by ABPM | PPS | | LAYBETW0<br>01 |
| DAY_SBP_<br>CHG | T | Change from baseline to<br>Week 8 in 24-hour mean<br>daytime systolic blood<br>pressure (DBP) as measured<br>by ABPM by treatment group | PPS | | LAYBASE0<br>01 |
| DAY_SBP_<br>ANCOVA | T | ANCOVA for change from<br>baseline to Week 8 in mean<br>daytime systolic blood<br>pressure (SBP) as measured<br>by ABPM | PPS | | LAYBETW0<br>01 |
| NIGHT_SBP<br>_CHG | T | Change from baseline to<br>Week 8 in 24-hour mean<br>night time systolic blood<br>pressure (SBP) as measured<br>by ABPM by treatment group | PPS | | LAYBASE0<br>01 |

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| NIGHT_SBP<br>_ANCOVA | Т | ANCOVA for change from<br>baseline to Week 8 in mean<br>night time systolic blood<br>pressure (SBP) as measured<br>by ABPM | PPS | | LAYBETW0<br>01 |
| MIXED_DB<br>P_W2_W4_<br>W8_W10 | T | Mixed model for changes<br>from baseline to Weeks 2, 4,<br>8 and 10 in mean trough<br>sitting diastolic blood<br>pressure (SiDBP, OC) as<br>measured by OBPM | PPS | | LAYBETW0<br>01 |
| MIXED_SBP<br>_W2_W4_W<br>8_W10 | T | Mixed model for changes<br>from baseline to Weeks 2, 4,<br>8 and 10 in mean trough<br>sitting systolic blood pressure<br>(SiSBP, OC) as measured by<br>OBPM | PPS | | LAYBETW0<br>01 |
| ABPM | L | Listing of individual diastolic<br>and systolic blood pressure<br>measured by ABPM | FAS | | LSTCSR09<br>32 |
| DN_ABPM | L | Listing of 24-hour mean,<br>daytime mean and night time<br>mean diastolic and systolic<br>blood pressure measured by<br>ABPM | FAS | | LSTCSR09<br>32 |

<sup>\*</sup> T = Summary Table; L = Listing.

ABPM = ambulatory blood pressure monitoring; ANCOVA = analysis of covariance; DBP = diastolic blood pressure; FAS = Full Analysis Set; MCP-Mod = Multiple Comparison Procedure – Modeling; OBPM = automated office blood pressure measurement; PPS = Per-Protocol Set; SBP = systolic blood pressure; SiDBP = sitting diastolic blood pressure; SiSBP = sitting systolic blood pressure.

ABPM analyses are based on the subset of PPS subjects describe d in Section 5.5.

# 13.9 Safety analyses

## 13.9.1 Adverse events

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| AEOV | Т | Overview of double-blind<br>treatment-emergent adverse<br>events (AEs) | SAF | Yes | LAYAE004 |
| TEAESCPR | T | Double-blind treatment-<br>emergent adverse events<br>(AEs) by primary system<br>organ class (SOC) and<br>preferred term | SAF | | LAYAE001 |
| TEAEPR | Т | Double-blind treatment-<br>emergent adverse events<br>(AEs) by preferred term | SAF | | LAYAE002 |
| TEAERESC<br>PR | T | Double-blind treatment-<br>emergent adverse events<br>(AEs) related to study<br>treatment by primary system<br>organ class (SOC) and<br>preferred term | SAF | | LAYAE001 |
| TEAEREPR | T | Double-blind treatment-<br>emergent adverse events<br>(AEs) <i>related to study</i><br><i>treatment</i> by preferred term | SAF | | LAYAE002 |
| TEAEPRIN | Т | Double-blind treatment-<br>emergent adverse events<br>(AEs) by maximum intensity | SAF | | LAYAE003 |
| AEOV | Т | Overview of run-in<br>treatment-emergent adverse<br>events (AEs) | RIS | | LAYAE004 |
| TEAEPR | Т | Run-in treatment-emergent<br>adverse events (AEs) by<br>preferred term | RIS | | LAYAE002 |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| AE | L | Listing of adverse events | RIS | | LSTCSR071 |


AE = adverse event; RIS = Run-in Set; SAF = Safety Set.

#### 13.9.2 **Deaths**

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| DEATH | L | Listing of deaths | SAF | | LSTCSR072 |

(AEs)

### 13.9.3 Serious adverse events

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| TESAESCPR | T | Double-blind treatment-<br>emergent serious<br>adverse events (SAEs)<br>by primary system organ<br>class (SOC) and<br>preferred term | SAF | Yes | LAYAE001 |
| TESAEPR | T | Double-blind treatment-<br>emergent serious<br>adverse events (SAEs)<br>by preferred term | SAF | | LAYAE002 |
| TESAERESCPR | T | Double-blind treatment-<br>emergent serious<br>adverse events (SAEs)<br>related to study<br>treatment by preferred<br>term | SAF | | LAYAE002 |

<sup>\*</sup> T = Summary Table; L = Listing.

<sup>\*</sup> L= Listing, SAF=Safety set.

| _ | | | |
|-----|-------|------|-------------|
| 5 N | Λav 2 | 2017 | page 89/110 |

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| TESAEPR | T | Run-in treatment-<br>emergent serious<br>adverse events (SAEs)<br>by preferred term | RIS | | LAYAE002 |
| SAE | L | Listing of serious adverse events (SAEs) | RIS | | LSTCSR071 |

<sup>\*</sup> T = Summary Table; L = Listing.

### 13.9.4 Adverse events leading to treatment discontinuation

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock<br>layout(AEs) |
|---|---|---|---|---|---|
| TEAEPDSCPR | T | Double-blind treatment-<br>emergent adverse events<br>(AEs) leading to premature<br>discontinuation of study<br>treatment by primary<br>system organ class (SOC)<br>and preferred term | SAF | Yes | LAYAE001 |
| TEAEPDPR | T | Double-blind treatment-<br>emergent adverse events<br>(AEs) leading to premature<br>discontinuation of study<br>treatment by preferred term | SAF | | LAYAE002 |
| TEAEPDPR | T | Run-in treatment-emergent<br>adverse events (AEs)<br>leading to premature<br>discontinuation of study<br>treatment by preferred term | RIS | | LAYAE002 |
| AEPD | L | Listing of adverse events (AEs) leading to premature discontinuation of study treatment | SCR | | LSTCSR071 |

RIS = Run-in Set; SAE = serious adverse event; SAF = Safety Set; SOC = system organ class.

<sup>\*</sup> T = Summary Table; L = Listing. AE = adverse event; RIS = Run-in Set; SAF = Safety Set; SOC = system organ class.

# 13.10 Electrocardiogram (ECG)

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| ECG_CHG | T | ECG parameters: changes from baseline to end of double-blind treatment | SAF | | LAYBASE00 |
| ECGQTCP<br>T | T | Number of subjects with<br>double-blind treatment-<br>emergent ECG abnormalities<br>(based on Fridericia's formula) | SAF | | LAYECG001 |
| ECGMA | L | Listing of 12-lead ECG variables in subjects with at least one double-blind treatment-emergent ECG abnormalities | SAF | | LSTCSR0931 |
| ECG | L | Listing of 12-lead ECG variables and abnormalities | SCR | | LSTCSR093 |

\* T = Summary Table; L = Listing. ECG = electrocardiogram; SAF = Safety Set; SCR = Screened Set.

# 13.11 Laboratory tests

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| HEMAV_VIS | T | Hematology<br>parameters:<br>absolute values by<br>visit | SAF | | LAYLAB003a |
| HEM_CHG | T | Hematology<br>parameters:<br>changes from<br>baseline to<br>post-baseline visits | SAF | Yes | LAYLAB002a |

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| HEM_CHG | F | Mean change from<br>baseline to post-<br>baseline visits in<br>hemoglobin by<br>treatment group | SAF | | LAYTIME |
| CHEAV_VIS | T | Chemistry parameters: absolute values by visit | SAF | | LAYLAB003a |
| CHE_CHG | T | Chemistry parameters: changes from baseline to post-baseline visits | SAF | | LAYLAB002a |
| UACRAV_VIS | Т | Urine parameter:<br>UACR absolute<br>values by visit | SAF | | LAYLAB003a |
| UACR_CHG | Т | Urine parameter:<br>UACR changes<br>from baseline to<br>post-baseline visits | SAF | Yes | LAYLAB002a |
| | T | Definition of<br>abnormal<br>laboratory values | NA | | |
| HEM_TEMA | T | Hematology<br>parameters:<br>treatment-emergent<br>marked<br>abnormalities | SAF | | LAYLAB001 |
| CHE_TEMA | Т | Chemistry parameters: treatment-emergent marked abnormalities | SAF | | LAYLAB001 |
| CHE_ALT_BIL | T | Number of subjects with ALT > 3 × ULN and bilirubin > 2 × ULN | SAF | | LAYCAT002 |

| Output name | Display* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| LABMLA | L | Listing of<br>definitions of<br>marked laboratory<br>abnormality | - | | L_LABMLA |
| LAB | L | Listing of individual laboratory measurements (SI units) | SCR | | LSTCSR081 |
| HEM_CHG | F | Density of change<br>from baseline to<br>post-baseline visits<br>in hemoglobin by<br>treatment group | SAF | | LAYDENS |
| HEM_MCPMOD1 | T | MCP-Mod test for<br>dose-response in<br>change from<br>baseline to Week 8<br>in hemoglobin | SAF | | LAYMCP1 |
| HEM_MCPMOD2 | T | MCP-Mod<br>estimation of<br>dose-response in<br>change from<br>baseline to Week 8<br>in hemoglobin | SAF | | LAYMCP2 |
| HEM_MCPMOD | F | MCP-Mod<br>estimation of dose-<br>response in change<br>from baseline to<br>Week 8 in<br>hemoglobin | SAF | | LAYMCP3 |

\* T = Summary Table; L = Listing; F = Figure. ALT = alanine aminotransferase; MCP-Mod = Multiple Comparison Procedure – Modeling; SAF = Safety Set; SCR = Screened Set; SI = Standard International; UACR = urine albumin-to-creatinine ratio; ULN = upper limit of normal; NA = not applicable.

# 13.12 Physical examination, vital signs and body weight

| Output name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| VSW_VI | T | Pulse rate and body weight: values by visit | SAF | | LAYBASE0<br>01 |
| VSW_C<br>HG | Т | Pulse rate and body weight:<br>changes from baseline to<br>post-baseline visit | SAF | Yes | LAYBASE0<br>01 |
| VSW_C<br>HG | F | Mean change from baseline to post-baseline visits in body weight by treatment group | SAF | | LAYTIME |
| VSW_C<br>HG | F | Density of change from baseline<br>to post-baseline visits in body<br>weight by treatment group | SAF | | LAYDENS |
| VSW | L | Listing of pulse rate and body weight | SCR | | LSTCSR091 |
| PHYSF | L | Listing of physical findings | SCR | | LSTCSR094 |
| WGT_M<br>CPMOD<br>1 | Т | MCP-Mod test for dose-response in change from baseline to Week 8 in body weight | SAF | | LAYMCP1 |
| WGT_M<br>CPMOD<br>2 | Т | MCP-Mod estimation of dose-<br>response in change from baseline<br>to Week 8 in body weight | SAF | | LAYMCP2 |
| WGT_M<br>CPMOD | F | MCP-Mod estimation of dose-<br>response in change from baseline<br>to Week 8 in body weight | SAF | | LAYMCP3 |

\* T = Summary Table; L = Listing; F = Figure. MCP-Mod = Multiple Comparison Procedure - Modeling; SAF = Safety Set; SCR = Screened Set.

### 13.13 Other safety variables

Not applicable.

#### 13.14 Other evaluations

#### 13.14.1 PK

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| PRDEVP<br>K | T | Protocol deviations leading to exclusion from PK set | FAS | | LAYPD002 |
| PK1 | T | Summary of ACT 132577 plasma concentrations in the double-blind treatment period | PK | | LAYPKPD |
| PKAGE | T | Summary of ACT 132577 plasma concentrations in the double-blind treatment period - by age category | PK | | LAYPKSUB |
| PKGEN | T | Summary of ACT 132577 plasma concentrations in the double-blind treatment period - by gender | PK | | LAYPKSUB |
| PKRAC<br>E | T | Summary of ACT 132577 plasma concentrations in the double-blind treatment period - by race | PK | | LAYPKSUB |
| PKTRO<br>UGH | L | ACT-132577 plasma<br>concentrations in the<br>double-blind treatment period | PK | | LSTCSR051<br>b |

<sup>\*</sup> T = Summary Table, L = Listing.

### 13.14.2 PD

| Output<br>name | Display<br>* | Title (Description) | Analysis set(s) | Key | Mock layout |
|---|---|---|---|---|---|
| PD1 | T | Summary of trough ET-1 plasma<br>concentrations in the<br>double-blind treatment period | PK | | LAYPKPD |
| PDTRO<br>UGH | L | Listing of individual trough ET-1 plasma concentrations in the double-blind treatment period | PK | | LSTCSR051<br>b |

<sup>\*</sup> T = Summary Table, L = Listing.

PK = pharmacokinetic.

ET = endothelin; PK = pharmacokinetic.

#### 14 REFERENCES

- [D-16.063] A multi-center, double-blind, double-dummy, randomized, placebo- and active-reference, parallel group, Phase 2 dose-finding study with ACT-132577 in subjects with essential hypertension (grade 1 and 2). Actelion Pharmaceuticals Ltd; Protocol AC-080A201, 30 May 2016.
- [Bornkamp 2016] Bornkamp B, Pinheiro J, Bretz F. Planning and analyzing dose finding experiments. 2016. Available from: cran.r-project.org/web/packages/DoseFinding. Accessed on: 27 July 2016.
- [Bretz 2005] Bretz F, Pinheiro JC, Branson M. Combining multiple comparisons and modeling techniques in dose-response studies. Biometrics. 2005;61(3):738-48.
- [EMA 2010] European Medicines Agency, EMA/CPMP/EWP/1776/99 Rev. 1. Guideline on Missing Data in Confirmatory Clinical Trials. Available from: http://www.ema.europa.eu/docs/en GB/document library/Scientific guideline/201 0/09/WC500096793.pdf
- [EMA 2014] European Medicines Agency, EMA/CHMP/SAWP/757052/2013. Qualification Opinion of MCP-Mod as an efficient statistical methodology for model-based design and analysis of Phase II dose finding studies under model uncertainty.

Available from:

- http://www.ema.europa.eu/docs/en GB/document library/Regulatory and procedu ral guideline/2014/02/WC500161027.pdf
- [FDA 2007]. Food and Drug Administration, Center for Drug Evaluation and Research. Medical reviews of Aliskiren.

Available from:

- https://www.accessdata.fda.gov/drugsatfda docs/nda/2007/021985s000toc.cfm
- [Leung 2016]. Leung AA, Nerenberg K, Daskalopoulou SS, McBrien K, Zarnke KB, Dasgupta K, et al. Hypertension Canada's 2016 Canadian Hypertension Education Program Guidelines for Blood Pressure Measurement, Diagnosis, Assessment of Risk, Prevention, and Treatment of Hypertension. Canadian Journal of Cardiology. 2016;32:569-88.
- [O'Brien 2013] O'Brien E, Parati G, Stergiou G. Ambulatory blood pressure measurement - What is the international consensus. Hypertension. 2013;62:988-94.
- [Omboni 1995] Omboni S, Parati G, Zanchetti A, Mancia G. Calculation of trough: peak ratio of antihypertensive treatment from ambulatory blood pressure: methodological aspects. Journal of Hypertension 1995;13:1105-12.

- [Pinheiro 2006] Pinheiro J, Bornkamp B, Bretz F. Design and analysis of dose-finding studies combining multiple comparisons and modeling procedures. J Biopharm Stat. 2006;16(5):639-56.
- [Pinheiro 2014] Pinheiro J, Bornkamp B, Glimm E, Bretz F. Model-based dose finding under model uncertainty using general parametric models. Statistics in Medicine 2014;33(10):1646-61.

# 15 APPENDICES

#### **Protocol synopsis** A.

| TITLE | Multi-center, double-blind, double-dummy, randomized, placebo- and active-reference, parallel group, Phase 2 dose-finding study with ACT-132577 in subjects with essential hypertension (grade 1 and 2) |
|---|---|
| OBJECTIVES | Primary objective The primary objective of the study is to explore the dose-response of ACT-132577 on diastolic blood pressure (DBP) in subjects with essential hypertension (grade 1 and 2). |
| | <ul> <li>Secondary objectives</li> <li>Evaluate the dose-response of ACT-132577 on:</li> <li>Systolic blood pressure (SBP)</li> <li>Control and response rates of blood pressure (BP)</li> <li>24-h ambulatory blood pressure monitoring (ABPM)</li> </ul> |
| | Evaluate the safety and tolerability of a once a day oral regimen of 4 doses of ACT-132577. |
| | Other objectives Other objectives are described in Section 2.3. |
| DESIGN | Prospective, multi-center, double-blind, double-dummy, randomized, placebo- and active-reference, parallel group, Phase 2 dose-finding study |
| PERIODS | Pre-screening: |
| | Subjects without a confirmation of hypertension are offered the possibility of having their BP measured (at trough if subjects are on antihypertensive treatment) with an automated office BP device before entering the screening period. |
| | Screening: |
| | Visit 1 (screening period) lasts up to 72 h to allow for informed consent to be obtained and study assessments to be performed (e.g., laboratory tests) to determine whether the subject is eligible for the study. |
| | <b>Run-in Period (Period I)</b> is a single-blind (SB) placebo period of between 4 to 6 weeks. |
| | It commences at the end of Visit 1 and ends at Visit 4 / Randomization (after completion of the baseline 24-h ABPM |

| | recording on the last dose of SB study treatment (placebo). |
|---|---|
| | For subjects on anti-hypertensive treatment at first visit (Visit 1) the SB placebo period is 6 weeks including a 2-week wash-out period for anti-hypertensive treatment. |
| | For anti-hypertensive treatment naïve subjects at first visit, the SB placebo period is 4 weeks. Visit 1 is combined with Visit 2. |
| | <b>Treatment Period (Period II)</b> is a double-blind (DB) treatment period of 8 weeks which starts at Visit 4 / Randomization with the first dose of DB study treatment and ends at Visit 7 / Part 2 (after completion of 24-h ABPM recording on the last dose of DB study treatment). |
| | Withdrawal Period (Period III) is an SB placebo period of 2 weeks which starts at Visit 7 / Part 2 with the first dose of SB study treatment (placebo) and ends at Visit 8 (withdrawal End-of-Treatment [WD-EOT]). |
| | <b>Follow-up Period</b> starts after the last dose of withdrawal study treatment and ends at least 2 weeks thereafter, by the follow-up telephone call, or follow-up visit only for women of childbearing potential to perform a pregnancy test at the site. |
| | <b>End-of-Study (EOS)</b> for a single subject is defined as the date of the follow-up telephone call or the date of the follow-up visit. |
| | If a subject withdraws consent and does not wish to participate in further visits, the date of consent withdrawal is EOS for this subject. If a subject is declared lost to follow-up [see also Section 9.2] date of last contact is EOS for this subject. |
| | The overall study is considered completed when all subjects have completed their safety follow-up telephone call or follow-up visit. |
| PLANNED DURATION | Approximately 16 months from First subject first visit (i.e., Screening Visit) to Last subject last visit (i.e., 30-day follow-up telephone call / visit). |
| SITE(S)<br>/ COUNTRY(IES) | Approximately 100 sites in 3 to 4 countries in North America and Israel (planned). |
| SUBJECTS / GROUPS | Approximately 1000 subjects will be enrolled in the SB placebo run-in period, in order to have at least 540 subjects randomized in 6 groups (90 subjects per group) in a 1:1:1:1:1: |

| | ratio. |
|---|---|
| | At least 420 subjects (70 per group) are expected to complete the trial. |
| INCLUSION CRITERIA | This study will enroll adult male and female subjects aged 18 to 75 years with mild-to-moderate (grade 1 and 2) essential hypertension with or without ongoing anti-hypertensive treatment. |
| | Women of childbearing potential must have a negative pregnancy test at screening and randomization, and must agree to use reliable methods of contraception from Visit 1 (Screening) until up to 30 days after DB study treatment discontinuation. |
| | Eligible subjects must be able and willing to give informed consent for participation in the clinical study. |
| | For the complete list of inclusion criteria, please see Section 4.3. |
| EXCLUSION CRITERIA | Subjects with severe hypertension (grade 3) or secondary hypertension. |
| | Subjects with clinically relevant medical or surgical conditions that, in the opinion of the investigator, would put the subject at risk by participating in the study. |
| | For the complete list of exclusion criteria, please see Section 4.4. |
| STUDY TREATMENTS | <b>Investigational treatment</b> ACT-132577 5 mg, 10 mg (2 × 5 mg), 25 mg, and 50 mg administered as capsules orally once a day (o.d.) in the morning irrespective of food intake during the DB treatment period. |
| | Comparator Lisinopril is used as active reference drug. It is administered as 20 mg capsules orally o.d. in the morning irrespective of food intake during the DB treatment period. |
| | Placebo Placebo matching ACT-132577 and placebo matching lisinopril capsules will be administered concomitantly orally o.d. during the SB placebo run-in period and SB placebo withdrawal period to all subjects and during the DB treatment period to those subjects who have been randomized to the |

| | placebo group. |
|---|---|
| CONCOMITANT<br>THERAPY | Allowed concomitant therapy Treatments considered necessary for the subject's wellbeing and not categorized as prohibited concomitant medications are allowed during the study. |
| | Intermittent use of topical/nasal corticosteroid applications are allowed during the study. |
| | In addition, the following therapies are allowed with the provision that they have been initiated at least one month prior to the Screening visit (Visit 1) and that the dose is kept stable until the WD-EOT visit (i.e., Visit 8): |
| | Hormonal contraceptives. |
| | Estrogen-replacement treatment. |
| | Non-steroidal anti-inflammatory drugs (e.g., low dose acetylsalicylic acid for prevention of cardiovascular disease). |
| | • <u>Selective serotonin reuptake inhibitors</u> and anxiolytics. |
| | Forbidden concomitant therapy The following concomitant therapies are forbidden from Screening visit (i.e., Visit 1) until the WD-EOT visit (i.e., Visit 8), see Section 5.2.4: |
| | • Any drug, including ophthalmic preparation, which may affect blood pressure, see Appendix 3. Endothelin receptor antagonists (ERAs) and PDE5 inhibitors. |
| | • Strong inhibitors or inducers of cytochrome P450 3A4 isoenzyme (CYP3A4), see Appendix 4. |
| ENDPOINTS | Primary efficacy endpoint(s) The primary efficacy variable is the change from baseline to Week 8 of DB treatment period (Period II) in mean trough sitting DBP (SiDBP), measured by office blood pressure measurement (OBPM). |
| | Secondary efficacy endpoints Secondary efficacy variables include (measured by OBPM, unless specified otherwise): |
| | • Change from baseline to Week 8 of DB treatment period (Period II) in mean trough sitting systolic BP (SiSBP); |
| | • Control and response rates at Week 8 of DB treatment |

| | period (Period II) based on trough SiDBP [defined as in Section 7.2.1.1]; |
|---|---|
| | • Control and response rates at Week 8 of DB treatment period (Period II) based on trough SiSBP [defined as in Section 7.2.1.1]; |
| | • Change from baseline to Week 8 of DB treatment period (Period II) in 24-h mean DBP, measured by ABPM; |
| | • Change from baseline to Week 8 of DB treatment period (Period II) in 24-h mean SBP, measured by ABPM; |
| | Trough to peak ratio for DBP based on ABPM. |
| | Other efficacy endpoints Other efficacy endpoints are described in Section 6.1.3. |
| | <ul> <li>Safety endpoints</li> <li>Treatment-emergent adverse events (AEs);</li> <li>AEs leading to premature discontinuation of study</li> </ul> |
| | treatment; |
| | • Treatment-emergent deaths; |
| | Treatment-emergent serious adverse events; |
| | • Treatment-emergent ECG abnormalities; |
| | Treatment-emergent marked laboratory abnormalities; |
| | • Changes from baseline to Weeks 2, 4 and 8 of DB treatment period (Period II) in laboratory parameters; |
| | • Changes from baseline to Weeks 4 and 8 of DB treatment period (Period II) in ECG parameters (PR, QRS, QT, QTcB, QTcF); |
| | • Changes from baseline to Weeks 2, 4 and 8 of DB treatment period (Period II) in body weight and heart rate. |
| | See Section 10.1.1 for definition of 'treatment-emergent'. |
| | Pharmacokinetic/pharmacodynamic endpoints Pharmacokinetic / pharmacodynamic endpoints are described in Section 6.3. |
| ASSESSMENTS | Refer to the schedule of assessments in Table 1. |
| STATISTICAL<br>METHODOLOGY | The Full Analysis Set (FAS) includes all subjects randomized to a study treatment, who have a baseline mean trough SiDBP. |
| | The Per-Protocol Set (PPS) includes all subjects from the FAS |

who have a mean trough SiDBP at Week 8 of DB treatment period (Period II) and do not have any major protocol deviation. Major protocol deviations will be described in the Statistical Analysis Plan.

The Safety Set includes all subjects who received at least one dose of study treatment in DB treatment period (Period II).

#### Statistical hypotheses

The null hypothesis to be tested is that there is no dose-response for the primary endpoint.

$$H_0$$
:  $\mu_0 = \mu_1 = \mu_2 = \mu_3 = \mu_4$ 

Here,  $\mu_i$  denotes the mean change from baseline to Week 8 in mean trough SiDBP ( $\mu$ ) for ACT-132577 dose (i) (where i = 0 corresponds to placebo). A value of  $\mu_i < 0$  corresponds to a decrease in SiDBP.

The alternative hypothesis is that there is a monotonic dose-response for the primary endpoint.

H<sub>1</sub>: 
$$\mu_0 \ge \mu_1 \ge \mu_2 \ge \mu_3 \ge \mu_4$$
 and  $\mu_i > \mu_j$  for at least one  $i > j$  or  $\mu_0 \le \mu_1 \le \mu_2 \le \mu_3 \le \mu_4$  and  $\mu_i < \mu_j$  for at least one  $i > j$ 

Note that larger values of  $\mu_i$  –corresponding to less decrease (or more increase) from baseline to Week 8 in mean trough SiDBP with increasing dose of ACT-132577– are less favorable. The first part of the alternative hypothesis corresponds to ACT-132577 being superior to placebo.

#### Type I and II errors and power

The type I error ( $\alpha$ ) is set to 0.05 (two-sided). The type II error is set to 0.10 and therefore the power to 90%.

#### **Primary analysis**

The primary analysis will be conducted on the PPS.

Change from baseline to Week 8 in mean trough office SiDBP will be analyzed using the MCP-Mod approach. In brief, it consists of a set of Multiple Contrast Tests (MCTs) to establish the existence of a dose-response and a set of pre-specified dose-response models to describe the dose-response curve.

Six candidate dose-response models will be considered: linear, linear in log-dose, quadratic,  $E_{max}$ , sigmoidal  $E_{max}$  and logistic. The analysis will be performed using the R-package DoseFinding. A dose-response relationship is demonstrated if

at least one of the six MCTs has an adjusted p-value < 0.05.

Supportive and sensitivity analyses will be conducted on the PPS and FAS. Change from baseline to Week 8 of DB treatment period (Period II) in mean trough SiDBP (imputed by last observation carried forward, if applicable) will also be analyzed using an analysis of covariance model with a factor for treatment group (placebo and four doses of ACT-132577) and a covariate for baseline mean trough SiDBP. Each of the four doses of ACT-132577 will be compared to placebo applying the Dunnett's test.

#### Secondary analyses

Secondary efficacy variables will be analyzed for the PPS at  $\alpha = 0.05$  (two-sided) using 95% confidence intervals (CIs). No correction for multiple testing will be applied for these analyses.

#### Safety analyses

Safety analyses will be performed on the Safety Set. Safety data will be summarized using descriptive statistics.

#### **Interim** analysis

No formal interim analysis is planned.

#### Sample size

In a previous study with macitentan in essential hypertension (AC-055-201) the within-group standard deviation (SD) for the change from baseline to Week 8 in SiDBP was 7.4 mmHg (90% CI: 7.0–8.0).

It is assumed that the maximum difference versus placebo is achieved at the highest dose of ACT-132577.

For the sample size it was required that the power to demonstrate the existence of a dose-response relationship—conservatively assuming a maximum difference versus placebo of 4 mmHg and an SD = 9 mmHg— is 90%. A total of 70 subjects per group in the PPS (i.e., 420 subjects in total) satisfied this condition and would also allow for sufficiently precise estimation of the dose-response curve. Assuming a drop-out rate of approximately 20%, a total of 90 patients per group would need to be randomized (i.e., 540 in total).

| | A blinded sample size re-estimation will be performed by the sponsor after 100 subjects have been randomized and their Week 8 BP data are available for analysis. The sample size will be recalculated considering the overall SD of the primary endpoint (change from baseline to Week 8 in mean trough SiDBP, measured by OBPM) in the PPS. The recalculated size of the PPS is expected to be between 280 subjects and the originally foreseen 420 subjects. The associated number of subjects to be randomized will also be re-estimated and is expected to be between 300 subjects and the originally planned 540 subjects. See Section 11.5.3 for more details. |
|---|---|
| STUDY COMMITTEES | An Independent Liver Safety Data Review Board (an external expert committee of hepatologists) provides ongoing assessment and advice regarding any hepatic events that may require further evaluation during the study. |

#### B. Calculation of mean blood pressure measurements based on ABPM

Example code. The SAS code to implement the trapezoidal rule

$$\int_a^b f(x)\,dx pprox rac{1}{2} \sum_{k=1}^N \left(x_{k+1} - x_k
ight) \left(f(x_{k+1}) + f(x_k)
ight).$$

is given below. Here it is assumed that the input data set (&dset) contains variables *subjid*, *visited*, *abgrpid* (to separate ABPMs of the same subject at the same visit, in the unlikely event that two ABPMs were taken).

Variable *ABBPTM* contains the 48-hour clock time of the measurement. For measurements taken on the second day 24 hours will be added to the 24-hour clock time. Variables ABDIA and ABSYS contain the DBP and SBP (mmHg), respectively.



**Example data.** The data plotted in Figure 1 are:

| ABPM date blood<br>pressure reading | | ABPM diastolic blood pressure (mmHg) | • |
|---|---|---|---|
| 18MAY2016 | 10:29 | 107 | 146 |
| 18MAY2016 | 10:31 | 100 | 150 |
| 18MAY2016 | 10:33 | 103 | 154 |
| 18MAY2016 | 10:35 | 101 | 157 |
| 18MAY2016 | 10:40 | 100 | 144 |
| 18MAY2016 | 11:00 | 107 | 146 |

| ABPM date blood pressure reading | ABPM time of blood pressure reading | ABPM diastolic blood pressure (mmHg) | ABPM systolic blood pressure (mmHg) |
|---|---|---|---|
| 18MAY2016 | 11:20 | 100 | 146 |
| 18MAY2016 | 11:40 | 114 | 150 |
| 18MAY2016 | 12:00 | 109 | 140 |
| 18MAY2016 | 12:23 | 122 | 167 |
| 18MAY2016 | 12:43 | 73 | 91 |
| 18MAY2016 | 13:00 | 109 | 148 |
| 18MAY2016 | 13:20 | 95 | 147 |
| 18MAY2016 | 13:40 | 94 | 141 |
| 18MAY2016 | 14:00 | 95 | 126 |
| 18MAY2016 | 14:20 | 89 | 120 |
| 18MAY2016 | 14:40 | 84 | 135 |
| 18MAY2016 | 15:00 | 96 | 140 |
| 18MAY2016 | 15:20 | 95 | 139 |
| 18MAY2016 | 15:40 | 82 | 138 |
| 18MAY2016 | 16:03 | 100 | 135 |
| 18MAY2016 | 16:23 | 103 | 144 |
| 18MAY2016 | 16:40 | 98 | 137 |
| 18MAY2016 | 17:20 | 102 | 147 |
| 18MAY2016 | 17:43 | 93 | 145 |
| 18MAY2016 | 18:00 | 93 | 159 |
| 18MAY2016 | 18:20 | 107 | 151 |
| 18MAY2016 | 18:40 | 95 | 135 |
| 18MAY2016 | 19:00 | 100 | 129 |
| 18MAY2016 | 19:20 | 99 | 130 |
| 18MAY2016 | 19:40 | 96 | 129 |
| 18MAY2016 | 20:00 | 101 | 129 |
| 18MAY2016 | 20:20 | 94 | 126 |
| 18MAY2016 | 20:40 | 91 | 124 |
| 18MAY2016 | 21:00 | 86 | 118 |
| 18MAY2016 | 21:23 | 83 | 116 |
| 18MAY2016 | 21:40 | 90 | 123 |
| 18MAY2016 | 22:00 | 86 | 121 |

| ABPM date blood | ABPM time of blood | ABPM diastolic blood | ABPM systolic blood |
|---|---|---|---|
| pressure reading | pressure reading | pressure (mmHg) | pressure (mmHg) |
| 18MAY2016 | 22:40 | 94 | 169 |
| 18MAY2016 | 23:00 | 95 | 150 |
| 18MAY2016 | 23:30 | 97 | 135 |
| 19MAY2016 | 00:03 | 144 | 180 |
| 19MAY2016 | 01:00 | 83 | 117 |
| 19MAY2016 | 01:30 | 74 | 129 |
| 19MAY2016 | 02:00 | 70 | 127 |
| 19MAY2016 | 02:30 | 62 | 124 |
| 19MAY2016 | 03:00 | 60 | 121 |
| 19MAY2016 | 03:30 | 66 | 127 |
| 19MAY2016 | 04:00 | 71 | 137 |
| 19MAY2016 | 04:30 | 95 | 140 |
| 19MAY2016 | 05:00 | 97 | 140 |
| 19MAY2016 | 05:30 | 92 | 161 |
| 19MAY2016 | 06:00 | 111 | 180 |
| 19MAY2016 | 06:20 | 115 | 178 |
| 19MAY2016 | 06:40 | 121 | 177 |
| 19MAY2016 | 07:00 | 117 | 173 |
| 19MAY2016 | 07:20 | 120 | 177 |
| 19MAY2016 | 07:40 | 112 | 173 |
| 19MAY2016 | 08:00 | 113 | 161 |
| 19MAY2016 | 08:20 | 130 | 221 |
| 19MAY2016 | 09:00 | 121 | 167 |
| 19MAY2016 | 09:20 | 100 | 177 |
| 19MAY2016 | 09:40 | 117 | 174 |
| 19MAY2016 | 10:20 | 117 | 179 |
| 19MAY2016 | 10:43 | 89 | 161 |
| 19MAY2016 | 11:00 | 92 | 190 |
| 19MAY2016 | 11:04 | 104 | 158 |

ABPM = ambulatory blood pressure monitoring.
**Example calculations.** The total duration of the ABPM (24h 35 mins) was shorter than 25 hours, so all measurements were included in the calculation of the 24-hour mean DBP and SBP for this subject at this visit. The calculations based on these data are:

- The areas under the DBP and SBP curves are 8,640,870 and 12,956,970 mmHg sec, respectively. Dividing both areas by the time span of 88,500 seconds gives a 24-hour means of 97.6 and 146.4 mmHg, respectively.
- The mean daytime DBP = (3,705,300 + 801,570) / (37,860 + 7440) = 99.5 mHg.
- The mean daytime SBP = (5,224,530 + 1,295,970) / (37,860 + 7440) = 143.9 mmHg.
- The mean night time DBP = 1,411,200 / 18,000 = 78.4 mmHg.
- The mean night time SBP = 2,438,100 / 18,000 = 135.5 mmHg.

Note that measurements between 21:00 on the first day and 01:00 on the second day (limits excluded) and between 06:00 and 09:00 on the second day (limits excluded) are included in the calculation of the 24-hour means, but not in the calculation of the daytime or night time means.

#### C. Calculation of trough-peak ratios based on ABPM

The figure below shows the mean diastolic ABPM by hour for a single treatment group at baseline (black) and Week 8 (red).

- The mean diastolic ABPM at trough is the average difference between the curves between 20 and 24 hours (circles)
- The mean diastolic ABPM at peak is the average difference between the curves between 2 and 6 hours (circles)

The trough to peak ratio for DBP based on ABPM is the ratio of the two.

The trough to peak ratio for SBP based on ABPM is calculated similarly.



## D. Document history

| Version | Effective Date | Reason |
|----------------|----------------|-----------------------|
| 1.0 8 May 2017 | | New |
| 2.0 | 15 May 2017 | Update pre-unblinding |



## STATISTICAL ANALYSIS PLAN

## FOR SAMPLE SIZE RE-ESTIMATION

## **STUDY AC-080A201**

Purpose of Analysis Blinded Sample Size Re-estimation

Investigational Drug ACT-132577

Protocol Number AC-080A201

Idorsia Document Number D-17.086

Document Status/Version Number Final Version 2

Date 3 November 2017

Author , Expert Statistician

Reviewers Senior Expert Statistician

, VP Science Medical Expert

Property of Idorsia Pharmaceuticals Ltd


May not be used, divulged, published or otherwise disclosed without the consent of Idorsia Pharmaceuticals Ltd

## TABLE OF CONTENTS

| ST OF ABBREVIATIONS AND ACRONYMS | 4 |
|---|---|
| INTRODUCTION | 5 |
| 2.1 Study design | 5 |
| OBJECTIVES | 9 |
| CHANGES OR CLARIFICATIONS TO ANALYSES PLANNED IN THE STUDY PROTOCOL | 9 |
| 5.2 Subject characteristics 5.3 Study treatment exposure and compliance 5.4 Study discontinuation 5.5 Efficacy variables 5.5.1 Primary efficacy endpoint(s) | 9<br>9<br>9 |
| DEFINITION OF PROTOCOL DEVIATIONS | 10 |
| 7.1 Definitions of analysis sets | 10<br>10 |
| DEFINITION OF SUBGROUPS | 10 |
| GENERAL STATISTICAL METHODOLOGY | 11 |
| 10.1 Overall testing strategy | 15 |
| | INTRODUCTION. STUDY DESIGN AND FLOW. 2.1 Study design |

| | 10.4 | Analyses of subject characteristics | 16 |
|---|---|---|---|
| | 10.5 | Analysis of study treatment exposure and compliance | |
| | 10.6 | Analysis of the primary efficacy variable(s) | |
| | | 6.1 Hypothesis and statistical model | |
| | | 6.2 Handling of missing data | |
| | | 6.3 Main analysis | |
| | 10.7 | Analysis of the secondary efficacy variables | |
| | 10.8 | Analysis of other efficacy variables | |
| | 10.9 | Analysis of safety variables | |
| | 10.10 | Analysis of quality of life variables | |
| | 10.11 | Analysis of pharmacoeconomic variables | 17 |
| | 10.12 | Analysis of epidemiological measures and risk-benefit evaluations | 17 |
| | 10.13 | Analysis of pharmacodynamic variables | 17 |
| | 10.14 | Analysis of pharmacokinetic variables | |
| 11 | GENER | AL DEFINITIONS AND DERIVATIONS | 17 |
| | 11.1 | Time windows | 17 |
| 12 | HANDI | LING OF MISSING/INCOMPLETE DATE AND TIME FIELDS | 18 |
| 12 | LICTO | E CHAMADY TADIES LISTINGS AND EIGHDES | 1.0 |
| 13 | LISTO | F SUMMARY TABLES, LISTINGS AND FIGURES | |
| | 13.1 | Subject disposition | |
| | 13.2 | Subject characteristics | |
| | 13.3 | Primary efficacy variable | |
| | 13.4 | Secondary efficacy analyses | 20 |
| 1.4 | DEFED | DNGEG | 20 |
| 14 | KEFEK | ENCES | 20 |
| 15 | ΔPPFN | DICES | 21 |
| 13 | | | |
| | 15.1 | Layouts | |
| | | 1.1 Layout T1 | |
| | | 1.2 Layout T2 | |
| | | 1.3 Layout T3 | |
| | | 1.4 Layout F1 | |
| | | 1.5 Layout F2 | |
| | 15.2 | R Program for power MCP-Mod approach | |
| | 10.3 | R Program to compare group standard deviations | |

Statistical Analysis Plan Sample Size Re-estimation Doc No D-17.086

## LIST OF ABBREVIATIONS AND ACRONYMS

| BP | Blood pressure |
|---------|-----------------------------------------------|
| eCRF | Electronic Case Report Form |
| FAS | Full Analysis Set |
| MCP-Mod | Multiple Comparison Procedure - Modeling |
| OBPM | (Automated) office blood pressure measurement |
| PD | Protocol deviation |
| PPS | Per-Protocol Set |
| RND | All Randomized Set |
| SAP | Statistical Analysis Plan |
| SD | Standard deviation |
| SiDBP | Sitting diastolic blood pressure |
| SiSBP | Sitting systolic blood pressure |
| SSR | Sample size re-estimation |

Statistical Analysis Plan Sample Size Re-estimation

Doc No D-17.086

#### INTRODUCTION

This Statistical Analysis Plan (SAP) describes statistical analyses required for the blinded sample size re-estimation (SSR) of Study AC-080A201, the Phase 2 dose-finding trial of the ACT-132577 project.

The objective is to provide the sizes of the Per-Protocol Set (PPS) and Full Analysis Set (FAS) which, given the observed variability at this point in time, will guarantee approximately 90% power to detect a dose response relationship and provide sufficient precision in the estimation of the dose response curve and of doses that will be selected for the Phase 3 program of ACT-132577.

The blinded SSR will be performed by the sponsor after 100 subjects have been randomized and their Week 8 blood pressure (BP) data are available for analysis. The sample size will be recalculated considering the overall standard deviation (SD) of the primary endpoint (change from baseline to Week 8 in mean trough sitting diastolic blood pressure [SiDBP], measured by automated office blood pressure measurement [OBPM]) in the Per-Protocol Set.

The re-calculated size of the PPS is expected to be between 280 subjects and the originally foreseen 420 subjects. The associated number of subjects to be randomized will also be re-estimated and is expected to be between 300 subjects and the originally planned 540 subjects. It is anticipated that the size of the PPS will be at least 80% of the size of the FAS.

This SAP is based on Version 3 of the Protocol dated 30 May 2016 [D-16.063].

Version 2 of this SAP was generated in order to make editorial corrections—no changes were made to analyses or statistical content—and to reflect the transfer of ownership of ACT-132577. ACT-132577 was previously developed by Actelion Pharmaceuticals Ltd. Actelion was recently acquired by Johnson & Johnson. As part of this transaction, Actelion spun off its drug discovery operations and early stage clinical development assets into an independent biopharmaceutical company, Idorsia Pharmaceuticals Ltd (Idorsia). ACT-132577 is now owned by Idorsia.

#### 2 STUDY DESIGN AND FLOW

#### 2.1 Study design

Study AC-080A201 is a prospective, multi-center, double-blind, double-dummy, randomized, placebo- and active-reference, parallel group, Phase 2 dose-finding study with ACT-132577 in subjects with essential hypertension (grade 1 and 2).

Approximately 1000 subjects are expected to be enrolled into the study (i.e., entered the run-in phase), in order to have at least 540 subjects randomized in the 6 following groups in a 1:1:1:1:1 ratio; placebo, 5 mg ACT-132577, 10 mg ACT-132577, 25 mg ACT-132577, 50 mg ACT-132577, lisinopril 20 mg. At least 420 subjects are expected to complete the trial.

## 2.2 Study visit and assessment schedule

Table 1 shows the study visit and assessments schedule.

Table 1 Visit and assessment schedule

| PERIODS | Name / duration | Period | I: Run-in / | Run-in / 4–6 weeks Period II: Double-blind / 8 weeks | | | Period III | I: withdrawal / 2 weeks | Premature<br>EOT | | Follow-up | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| VISITS | Number<br>Name | 1 <sup>6</sup><br>Week –6 | 2 <sup>6</sup><br>Week –4 | 3<br>Week -1 | 4 | 1 | 5<br>Week 2 | 6<br>Week 4 | Wee | 7<br>ek 8 | 8<br>Week 10 | 9 | U1, 2, 3, etc. <sup>10</sup> | Telephone<br>call <sup>9</sup> or visit <sup>11</sup> |
| | Name | Screening** | | | Randon | nization | | | DB- | EOT | WD-EOT | Within 7 days | Unscheduled | EOS |
| | TIME / Week | Day -42 | Day -28<br>(± 3 d) | Day -7<br>(± 4 d) | Pre-<br>Day -1 | Day 1 | 2<br>Day 14<br>(± 3 d) | 4<br>Day 28<br>(± 3 d) | Part 1 Day 55 (± 5 d) | Part 2<br>Day 56 | 10<br>Day 70<br>(± 3 d) | after last study<br>treatment<br>intake | | 30–33 d after last<br>dose of DB treatment |
| Infor | med consent | X | | | | | | | | | | | | |
| E | ligibility | X | X | X | X | | | | | | | | | |
| Med | lical history | X | | | | | | | | | | | | |
| Physic | al examination | X | X | X | X | | X | X | X | | X | X | X | |
| Concomi | itant medications | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HR*, bod | ly weight, height <sup>1</sup> | X | X | X | X | | X | X | X | | X | X | X | |
| 12-lead ECG | * | X <sup>4</sup> | | | X <sup>9</sup> | | | X | X | | X | X <sup>9</sup> | X | |
| Laboratory in | ncl. pregnancy tests*2 | X <sup>5</sup> | | X <sup>9</sup> | X <sup>9</sup> | | X | X | X | | X | X <sup>9</sup> | X | X <sup>2</sup> |
| τ | Jrinalysis | | X <sup>7, 9</sup> | | X <sup>9</sup> | | X | X | X | | X | X <sup>9</sup> | X | |
| Office B | P measurement* | X | X | X | X | | X | X | X | | X | X | X | |
| Home | e BP device <sup>12</sup> | X | | | | | | | | | | | <b>&gt;</b> | |
| Ambulatory | BP measurement* | | | | X | | | | X | | | | | |
| PK and | PD sampling <sup>13</sup> | | | | | | X | X | X | | | | | |
| Compliance | with study treatment | | X <sup>9</sup> | X <sup>9</sup> | X | | X | X | X | | X | X | X | |
| Study treatm | ent dispensing/return | X | X <sup>8</sup> | | X | X | | X | X | X | X | X | X | |
| Adv | erse events <sup>3</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serious | adverse events <sup>3</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |

# Statistical Analysis Plan Confidential Sample Size Re-estimation Doc No D-17.086

#### \*Electronically transferred to sponsor.

\*\* Visit 1 (screening) can last up to 72 h for obtaining informed consent and performing required assessments.

- 1. Height is only measured at Visit 1.
- 2. Serum pregnancy test only for women of childbearing potential. Result is transferred electronically to sponsor.
- 3. All AEs and SAEs that occur after signing the Informed Consent Form and up to 30 days after last DB study treatment intake must be reported.
- 4. Historical ECG is accepted if not older than 6 months.
- 5. Historical blood laboratory data is accepted to check exclusion criterion 15, if not older than 3 months. In such a case, for women of childbearing potential a urine pregnancy test must be performed. If no historical report is available, a blood sample to be taken for laboratory analysis (including pregnancy test for women of childbearing potential) by central laboratory.
- 6. Run-in period is 4 weeks before randomization for anti-hypertensive treatment naïve subjects. Visit 1 is combined with Visit 2. Run-in period is 6 weeks before randomization for subjects on anti-hypertensive treatment. Visit 1 and Visit 2 must be performed.
- 7. Only urine pregnancy test for women of childbearing potential. Result is captured in the eCRF.
- 8. Only for subjects who were on anti-hypertensive drugs at Visit 1 (i.e., had to perform a Visit 2).
- 9. If subject discontinued study treatment during run-in period (i.e., between run-in visits) or at an in-person run-in visit (e.g., Visit 3), these tests may not be performed
- 10. Unscheduled visits may be performed at any time during the study and may include all or some of the indicated assessments, based on the judgment of the investigator.
- 11. For women of childbearing potential a visit must be organized instead of the telephone call to perform the serum pregnancy test at the site. However, if a woman of childbearing potential discontinued study treatment during the run-in period, a telephone call can be made instead of the visit.
- 12. Upon investigator's judgment, a home monitoring device will be dispensed to monitor BP at home, if necessary.
- 13. Sample to be taken at trough (i.e., prior to study treatment intake).

AE = adverse event; BP = blood pressure; DB = double-blind; ECG = electrocardiogram; eCRF = electronic case report form; EOS = End-of-Study; EOT = End-of-Treatment; HR = heart rate; PD = pharmacodynamics; PK = pharmacokinetics; SAE = serious adverse event; WD = withdrawal.

#### 3 OBJECTIVES

The objective of this Sample Size Re-estimation is to provide the sizes of the PPS and FAS which, given the observed variability at this point in time, will guarantee approximately 90% power to detect a dose response relationship and provide sufficient precision in the estimation of the dose response curve and of doses that will be selected for the Phase 3 program of ACT-132577.

# 4 CHANGES OR CLARIFICATIONS TO ANALYSES PLANNED IN THE STUDY PROTOCOL

Not applicable.

#### 5 DEFINITIONS OF VARIABLES

Baseline refers to the last non-missing value before double-blind treatment start date.

#### 5.1 Screening failures

Not applicable.

#### 5.2 Subject characteristics

Not applicable.

### 5.3 Study treatment exposure and compliance

Not applicable.

#### 5.4 Study discontinuation

Not applicable.

#### 5.5 Efficacy variables

#### 5.5.1 Primary efficacy endpoint(s)

The primary efficacy endpoint is the change from baseline to Week 8 of double-blind treatment period (Period II) in mean trough (i.e., 24 hours post-dose) SiDBP, measured by OBPM.

Here, baseline is defined as in Section 5 and Week 8 is the time window of Visit 7 [Section 11.1]. OBPM SiDBP is measured by BpTRU<sup>®</sup> (automated; average over five measurements) and is collected via electronic data transfer from an external will not be (re-)calculated by the sponsor.

All assessments (including the unscheduled ones) are considered and re-assigned to the most appropriate visit according to the time windows described in Section 11.1.

#### 5.5.2 Secondary efficacy endpoint

Of the secondary efficacy endpoints defined in the protocol, the following is considered as supportive for the sample size re-estimation:

• Change from baseline to Week 8 of double-blind treatment period (Period II) in mean trough SiSBP, measured by OBPM.

Here, baseline is defined as in Section 5 and Week 8 is the time window of Visit 7 [Section 11.1]. OBPM SiSBP is collected via electronic data transfer and will not be (re-)calculated by the sponsor.

All assessments (including the unscheduled ones) are considered and re-assigned to the most appropriate visit according to the time windows described in Section 11.1.

#### 5.6 Safety variables

Not applicable.

#### 6 DEFINITION OF PROTOCOL DEVIATIONS

For the purpose of this SSR only two major protocol deviations (PDs) will be considered in the definition of the PPS [see Section 7.1.3].

- Not completing the double-blind treatment period: no Week 8 (i.e., time window Visit 7) efficacy data available.
- Use of forbidden medication, indicated as protocol deviation (PD code list version 2, PV MM.503).

#### 7 ANALYSIS SETS

#### 7.1 Definitions of analysis sets

#### 7.1.1 All Randomized Set

The All Randomized Set (RND) includes all subjects with answer 'YES' to the question 'Was the subject randomized?' in the **Randomization** eCRF.

#### 7.1.2 Full Analysis Set

The FAS includes all subjects in the RND Set, who have a baseline mean trough SiDBP.

#### 7.1.3 Per-Protocol Set

The PPS includes all subjects from the FAS who have a mean trough SiDBP at Week 8 (i.e., time window Visit 7) and did not use forbidden medication deviation as defined in Section 6.

#### 8 DEFINITION OF SUBGROUPS

Not applicable.

#### GENERAL STATISTICAL METHODOLOGY

A blinded SSR will be performed by the sponsor after 100 subjects have been randomized and their Week 8 (time window Visit 7) OBPM data are available for analysis. The SSR will consider the overall standard deviation (i.e., based on pooled treatment groups as the SSR is blinded) of the primary endpoint (change from baseline to Week 8 [time window Visit 7] in mean trough SiDBP, measured by OBPM) in the PPS.

The primary endpoint (change from baseline to Week 8 [time window Visit 7] of double-blind treatment period in mean trough SiDBP) will be analyzed using the MCP-Mod approach [Bretz 2005, Pinheiro 2006, EMA 2013]. The blinded SSR will be based on the average power achieved in the MCP-Mod approach, to detect a dose response when the 'true' dose-response curve is among the four curves displayed in (copied from protocol figure 2). All four assume that the minimum Figure 1 response will be obtained with placebo (0 mg) and the maximum response (4–5 mmHg, placebo corrected) will be reached at the highest dose of ACT-132577 (50 mg).

Figure 1 Dose response relationships used in power calculations



For each of the four dose-response curves the power will be calculated using the powMCT function in the R-package DoseFinding [Bornkamp 2016]. R-code is included in Appendix 15.1.

Statistical Analysis Plan Sample Size Re-estimation Doc No D-17.086

The calculation requires an estimate of the standard deviation of the primary endpoint [see Section 10.6] in the PPS. The *average* power is displayed in Figure 2 for primary endpoint SDs ranging from 6-9 mmHg. (For the original sample size calculation 9 mmHg was assumed and > 95% power was required for each of the four scenarios separately.)

Figure 2 Average power to detect dose response

Black SD = 6.0; Red SD = 6.5; Blue SD = 7.0; Green SD = 7.5; Orange SD = 8.0; Purple SD = 8.5; Grey SD = 9.0.



The associated sample sizes (PPS) for 80–95% average power are given in Table 2.

Table 2 Sample size (PPS) needed for 80–95% power to detect a dose-response across various SDs

| | SD = 6.0 | SD = 6.5 | SD = 7.0 | SD = 7.5 | SD = 8.0 | SD = 8.5 | SD = 9.0 |
|---|---|---|---|---|---|---|---|
| 80% power | | | | | | | |
| - PPS size | 126 | 150 | 174 | 198 | 222 | 252 | 282 |
| - per group* | 21 | 25 | 29 | 33 | 37 | 42 | 47 |
| 85% power | | | | | | | |
| - PPS size | 144 | 168 | 198 | 222 | 258 | 288 | 318 |
| - per group* | 24 | 28 | 33 | 37 | 43 | 48 | 53 |
| 90% power | | | | | | | |
| - PPS size | 174 | 198 | 234 | 264 | 300 | 336 | 378 |
| - per group* | 29 | 33 | 39 | 44 | 50 | 56 | 63 |
| 95% power | | | | | | | |
| - PPS size | 210 | 252 | 288 | 330 | 372 | 420 | 474 |
| - per group* | 35 | 42 | 48 | 55 | 62 | 70 | 79 |

<sup>\*</sup>Expected number. Power based on the MCT test in the MCP-Mod procedure as implemented in the R DoseFinding package, averaged over the four dose-response curves in Figure 2 of this protocol.

Here, SD is the standard deviation of the primary endpoint (independent of treatment assignment, as this is blinded). It is acknowledged that this could be an overestimation of the (unobserved) within group SD, but, given the range of anticipated treatment group differences, this overestimation is likely to be small (< 5%; simulation program in Appendix 15.2). The re-calculated size of the PPS is expected to be between 280 subjects and the originally foreseen 420 subjects.

The associated number of subjects to be randomized will be calculated by dividing PPS size by the proportion of randomized subjects who were included in the PPS. That proportion will be estimated based on the same 100 randomized subjects considered for the blinded sample size re-estimation. To be conservative, the lower limit of the 95% CI around the proportion will be employed, of which some examples are given in Table 3.

MCP-Mod = Multiple Comparison Procedure - Modeling; MCT = Multiple Contrast Test; PPS = Per-Protocol Set; SD = standard deviation.

Table 3 Number and proportion of subjects in PPS and 95% CIs for the proportion at the time of the sample size re-estimation

| Number | Number | Proportion | 95% CI* | |
|------------|--------|------------|---------|------|
| Randomized | in PPS | in PPS | | |
| 100 | 95 | 0.95 | 0.89 | 0.98 |
| 100 | 90 | 0.90 | 0.82 | 0.95 |
| 100 | 85 | 0.85 | 0.76 | 0.91 |
| 100 | 80 | 0.80 | 0.71 | 0.87 |

<sup>\*</sup>Clopper-Pearson [Clopper 1934]

The re-calculated number of subjects randomized is expected to be between 300 subjects and the originally foreseen 540 subjects.

#### 10 STATISTICAL ANALYSES

#### 10.1 Overall testing strategy

The SSR will be based on blinded data. No statistical testing will be performed.

#### 10.2 General rules for data presentations

Output titles should include the name of the analysis set used for the analysis, and if specific period used, also the time period.

Table column headers should provide the number of subjects of the used analysis set.

The footer should provide the following information:

- the date and time of the data extraction from the database and the cut-off date,
- the date and time of the output generation,
- the SAS program that produces the output and the author,

No acronym/abbreviation should be used unless documented in the footer.

For categorical parameters, frequencies/numbers and percentages should be used. Percentages should be presented with one decimal place (e.g., 18.2%).

Descriptive statistics for continuous variables are given in Table 4.

The number of subjects to be randomized will also take into account the need to collect sufficient exposure and safety data and is expected to be between 300 subjects and the originally planned 540 subjects.

CI = confidence interval; PPS = Per-Protocol Set.

Table 4 Descriptive statistics for continuous variables

| Statistics | Display | Number of decimals | Example |
|---|---|---|---|
| N | N | None | 99 |
| Mean | Mean | Original digit + 1 | 45.2 |
| Standard Deviation | Standard<br>Deviation | Original digit + 1 | 38.5 |
| Median | Median | Original digit + 1 | 45.3 |
| Minimum-Maximum | Min-Max | Original digit | 125–250 |
| $1^{\text{st}}$ quartile (25%) $-3^{\text{rd}}$ quartile (75%) | Q1-Q3 | Original digit + 1 | 35.2–58.5 |

### 10.3 Display of patient disposition and analysis sets

The number of patients in the FAS and PPS will be tabulated on pooled treatment groups.

## 10.4 Analyses of subject characteristics

Not applicable.

#### 10.5 Analysis of study treatment exposure and compliance

Not applicable.

#### 10.6 Analysis of the primary efficacy variable(s)

The primary efficacy variable will be analyzed in the PPS and FAS, based on pooled treatment groups.

#### 10.6.1 Hypothesis and statistical model

Not applicable.

#### 10.6.2 Handling of missing data

The PPS analysis will be based on observed data.

In the FAS, last post-baseline measurement will be carried forward.

#### 10.6.3 Main analysis

The changes from baseline to Weeks 2, 4 and 8 of double-blind treatment period (time window Visits 5, 6 and 7 respectively) in mean trough SiDBP (measured by OBPM) will be summarized using descriptive statistics.

The distribution of the changes from baseline in SiDBP will be displayed in a density plot.

#### 10.7 Analysis of the secondary efficacy variables

Secondary efficacy endpoints will be analyzed in the PPS.

Statistical Analysis Plan Sample Size Re-estimation Doc No D-17.086

rantment paried (time

The changes from baseline to Weeks 2, 4 and 8 of double-blind treatment period (time window Visits 5, 6 and 7, respectively) in mean trough SiSBP (measured by OBPM) will be summarized using descriptive statistics.

The distribution of the changes from baseline in SiSBP will be displayed in a density plot.

#### 10.8 Analysis of other efficacy variables

Not applicable.

#### 10.9 Analysis of safety variables

Not applicable.

#### 10.10 Analysis of quality of life variables

Not applicable.

#### 10.11 Analysis of pharmacoeconomic variables

Not applicable.

#### 10.12 Analysis of epidemiological measures and risk-benefit evaluations

Not applicable.

#### 10.13 Analysis of pharmacodynamic variables

Not applicable.

#### 10.14 Analysis of pharmacokinetic variables

Not applicable.

#### 11 GENERAL DEFINITIONS AND DERIVATIONS

#### 11.1 Time windows

To allow analysis of data at the relevant planned (scheduled) visits, all recorded assessments, including unscheduled ones, are re-assigned to the most appropriate visit according to the best fitting time-window for that visit [see Table 5].

Table 5 Visit time windows

| Visit | Period | Target day | Min day | Max day |
|----------------|------------------|------------|---------|----------|
| 1 | I: Run-in | -42 | _ | -35 |
| 2 | | -28 | -34 | -18 |
| 3 | | -7 | -17 | -4 |
| 4 <sup>a</sup> | | -1 | -3 | -1 |
| 5 <sup>b</sup> | II: Double-blind | 14 | 1 | 21 |
| 6 <sup>b</sup> | | 28 | 22 | 42 |
| 7 <sup>b</sup> | | 55 | 43 | EOT |
| 8° | III: Follow-up | 70 | EOT | No limit |

<sup>&</sup>lt;sup>a</sup>Measurements mapped to Visit 4 must be before randomization; otherwise map to Visit 3

EOT = End-of-Treatment.

If more than one assessment falls within the same time window, the closest value to the planned time point will be assigned to the re-mapped visit. In the event of equidistant values from the planned time point, the last assessment will be considered for the analyses.

## 12 HANDLING OF MISSING/INCOMPLETE DATE AND TIME FIELDS Not applicable.

#### 13 LIST OF SUMMARY TABLES, LISTINGS AND FIGURES

All outputs will be generated based on blinded data.

The TLF naming conventions consider three components: Type (T, L, F), Name (free text, in general not more than eight characters, but if required to maintain uniqueness, up to a maximum of ten characters), Suffix (for example, for analysis sets, or subgroups, not longer than four characters) - multiple suffixes can be added. Components/suffixes are separated by ' '. Example: T TEAE RND, summary table (T) of treatment-emergent adverse events (TEAE) on all randomized analysis set (RND).

## 13.1 Subject disposition

| Output name | Display* | Title (Description) | Analysis set(s)** | Mock layout |
|---|---|---|---|---|
| ANSETOV | T | Composition of FAS and PPS | RND | T1 |

<sup>\*</sup>T = Summary table, L = Listing, F = Figure, \*\*RND = All Randomized Set, FAS = Full Analysis Set, PPS = Per-Protocol Set

<sup>&</sup>lt;sup>b</sup>Measurements mapped to Visit 5, 6 or 7 must be before the patient's EOT; otherwise map to Visit 8

<sup>&</sup>lt;sup>c</sup>Measurements taken on Visit 8 must be after the patient's EOT; otherwise map to Visit 7

## 13.2 Subject characteristics

| Output<br>name | Display* | Title (Description) | Analysis set(s)** | Mock layout |
|---|---|---|---|---|
| DEM | T | Demographic Characteristics | R | T2 |

<sup>\*</sup> T = Summary table, L = Listing, F = Figure, \*\*SC = Screened Analysis Set, R = All Randomized Set

## 13.3 Primary efficacy variable

| Output name | Display* | Title (Description) | Analysis set(s)** | Mock<br>layout |
|---|---|---|---|---|
| DIA_OBPM_CHG | T | Change from baseline in<br>Sitting Diastolic Blood<br>Pressure as Measured by<br>OBPM by Visit | FAS, PPS | Т3 |
| DIA_OBPM_CHG | F | Distribution of Change from<br>baseline in Sitting Diastolic<br>Blood Pressure as Measured<br>by OBPM by Visit | PPS | F1 |

<sup>\*</sup>T = Summary table, L = Listing, F = Figure, \*\*RND = All Randomized Set, FAS = Full Analysis Set, PPS = Per-Protocol Set

#### 13.4 Secondary efficacy analyses

| Output name | Display* | Title (Description) | Analysis set(s)** | Mock layout |
|---|---|---|---|---|
| SYS_OBPM_CHG | T | Change from baseline in<br>Sitting Systolic Blood<br>Pressure as Measured by<br>OBPM by Visit | PPS | Т3 |
| SYS_OBPM_CHG | F | Distribution of Change from<br>baseline in Sitting Systolic<br>Blood Pressure as Measured<br>by OBPM by Visit | PPS | F1 |
| COR_OBPM_CHG | F | Correlation between change<br>from baseline in Diastolic<br>and Systolic Blood Pressure<br>by Visit | PPS | F2 |

<sup>\*</sup>T = Summary table, L = Listing, F = Figure, \*\*RND = All Randomized Set, FAS = Full Analysis Set, PPS = Per-Protocol Set

#### 14 REFERENCES

- [Bornkamp 2016] Bornkamp B, Pinheiro J, Bretz F. Planning and Analyzing Dose Finding experiments. Retrieved from: cran.r-project.org/web/packages/DoseFinding
- [Bretz 2005] Bretz F, Pinheiro, JC, Branson M. Combining multiple comparisons and modeling techniques in dose-response studies Biometrics. 2005;61:738–48.
- [Clopper 1934] Clopper C, Pearson ES. The use of confidence or fiducial limits illustrated in the case of the binomial. Biometrika 1934;26:404–13.
- [Pinheiro 2006] Pinheiro JC, Bornkamp B, Bretz F. Design and analysis of dose-finding studies combining multiple comparisons and modeling procedures, J Biopharm Stat. 2006;16:639–56.
- [EMA 2013] EMA/CHMP/SAWP/757052/2013. Qualification Opinion of MCP-Mod as an efficient statistical methodology for model-based design and analysis of Phase II dose finding studies under model uncertainty.

Statistical Analysis Plan Sample Size Re-estimation Doc No D-17.086

## 15 APPENDICES

## 15.1 Layouts

### 15.1.1 Layout T1

ACT-132577

Protocol: AC-080A201/Essential Hypertension

<Title>

Analysis set: <analysis set>

<overall, site x>

| | Tre | inded<br>atment<br>= XX<br>(%) |
|--------------------------|-----|--------------------------------|
| Subjects Randomized | xx | (уу.у) |
| Subjects Included in FAS | XX | (yy.y) |
| Subjects Included in PPS | XX | (уу.у) |

Output: XXXX, Produced by xxxxxxxx on ddmmmyyyy hh:mm (CET), Data Extraction Date: ddmmmyyyy,

Cut-Off Date: ddmmmyyyy

Program: prod\_ccm/program\_output/program\_name.sas

Page x of x

## 15.1.2 Layout T2

ACT-132577

Protocol: AC-080A201/Essential Hypertension

<Title>

Analysis set: <analysis set>

| | Blinded<br>Treatment<br>N = XX |
|---|---|
| Age (years) | xx |
| Mean | XX.XX |
| Standard Deviation | XX.XX |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| Min, Max | XX.X, XX.X |
| Sex [n (%)] Females Males Missing | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |
| Race [n (%)] Black or African American American Indian or Alaska Native Native Hawaiian or Other Pacific Islander Asian White Other Missing | xx (xx.x) |
| Ethnicity [n (%)] Hispanic or Latino Not Hispanic or Latino Missing | xx (xx.x)<br>xx (xx.x)<br>xx (xx.x) |

Output: XXXX, Produced by xxxxxxxx on ddmmmyyyy hh:mm (CET), Data Extraction Date: ddmmmyyyy, Cut-Off Date: ddmmmyyyy

Program: prod\_ccm/program\_output/program\_name.sas

Page x of x

Statistical Analysis Plan Sample Size Re-estimation Doc No D-17.086

## 15.1.3 Layout T3

ACT-132577

Protocol: AC-080A201/Essential Hypertension

<Title>

Analysis set: <analysis set>

<Parameter (unit)>, Time point x>

| N = XX |
|--------------|
| XX |
| XX.XX |
| XX.XX |
| XX.X |
| XXX.X, XXX.X |
| xx.x, xx.x |
| XX |
| XX.XX |
| XX.XX |
| XX.X |
| xxx.x, xxx.x |
| XX.X, XX.X |
| oint x> |
| XX |
| XX.XX |
| XX.XX |
| XX.X |
| XXX.X, XXX.X |
| XX.X, XX.X |

Output: XXXX, Produced by xxxxxxxx on ddmmmyyyy hh:mm (CET), Data Extraction Date: ddmmmyyyy,

Cut-Off Date: ddmmmyyyy

Program: prod\_ccm/program\_output/program\_name.sas

Page  $\mathbf{x}$  of  $\mathbf{x}$ 

#### 15.1.4 Layout F1

ACT-132577 Protocol: AC-080A201/Essential Hypertension Analysis set: <analysis set> <Parameter (unit)>



```
proc kde data=<dset>;
 by avisitn;
 univar chg (bwm=1) / out=dens gridl=-40 gridu=20;
proc gplot data=dens;
 plot density*value=avisitn/ haxis=axis1 vaxis=axis2;
  symbol1 c=black i=j l=1;
  symbol2 c=red i=j l=1;
  symbol3 c=blue i=j l=1;
  axis1 order=(-40 to 20 by 5) minor=none;
 axis2 order=(0 to 0.06 by 0.01) minor=none;
run;
```

## 15.1.5 Layout F2

ACT-132577

Protocol: AC-080A201/Essential Hypertension

<Title>

Analysis set: <analysis set>



```
Some possible SAS statements
```

\* <dset> has change from baseline in DBP (cdbp) and in SBP (csbp)in separate columns;

```
proc corr data=<dset>;
                                                        proc sort;
                                                         by avisitn cdbp;
 by avisitn;
  var csbp cdbp;
                                                        run;
run;
                                                        proc gplot;
proc glm data=botht noprint;
                                                         by avisitn;
                                                          plot (csbp pred) *cdbp/ overlay;
 by avisitn;
 model csbp=cdbp;
                                                         run;
 output out=glmout predicted=pred;
```

## 15.2 R Program for power MCP-Mod approach

```
# powerDRssr.R JUN 2016
#setwd("<To be completed>")
## PRELIMINARIES
sigEmax <- function (ed50, ed90)
e0 <- 0
emax <- 1
hill < -log(9)/(log(ed90) - log(ed50))
c(ed50, round(hill,2))
} # Emax
# get ed50 and hill
# based on ed50 and ed90
black <- sigEmax (ed50=0.125, ed90=0.25)
red <- sigEmax (ed50=0.125, ed90=0.50)
blue <- sigEmax (ed50=0.25, ed90=0.50)
green \leftarrow sigEmax (ed50=0.25, ed90=0.75)
## FUNCTIONS
powerMCT <-function (doses, sigma, n, true) {</pre>
candMod <- Mods(linear = NULL, linlog = NULL, quadratic = -0.5, emax = 0.5,
                sigEmax = c(0.5, 0.5), logistic = c(0.5, 0.5), doses = doses)
contMat <- optContr(candMod, w = rep(n,length(doses)))</pre>
trueMod <- Mods(sigEmax = true, doses = doses)</pre>
power <- powMCT(contMat = contMat, altModels = trueMod, alpha = 0.05, alternative = "two.sided", n = n, sigma = sigma,
                placAdj = FALSE, df = NA, critV = TRUE, control = mvtnorm.control())
power
## MAIN
```

```
# load DoseFinding package
library(DoseFinding)
# doses in the study
d4 \leftarrow c(0, 0.05, 0.10, 0.25, 0.5)
# power
sigs < - seq (6,9,0.5)
nn < - seq (20,70,1)
pow<-matrix(NA,length(sigs)*length(nn),6)</pre>
k <- 1
for (i in 1:length(sigs)){
 for (j in 1:length(nn)){
    pow[k,1] <- sigs[i]
    pow[k,2] \leftarrow nn[j]
    pow[k,3] \leftarrow round(powerMCT (d4, sigs[i]/5, nn[j], black), 3)
    pow[k,4] \leftarrow round(powerMCT(d4, sigs[i]/4.5, nn[j], red), 3)
    pow[k,5] \leftarrow round(powerMCT (d4, sigs[i]/4.5, nn[j], blue), 3)
    pow[k,6] \leftarrow round(powerMCT (d4, sigs[i]/4, nn[j], green), 3)
    k <- k+1
  } # j
} # i
plot(pow[pow[,1]==6,2], rowMeans(pow[pow[,1]==6,3:6]), type="1", col="grey",
     xlab="group size (PPS)", ylab="power", xlim=c(20,70), ylim=c(0.6,1))
cols <- c("black","red","blue","green","orange","purple","grey")</pre>
for (i in 1:7) {
sel <- pow[pow[,1]==sigs[i],]</pre>
lines(sel[,2], rowMeans(sel[,3:6]), col=cols[i])
}
abline (h=c(0.8, 0.9, 0.95), col="grey")
```

3 November 2017, page 28/28

sim(n=90, means=m, sd=8, seed=1333)

## 15.3 R Program to compare group standard deviations

```
# simSD.R JUL 2016
# FUNCTIONS
sim <- function (n, means, sd, seed) {
  set.seed(seed)
  print (means)
  k <- length (means)
  var <- matrix(NA, nrep, 2)</pre>
  for (i in 1:nrep) {
    y \leftarrow rep(means, each=n) + rnorm(n*k, 0, sd)
    var[i,1] <- var(y) # overall variance</pre>
    x \leftarrow rep (1:k, each=n)
    A < -aov(y \sim as.factor(x))
    var[i,2] <- sum(A$residuals^2)/A$df.residual # within group variance</pre>
var <- colMeans(var)</pre>
print (round(c(var, var[1]/var[2]), 2))
sd <- sqrt(var)
round(c(sd, sd[1]/sd[2]), 2)
# MAIN
nrep <- 1000
m <- seq(0,5,length.out=6)
sim(n=90, means=m, sd=8, seed=1331)
m <- seq(0,6,length.out=6)
sim(n=90, means=m, sd=8, seed=1332)
m <- seq(0,8,length.out=6)</pre>
```